## **PROTOCOL PS0011 AMENDMENT 1**

A MULTICENTER, 48-WEEK, DOUBLE-BLIND,
PLACEBO-CONTROLLED, PARALLEL-GROUP EXTENSION
STUDY TO ASSESS THE LONG-TERM SAFETY,
TOLERABILITY, AND EFFICACY OF BIMEKIZUMAB IN ADULT
SUBJECTS WITH MODERATE TO SEVERE CHRONIC
PLAQUE PSORIASIS

PHASE 2B

EudraCT Number: 2016-001892-57

IND Number: 128707

Sponsor:

UCB Biopharma SPRL

Allée de la Recherche 60

B-1070 Brussels

**BELGIUM** 

| Protocol/Amendment number | Date | Type of amendment |
|---------------------------|-------------|-------------------|
| Final Protocol | 01 Jun 2016 | Not applicable |
| Protocol Amendment 1 | 12 Aug 2016 | Substantial |

## **Confidential Material**

## **Confidential**

This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB.


# STUDY CONTACT INFORMATION

## **Sponsor**

UCB Biopharma SPRL, Allée de la Recherche 60, B-1070 Brussels, Belgium

## **Sponsor Study Physician**

| Name: | |
|---|---|
| Address: | UCB BioPharma SPRL, Allée de la Recherche, 60, Brussels, Belgium, B-1070 |
| Phone: | Sign |
| Fax: | Tier. |

## **Clinical Project Manager**

| Name: | |
|---|---|
| Address: | UCB BioPharma SPRL, Allée de la Recherche, 60, Brussels, Belgium, B-1070 |
| Phone: | |
| Fax: | ALD istalling |

# Clinical Trial Biostatistician

| Name: | Nis. | |
|---|---|---|
| Address: | UCB Biosciences<br>27617 | , 8010 Arco Corporation Drive, Raleigh, NC |
| Phone: | | |
| Fax: | | |

# Clinical Monitoring Contract Research Organization

| Name: | PAREXEL International (IRL) Limited-Ireland |
|----------|-------------------------------------------------------------------|
| Address: | Ireland Limited at 70 Sir John Rogerson's Quay, Dublin 2, Ireland |
| Phone: | +353 (1) 477 3171 |
| Fax: | +353 (1) 477 3308 |


## **SERIOUS ADVERSE EVENT REPORTING**

| Fax |
|-------------|
| E 21 |
| Email Email |


# **TABLE OF CONTENTS**

| LIST OF ABBREVIATIONS | | 9 |
|---|---|---|
| 1 SUMMARY | | 12 |
| 2 INTRODUCTION | | 13 |
| 2.1 Psoriasis | | 13 |
| 2.1.1 Global epidemiology o | of psoriasis | 13 |
| | psoriasis | |
| 2.2 Bimekizumab | | <u>3</u> . 15 |
| 2.2.1 Clinical | | 15 |
| 2.2.2 Nonclinical | riables in service and army areas in the service and army areas in the service areas | 17 |
| 3 STUDY OBJECTIVES | ot in the second of the second | 17 |
| 3.1 Primary objective | | 17 |
| 3.2 Secondary objective | 200 | 17 |
| 3.3 Other objectives | Ø, | 17 |
| 4 STUDY VARIABLES | gijo' | 18 |
| 4.1 Safety variables | d dic | 18 |
| 4.1.1 Primary safety variable | · | 18 |
| 4.1.2 Other safety variables. | C ior | 18 |
| 4.2 Pharmacokinetic variable | | 18 |
| 4.3 Immunological variable | | 18 |
| 4.4 Efficacy variables | | 18 |
| 4.4.1 Secondary efficacy var | riables | 18 |
| 4.4.2 Other efficacy variable | 23/ <sub>11</sub> | 18 |
| 5 STUDY DESIGN | 801, | 19 |
| 5.1 Study description | | 19 |
| 5.1.1 Study duration per sub | ject | 20 |
| 5.1.2 Planned number of sub | pjects and sites | 20 |
| 5.1.3 Anticipated regions and | d countries | 20 |
| 5.2 Schedule of study assessments | 5 | 20 |
| 5.3 Schematic diagram | | 23 |
| | selection of dose | |
| 6 SELECTION AND WITHDR | AWAL OF SUBJECTS | 26 |
| 6 Inclusion criteria | | 26 |
| 6.3 Withdrawal criteria | | 27 |
| | ation criteria | |
| 7.1 Description of investigational | medicinal product | 30 |

| 7.2 | Treatments to be administered | 30 |
|---|---|---|
| 7.3 | Packaging | 30 |
| 7.4 | Labeling | 31 |
| 7.5 | Handling and storage requirements | 31 |
| 7.6 | Drug accountability | 31 |
| 7.7 | Procedures for monitoring subject compliance | 32 |
| 7.8 | Concomitant medication(s)/treatment(s). | 32 |
| 7 | 7.8.1 Permitted concomitant treatments (medications and therapies) | 32 |
| 7 | Prohibited concomitant treatments (medications and therapies) | 33 |
| 7.9 | Blinding. | 33 |
| 7 | Concomitant medication(s)/treatment(s). 8.1 Permitted concomitant treatments (medications and therapies). 8.2 Prohibited concomitant treatments (medications and therapies). Blinding. 9.1 Procedures for maintaining and breaking the treatment blind. 7.9.1.1 Maintenance of study treatment blind. 7.9.1.2 Breaking the treatment blind in an emergency situation. | 34 |
| | 7.9.1.1 Maintenance of study treatment blind | 34 |
| | 7.9.1.2 Breaking the treatment blind in an emergency situation | 34 |
| 7.10 | O Randomization and numbering of subjects | 35 |
| 8 | STUDY PROCEDURES BY VISIT | 35 |
| 8.1 | Baseline Visit | 35 |
| 8.2 | Week 4 (±3 days) | 36 |
| 8.3 | Week 8 (±3 days); Week 16 (±3 days); Week 32 (±3 days); and Week 40 (±3 days). | 37 |
| 8.4 | Week 12 (±3 days) | 38 |
| 8.5 | 7.9.1.2 Breaking the treatment blind in an emergency situation? Randomization and numbering of subjects STUDY PROCEDURES BY VISIT Baseline Visit Week 4 (±3 days) Week 8 (±3 days); Week 16 (±3 days); Week 32 (±3 days); and Week 40 (±3 days) Week 12 (±3 days) Week 20 (±3 days); Week 28 (±3 days); and Week 44 (±3 days) Week 24 (±3 days) Week 36 (±3 days) Week 48 (±3 days) Study Exit/Early Withdrawal SELL Visit (20 weeks after the last dose of bimekizumab or placebo: -3/±7 days) | 39 |
| 8.6 | Week 24 (±3 days) | 39 |
| 8.7 | Week 36 (±3 days) | 40 |
| 8.8 | Week 48 (±3 days) Study Exit/Early Withdrawal | 41 |
| 8.9 | SFU Visit (20 weeks after the last dose of bimekizumab or placebo; -3/+7 days) | 42 |
| 8.10 | O Early Withdrawal Visit | 42 |
| 8.11 | 1 Unscheduled Visit | |
| 9 | ASSESSMENT OF SAFETY | 43 |
| 9.1 | Adverse events. | 43 |
| | .1.1 Definition of AE | |
| 9 | 2.1.2 Procedures for reporting and recording AEs | 44 |
| 9 | 2.1.3 Description of AEs | 44 |
| 9 | 2.1.2 Procedures for reporting and recording AEs 2.1.3 Description of AEs 2.1.4 Follow up of AEs | 44 |
| .9 | 1.5 Rule for repetition of an AE | |
| ( <sup>©</sup> ) | Pregnancy Pregnancy | 44 |
| 9 | Suspected transmission of an infectious agent via a medicinal product | 45 |
| 9 | Overdose of investigational medicinal product | |
| 9 | 2.1.9 Safety signal detection | 46 |
| 9.2 | Serious adverse events | 46 |

| 9.2. | 1 Definition of SAE | 46 |
|---|---|---|
| 9.2.2 | 2 Procedures for reporting SAEs | 47 |
| 9.2.3 | Follow up of SAEs | 48 |
| 9.3 In | nmediate reporting of AEs | 48 |
| 9.4 A | nticipated SAEs | 48 |
| 9.5 A | dverse events of special interest | 48 |
| 9.6 A | dverse events for special monitoring | 49 |
| 9.7 L | aboratory measurements | 49 |
| 9.7. | Evaluation of PDILI | 50 |
| 9 | 9.7.1.1 Consultation with Medical Monitor and local hepatologist | 54 |
| 9 | 9.7.1.2 Immediate action: determination of IMP discontinuation | 54 |
| 9 | 9.7.1.3 Testing: identification/exclusion of alternative etiology | 54 |
| 9 | 9.7.1.4 Follow-up evaluation | 56 |
| 9.8 O | 9.7.1.4 Follow-up evaluation ther safety measurements | 56 |
| 9.8. | 1 Assessment and management of TB and TB risk factors | 56 |
| 9 | 9.8.1.1 TB assessment by IGRA | 58 |
| 9 | 9.8.1.2 Chest x-ray for TB. | 59 |
| 9 | 9.8.1.3 TB questionnaire | 59 |
| 9 | Assessment and management of TB and TB risk factors 9.8.1.1 TB assessment by IGRA 9.8.1.2 Chest x-ray for TB 9.8.1.3 TB questionnaire 9.8.1.4 TB management 2 Pregnancy testing 3 Vital signs 4 12-lead ECGs Physical examination 6 Assessment of suicidal bideation and behavior | 59 |
| 9.8.2 | Pregnancy testing Pregnancy testing | 60 |
| 9.8.3 | 3 Vital signs | 60 |
| 9.8.4 | 4 12-lead ECGs | 60 |
| 9.8. | 5 Physical examination | 60 |
| 9.8.0 | Assessment of suicidal ideation and behavior | 00 |
| 9.8. | 7 Data Monitoring Committee | 60 |
| | SSESSMENT OF PHARMACOKINETIC VARIABLES | |
| | SSESSMENT OF IMMUNOLOGICAL VARIABLES | |
| | SSESSMENT OF EFFICACY | |
| | soriasis Area and Severity Index | |
| | vestigator's Global Assessment | |
| | ermatology Life Quality Index | |
| | SA affected by psoriasis | |
| | Iodified Nail Psoriasis Severity Index | |
| | soriasis Scalp Severity Index | |
| | GADA for the arthritis VAS | |
| | 6-Item Short Form Health Survey | |
| | ospital Anxiety and Depression Scale | |
| 12 C' | THOV MANAGEMENT AND ADMINISTRATION | 65 |

| 13.1 Adherence to protocol | 65 |
|---|---|
| 13.2 Monitoring | 65 |
| 13.2.1 Definition of source data | 66 |
| 13.2.2 Source data verification | 66 |
| 13.3 Data handling | 66 |
| 13.3.1 eCRF completion | 66 |
| 13.3.2 Database entry and reconciliation | 67.0 |
| 13.3.3 Subject Enrollment log/Subject Identification Code list | 67 |
| 13.4 Termination of the study | 67 |
| 13.5 Archiving and data retention | |
| 13.6 Audit and inspection | <u>Ø</u> 68 |
| 13.7 Good Clinical Practices | 68 |
| 14 STATISTICS | 68 |
| 14.1 Definition of analysis sets | 68 |
| 14.2 General statistical considerations | 69 |
| 14.3 Planned safety analyses | 70 |
| 14.3.1 Primary safety analysis | 70 |
| 14.3.2 Other safety analyses | 71 |
| 14.4 Planned PK analyses | 71 |
| 13.3.2 Database entry and reconciliation 13.3.3 Subject Enrollment log/Subject Identification Code list 13.4 Termination of the study 13.5 Archiving and data retention 13.6 Audit and inspection 13.7 Good Clinical Practices 14 STATISTICS 14.1 Definition of analysis sets 14.2 General statistical considerations 14.3 Planned safety analyses 14.3.1 Primary safety analysis 14.3.2 Other safety analyses 14.4 Planned PK analyses 14.5 Planned immunological analyses 14.6 Planned efficacy analyses 14.7 Planned interim analysis and data monitoring | 71 |
| 14.6 Planned efficacy analyses | 71 |
| 14.7 Planned interim analysis and data monitoring | 72 |
| 14.8 Determination of sample size | 72 |
| 15 ETHICS AND REGULATORY REQUIREMENTS | 72 |
| 15.1 Informed consent | 72 |
| 15.2 Subject identification cards | 73 |
| 15.3 IRBs and IECs | 73 |
| 15.4 Subject privacy | 74 |
| 15.5 Protocol amendments | 74 |
| 16 FINANCE, INSURANCE, AND PUBLICATION | |
| 17 REFERENCES | |
| 18 APPENDICES | 77 |
| 18 APPENDICES | 77 |
| DECLARATION AND SIGNATURE OF INVESTIGATOR | 124 |
| 20 SPONSOR DECLARATION | |
| LIST OF TABLES | |
| Table 5–1: Schedule of study assessments | 21 |
| | <del>-</del> |

| Prohibited psoriasis medications during PS0011 | 33 |
|---|---|
| Anticipated SAEs for the population of subjects with moderate to severe chronic plaque psoriasis. | 48 |
| Laboratory measurements | 49 |
| Required investigations and follow-up for PDILI | 52 |
| PDILI laboratory measurements | 55 |
| PDILI information to be collected | 56 |
| Body areas for calculation of percent BSA for PASI | 62 |
| Parameters assessed for the PSSI. | 64 |
| LIST OF FIGURES | |
| Schematic diagram | 24 |
| ort any marketing | |
| | Prohibited psoriasis medications during PS0011 Anticipated SAEs for the population of subjects with moderate to severe chronic plaque psoriasis. Laboratory measurements Required investigations and follow-up for PDILI PDILI laboratory measurements PDILI information to be collected Body areas for calculation of percent BSA for PASI Parameters assessed for the PSSI LIST OF FIGURES Schematic diagram LIST OF FIGURES Schematic diagram LIST OF FIGURES Schematic diagram |


## LIST OF ABBREVIATIONS

AE adverse event

**AESM** 

**ALP** 

**ALT AST** 

**BSA** 

cAMP **CRO** 

**CTCAE** 

**DLOI** 

Contract Research Organization
Common Terminology Criteria for Adverse Events
Dermatology Life Quality Index
Data Monitoring Committee
exposure adjusted event rate
exposure adjusted incidence rate
electrocardiogram
electronic Case Report Form
electronic Columbia-Suicide Seelectronic data capture. **DMC EAER** 

**EAIR** 

ECG

**eCRF** 

eC-SSRS

**EDC** Full Analysis Set **FAS** 

Food and Drug Administration **FDA** 

Good Clinical Practice **GCP** 

gastrointestinal GI

Good Manufacturing Practice **GMP** 

Hospital Anxiety and Depression Scale **HADS** 

**HADS-A** Hospital Anxiety and Depression Scale-Anxiety Hospital Anxiety and Depression Scale-Depression HADS-D

high level term

Investigator's Brochure

International Council for Harmonisation

**Independent Ethics Committee** 

Investigator's Global Assessment

**IGRA** interferon gamma release assay ILinterleukin

**IMP** investigational medicinal product(s)

**IRB** 

iv

**IXRS** 

LTB mAb

**MCS** 

... Index
... imatory drug
... iny Index
... mNAPSI

**NSAID** 

**NTMB** 

**PASI** 

**PCS** 

PDE4

**PDILI** 

**PGADA** 

PK

**PK-PPS** 

**PRO** 

Patient Safet PS

**PSSI** Psoriasis Scalp Severity Index

PT preferred term every 4 weeks Q4W quality of life

serious adverse event

subcutaneous(ly)

36-Item Short Form Health Survey

Safety Follow-Up system organ class

Standard Operating Procedure

Safety Set tuberculosis TB

| TEAE | treatment-emergent adverse event |
|------|----------------------------------|

| TNF | tumor necrosis factor |
|-----|-----------------------|
| ULN | upper limit of normal |
| VAS | vicual analog coale |

The document control the used to support any treated in a superior of the use of the support of the use of the support of the used to support on the use of the use o


### 1 SUMMARY

PS0011 is a multicenter, 48-week, double-blind, placebo-controlled, parallel-group extension

During the Treatment Period, subjects will attend study visits at the study site every 4 weeks (Q4W) for study assessments and administration of bimekizumab or placebo by study site at a County through Week 48. Any subject who does not achieve a Psoriasis Area and County Week 12 or later in PS0011 will be a controlled by the decounty of the Early Withdree. the Early Withdrawal Visit assessments. Following completion or early withdrawal from the 48-week Treatment Period, subjects will return for a Safety Follow-Up (SFU) Visit 20 weeks after their last dose of bimekizumab or placebo in PS0011.

Subjects withdrawing early from the study will undergo the Early Withdrawal Visit assessments and will enter the SFU Period.

Subjects who received placebo or bimekizumab 64mg, 160mg, or 320mg loading dose + 160mg Q4W in PS0010 must achieve PASI90 response at Week 12 in PS0010 to enter the PS0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving placebo or bimekizumab 64mg Q4W will be assigned to receive bimekizumab 160mg Q4W on entering PS0011. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving bimekizumab 160mg or 320mg loading dose + 160mg Q4W will be assigned to receive bimekizumab 320mg Q4W on entering PS0011. Subjects who receive bimekizumab 320mg or 480mg Q4W in PS0010 will be assigned to receive bimekizumab 320mg Q4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010.

Up to 240 subjects are anticipated to enroll in PS0011 at approximately 40 sites in Europe, Canada, and the US, with possible extension to other regions and countries as required in PS0010.

The primary objective of the study is to assess the long-term safety and tolerability of bimekizumab. The secondary objective of the study is to assess the efficacy of bimekizumab administered Q4W over 48 weeks. The other objectives of the study are to assess the pharmacokinetics (PK) and immunogenicity of bimekizumab.

The primary safety variable is the incidence of treatment-emergent adverse events (TEAEs) adjusted by duration of subject exposure to treatment. The other safety variables are change from Baseline of PS0010 and PS0011 in clinical laboratory values (chemistry, hematology, and urinalysis), vital signs, physical examination, and 12-lead electrocardiogram (ECG) results.

The PK variable is plasma concentrations of bimekizumab and the immunological variable is anti-bimekizumab antibody levels prior to and following study treatment.

The efficacy assessments are PASI, Investigator's Global Assessment (IGA) Dermatology Life Quality Index (DLQI), body surface area (BSA) affected by psoriasis, modified Nail Psoriasis Valiations thereof. Severity Index (mNAPSI) score, Psoriasis Scalp Severity Index (PSSI), Patient's Global Assessment of Disease Activity (PGADA), 36-item Short Form Health Survey (SF-36), and the Hospital Anxiety and Depression Scale (HADS); a list of the secondary and other efficacy variables is presented in Section 4.4.

### 2 INTRODUCTION

### 2.1 **Psoriasis**

Psoriasis is a common, chronic inflammatory disease characterized by a series of linked cellular changes in the skin: hyperplasia of epidermal keratinocytes, vascular hyperplasia and ectasia, and infiltration of T lymphocytes, neutrophils, and other types of leukocytes in affected skin. Though the pathophysiology of psoriasis is not fully understood, the importance of T-cells and inflammatory cytokines has been demonstrated by the clinical benefit provided by therapies directed at these targets (Krueger and Ellis, 2005).

There are a variety of forms including plaque, guttate, inverse, pustular, and erythrodermic. Plaque psoriasis is the most common, comprising approximately 80% to 90% of all cases. Approximately 17% of those with psoriasis have moderate to severe disease (Kurd et al., 2008).

In addition to the impact on skin, psoriasis has a multitude of psychosocial and emotional effects on patients, including increased self-consciousness, frustration, fatigue, depression, and suicidal ideation. As a result, patients frequently report sleeping problems, difficulties at work, problems interacting with family members, disrupted leisure activities, and sexual difficulties (Dowlatshahi et al, 2014; Gottlieb, 2005; Mukhtar et al, 2004; Ortonne, 2004; Krueger et al. 2001).

A number of comorbidities have been associated with psoriasis, especially with more severe psoriasis. Psoriatic arthritis, cardiovascular disease, metabolic syndrome, chronic pulmonary disease, peptic ulcer disease, renal disease, and diabetes have all been demonstrated to have an increased prevalence in psoriasis patients (Yeung et al., 2013; Christophers et al., 2010; Gisondi et al, 2007; Gelfand et al, 2006).

### 2.1.1 Global epidemiology of psoriasis

Psoriasis affects approximately 3% of the adult US population (Rachakonda et al., 2014; Kurd and Gelfand, 2009) and its onset can begin at any age (Augustin et al, 2010; Icen et al. 2009). The reported worldwide incidence and prevalence of psoriasis varies greatly depending on age, gender, ethnicity, and geography primarily due to genetic and environmental factors. Estimates of incidence and prevalence include all types of psoriasis. Plaque psoriasis is the most common form of psoriasis therefore reported estimates of the magnitude of this condition are likely weighted heavily by this subtype. Both the incidence and prevalence of psoriasis are higher among Caucasians and those living in higher latitudes. Psoriasis affects approximately 2% to 4% of the population of western countries. Geographical differences are also influenced by case definition, study design, and the definition of prevalence (Parisi et al, 2013; Langley et al, 2005; Raychaudhuri and Gross, 2000).

## 2.1.2 Current treatments for psoriasis

Therapy for patients with psoriasis varies according to the severity of disease. Limited or mild disease is often treated with topical therapies such as corticosteroids and vitamin D analogs. Patients with more severe disease are often treated with chemophototherapy, methotrexate, the oral phosphodiesterase 4 (PDE4) inhibitor (apremilast), or biologic agents, such as tumor necrosis factor (TNF) antagonists, interleukin (IL) 12/23 inhibitors, and IL-17A inhibitors. The effectiveness of TNF inhibitors in the treatment of psoriasis has been demonstrated in many Phase 3 clinical studies and has led to the approval of multiple TNF inhibitors for use in patients with moderate to severe psoriasis. Interleukin inhibitors include secukinumab and ixekizumab, IL-17A inhibitors approved for treatment of moderate to severe psoriasis. Ustekinumab is an IL-12/23 antagonist approved for use in patients with moderate to severe psoriasis, and brodalumab, an IL-17 receptor antagonist, has completed pivotal Phase 3 studies in psoriasis. Standard therapies for psoriasis are listed below:

- Topical steroids (eg, triamcinolone, mometasone, clobetasol, betamethasone, hydrocortisone) are generally used as first-line treatment of psoriasis. High-strength steroids are typically reserved for use on the arms and legs. Areas such as the face and skin folds (axillary, inguinal regions, etc) are usually treated with a low potency steroid. Chronic use of topical steroids can lead to corticosteroid-related side effects and is generally discouraged.
- Vitamin D analogs (eg, calcipotriol and tacalcito) are commonly used to treat mild to moderate psoriasis, and work best within the mild patients. They are safe but lack efficacy for many moderate to severe patients.
- Chemophototherapy is a frequent option for moderate to severe patients, but the inconvenience of multiple treatment visits and varying efficacy limits its use in the market.
- Methotrexate is a systemic immunosuppressant and is used in moderate to severe patients. Toxicity concerns, particularly in older patients, are a major drawback.
- Apremilast is an oral small-molecule inhibitor of PDE4 that is also approved for treatment of adults with moderate to severe plaque psoriasis. Phosphodiesterase 4 inhibitors work intracellularly to modulate a network of pro-inflammatory and anti-inflammatory mediators. Phosphodiesterase 4 is a cyclic adenosine monophosphate (cAMP)-specific PDE and the dominant PDE in inflammatory cells. Phosphodiesterase 4 inhibition elevates intracellular cAMP levels, which in turn down-regulates the inflammatory response by modulating the expression of TNFα, IL-23, IL-17, and other inflammatory cytokines.
- Biologics, including TNFα inhibitors (adalimumab, etanercept, and infliximab), IL-12/23 inhibitors (ustekinumab), and IL-17A inhibitors are the treatment options of choice for patients with moderate to severe plaque psoriasis who are candidates for systemic therapy or phototherapy. These products are injected sc or delivered via intravenous (iv) infusion and while effective, TNFα inhibitors come with boxed warnings including the risk of serious infections and reports of lymphoma and malignancy in children and adolescent patients. The efficacy of TNFα inhibitors in treating psoriasis has been attributed to their inhibition of Th17-T cells. Different from the traditional systemic drugs that impact the entire immune system, biologics target specific parts of the immune system and offer reduced multi-organ toxicity and adverse effects associated with traditional treatments.

Secukinumab has been approved in the US and the EU for the treatment of moderate to severe plaque psoriasis in adult patients who are candidates for systemic therapy or phototherapy. Secukinumab is a monoclonal antibody (mAb) that inhibits the activity of the

Bimekizumab (also known as UCB4940) is an engineered, humanized, full-length immunoglobulin G1 mAb with high affinity for human IL-17A and IL-17F, important proinflammatory cytokines of the IL-17 family believed to play important roles in autoiman and inflammatory diseases. Interleukin-17A has been shown to have a role several autoimmune disorders and IL-17F has been increasing bathogenesis of a number of inflammatory distance. antibodies have demonstrated efficacy in patients with psoriasis, psoriatic arthritis, and ankylosing spondylitis, as yet, no therapeutic approach is available that fully inhibits the activity of IL-17F. Bimekizumab selectively and potently inhibits the activity of both IL-17A and IL-17F isoforms in vitro. Therefore, it permits an evaluation of the potential for additional efficacy, that may be conferred by dual inhibition of both cytokines, in patients suffering from diseases in

which both cytokines are active.

2.2.1 Clinical

Three clinical studies of bimekizumab have been completed: UP0008 in 39 subjects with mild to moderate plaque psoriasis, RA0124 in 30 healthy volunteers, and PA0007 in 53 subjects with psoriatic arthritis. Two studies (RA0123 and UP0031) are ongoing in subjects with moderate to severe rheumatoid arthritis and in healthy subjects, respectively.

UP0008 was a Phase 1, single ascending dose study in adults with mild to moderate psoriasis affecting ≤5% BSA. In this blinded study, single doses of up to 640mg (approximately 8mg/kg in an 80kg adult) were evaluated without any safety concerns. A total of 26 subjects with psoriasis with less than 5% of body surface involvement were treated with a range of single iv doses from 8 to 640mg. There were no clinically relevant safety findings identified at any dose and all doses were well tolerated. The pre-specified exploratory assessment of disease activity showed clinically relevant and statistically significant improvements at the higher doses studied.

RA0124 was a Phase 1, open-label, parallel-group, single-dose study in healthy subjects. The primary objective of this study was to determine the absolute bioavailability of single sc doses of proportionality of bimekizumab 80mg and 160mg sc, and to evaluate the safety and tolerability of these sc doses and 160mg given by iv infusion. In RA0124, the absolute bioavailability was similar for the 2 doses tested (0.656 and 0.631 for the bimekizumab 80mg and 160mg sc.) respectively). The PK of bimekizumab was linear in 41 following so admiproportionality of bimekizumab 80mg and 160mg sc, and to evaluate the safety and tolerability similar for the 2 doses tested (0.656 and 0.631 for the bimekizumab 80mg and 160mg sc doses, following sc administration was similar to that following iv administration (27.81 days and 28.25 days for bimekizumab 160mg sc and 160mg iv, respectively).

Bimekizumab has also been investigated in a Phase 1b, proof of concept, randomized, placebo-controlled, multiple dose study (PA0007). The primary objective of PA0007 was to attensions or variations thereof. assess the safety and PK of multiple dose administration of iv bimekizumab in subjects with psoriatic arthritis. Four active doses and a placebo were tested. Drug was administered as a loading dose at Week 0, and 2 additional doses were administered at Week 3 and Week 6. In each treatment group, subjects received a total of 3 doses of bimekizumab, administered every 3 weeks as shown below:

- 80mg loading dose followed by 40mg at Weeks 3 and 6
- 160mg loading dose followed by 80mg at Weeks 3 and 6
- 240mg loading dose followed by 160 mg at Weeks 3 and 6
- 560mg loading dose followed by 320mg at Weeks 3 and 6

The results of this study demonstrated that all doses of bimekizumab were well tolerated and there were no unexpected clinically relevant safety findings.

Infections (mostly nasopharyngitis) were the most commonly reported events in both the active treatment and the placebo group. None of the infections were considered serious or required treatment with antibiotics. Two subjects in the active treatment group experienced 1 local candida infection each (oropharhyngitis and vulvovaginitis, respectively) that were nonserious and resolved with topical therapy. There was a reduction in mean neutrophil count in the active treatment group, although this drop was not clinically relevant and a clear relationship with dose or time was not evident. Some increases in liver function tests were reported, but none had a convincing relationship to exposure to study medication. The exploratory analysis showed clinically relevant improvement in activity of psoriatic arthritis and in skin involvement in those subjects with concomitant active psoriatic lesions.

Two additional studies of bimekizumab are ongoing. RA0123 is a Phase 2a, double-blind, randomized, placebo-controlled, multiple dose study to evaluate the safety, PK, pharmacodynamics, and efficacy of multiple doses of bimekizumab administered as add-on therapy to stable certolizumab pegol therapy in subjects with moderate to severe rheumatoid arthritis. UP0031 is a Phase I open-label, parallel-group, single-dose study to evaluate the relative bioavailability and tolerability of bimekizumab 160mg sc in healthy subjects.

Additional information on the clinical data for bimekizumab is available in the current version of the Investigator's Brochure (IB).

The current study, PS0011, is a 48-week extension study for eligible subjects who complete PS0010, a Phase 2b, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study in adult subjects with moderate to severe chronic plaque psoriasis. In PS0010, subjects will be randomized 1:1:1:1:1 to receive the following blinded study treatment regimens for a treatment period of 12 weeks:

- Bimekizumab 64mg administered sc Q4W
- Bimekizumab 160mg administered sc Q4W
- Bimekizumab 320mg loading dose administered sc at Baseline followed by 160mg dose administered sc Q4W.

- Bimekizumab 320mg administered sc Q4W
- Bimekizumab 480mg administered sc Q4W

Parallel inhibition of IL-17A and IL-17F has been shown to be efficacious in a variety of animal models of inflammatory disease. Intravenously administered bimekizumab was well tolerated intravenously studies in Cynomolgus monkeys with of 200mg/kg/weel. The first intravenously administered bimekizumab was well tolerated in the first intravenously administered bimekizumab was well ad of 200mg/kg/week. The findings of note in toxicity studies were diarrhea related to infectious enteritis (observed in the single dose study) and asymptomatic mild colonic ulceration in a proportion of animals (in the repeat dose study); this latter finding was not associated with hematology abnormalities. Data suggest that bimekizumab has induced primary lesions to the mucosa-associated lymphoid tissue via a pharmacologically-related mechanism. In a second repeat-dose study, none of the minor apoptosis/necrosis findings observed in gut associated lymph nodes were revealed. In animals given the highest dose of bimekizumab in the study (20mg/kg/week), a slightly higher number of protozoa (Balantidium coli) was observed in the cecum and colon as compared to the control animals and low dose animals. Therefore gut associated lymph node lesions observed in the first study are considered to be accidental and/or linked to exaggerated pharmacology and proliferation of *Balantidium coli* and is considered the consequence of a change in local mucosal immunity. To date, similar findings have not been seen in studies in humans.

Additional information on the nonclinical data for bimekizumab is available in the current version of the IB.

## STUDY OBJECTIVES 3

## Primary objective 3.1

The primary objective of the study is to assess the long-term safety and tolerability of bimekizumab.

## Secondary objective 3.2

The secondary objective of the study is to assess the efficacy of bimekizumab administered Q4W over 48 weeks.

## 3.3 Other objectives

The other objectives of the study are:

- PK of bimekizumab

   To assess the immunogenicity of bimekizumab

### 4 STUDY VARIABLES

### 4.1 Safety variables

### 4.1.1 Primary safety variable

The primary safety variable is the incidence of TEAEs adjusted by duration of subject exposure to treatment.

### 4.1.2 Other safety variables

Change from Baseline variables will be defined relative to the Baseline measurements from both PS0010 and PS0011.

The other safety variables are:

- Change from Baseline in clinical laboratory values (chemistry, hematology, and urinalysis)
- Change from Baseline in vital signs
- Change from Baseline in physical examination
- Change from Baseline in 12-lead ECG results

### 4.2 Pharmacokinetic variable

The PK variable is plasma concentrations of bimekizumab.

### 4.3 Immunological variable

The immunological variable is anti-bimekizumab antibody levels prior to and following study treatment.

## 4.4 Efficacy variables

Change from Baseline variables will be defined relative to the Baseline measurements from both PS0010 and PS0011.

## 4.4.1 Secondary efficacy variables

The secondary efficacy variables are:

- PASI90 response over time
- IGA response Clear or Almost Clear with at least a 2 category improvement from Baseline on a 5-point scale) over time

# Other efficacy variables

The efficacy variables are listed below and will be evaluated at all scheduled visits in accordance with the schedule of assessments in Table 5–1.

PASI75 and PASI100 response

- Absolute and percent change from Baseline in PASI score
- Shift from Baseline in IGA score
- Change from Baseline in DLQI

- Percent of subjects achieving a DLQI score of 0 or 1
- Absolute and percent change from Baseline in the BSA affected by psoriasis

- Change from Baseline in the PGADA for the arthritis visual analog scale (VAS)

  Change from Baseline in SF-36 Physical Component Summary (PCS) score, Mental Component Summary (MCS) score, and individual domains

  Change from Baseline in the HADS Anxiety (HADS-A) and Development Summary (PCS) scores with scores below of scores.

### 5 STUDY DESIGN

### 5.1 Study description

PS0011 is a multicenter, 48-week, double-blind, placebo-controlled, parallel-group, extension study to assess the long-term safety, tolerability, and efficacy of bimekizumab in eligible adult subjects with moderate to severe chronic plaque psoriasis who complete PS0010. At Week 12 of PS0010, all eligible subjects continuing into PS0011 will undergo the PS0010 Week 12 study assessments and any additional PS0011 Baseline assessments, and will then receive their first dose of bimekizumab or placebo in PS0011.

During the Treatment Period, subjects will attend study visits at the study site Q4W for study assessments and administration of bimekizumab or placebo by study site staff through Week 48. Any subject who does not achieve PASI75 response at Week 12 or later in PS0011 will be withdrawn from study treatment and will return to complete the Early Withdrawal Visit assessments. Following completion or early withdrawal from the 48-week Treatment Period, subjects will return for a SFU Visit 20 weeks after their last dose of bimekizumab or placebo in PS0011.

Subjects withdrawing early from the study will undergo the Early Withdrawal Visit assessments and will enter the SFU Period.

Subjects who received placebo or bimekizumab 64mg, 160mg, or 320mg loading dose + 160mg O4W in P\$0010 must achieve PASI90 response at Week 12 in P\$0010 to enter the P\$0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving placebo or bimekizumab 64mg Q4W will be assigned to receive bimekizumab 160mg Q4W on entering PS0011. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving bimekizumab 160mg or 320mg loading dose + 160mg Q4W will be assigned to receive bimekizumab 320mg Q4W on entering PS0011. Subjects who receive bimekizumab 320mg or 480mg Q4W in PS0010 will be assigned to receive bimekizumab 320mg O4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010.

A schedule of study assessments in presented in Table 5–1.

presented in

Jubject

is estimated to be up

weeks

At the last dose of bimekizumab.

Afined as the date of the last visit of the last vi Dep to a maximum of 64 weeks:

Dep to a maximum of 64 weeks:

Dep to weeks

Dep to a maximum of 64 weeks:

Dep to 240 weeks after the last dose of bimekizumab or placebo

The end of the study is defined as the date of the last visit of the last subject in the study. The study of the study The regions planned for study conduct are Europe, Canada, and the US, with possible extension

| UCB<br>Clinical Study Protocol | | | В | simekiz | umab | | | | | | | | Street 12 A | •<br>Aug 2016<br>PS0011 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 5–1: Schedule of study assessments | | | | | | | | | | | | | | |
| Visit Week <sup>a</sup> | PS0011 | Treatment Period | | | | | | | | | | | | |
| | Baseline | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Wk | Wk. | -Wk | Wk | Wk 48/ | |
| Protocol activity | | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 360 | 40 | 44 | WD | SFU <sup>b</sup> |
| Informed consent | X <sup>c</sup> | | | | | | | | T. | S), | | | | |
| Inclusion/exclusion | X d | | | | | | | | 70, | | | | | |
| Physical exam <sup>e</sup> | X <sup>f</sup> | | | | | | | > ? | <i>C</i> , | | | | X | X |
| Body weight | X <sup>f</sup> | | | | | | | SUC | | | | | X | X |
| Vital signs <sup>g</sup> | X <sup>f</sup> | X | X | X | X | X | XO | X | X | X | X | X | X | X |
| Hematology/biochemistry | X <sup>f</sup> | X | X | X | X | X | cX | X | X | X | X | X | X | X |
| Urinalysis | $X^{f}$ | | | X | 07 | 200 | X | | | X | | | X | X |
| 12-lead ECG | X <sup>f</sup> | | | | .0` | 6.0 | X | | | | | | X | X |
| Pregnancy testing h | X <sup>f</sup> | X | X | $\langle \hat{\mathbf{X}} \rangle$ | 1X | X | X | X | X | X | X | X | X | X |
| eC-SSRS | X <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| IGRA TB test i | j | | 10P | aliti | | | | | | | | | X | |
| TB questionnaire | X <sup>f</sup> | < | 2000 | X | | | X | | | X | | | X | |
| Blood sample for bimekizumab plasma concentrations k | X <sup>f</sup> | X | ŁŠX | X | X | | | X | | | X | | X | X |
| Blood sample for anti-bimekizumab antibodies <sup>k</sup> | X f | NX | X | X | X | | | X | | | X | | X | X |
| PASI | XQ | X | X | X | X | X | X | X | X | X | X | X | X | X |
| IGA | cuX <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| DLQI | X f | X | | X | | | X | | | X | | | X | |
| BSA | X <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | |
| mNAPSI | X <sup>f</sup> | X | | X | | | X | | | X | | | X | |
| PSSI | X <sup>f</sup> | X | | X | | | X | | | X | | | X | |
| PGADA | X <sup>f</sup> | | | X | | | X | | | X | | | X | |
| SF-36 | X <sup>f</sup> | | | X | | | X | | | X | | | X | |

| Table 5–1: Schedule of study assessmen | ts |
|----------------------------------------|----|
|----------------------------------------|----|

| Visit Week <sup>a</sup> | DGGGG | Treatment Period | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | PS0011<br>Baseline | Wk<br>4 | Wk<br>8 | Wk<br>12 | Wk<br>16 | Wk<br>20 | Wk<br>24 | Wk<br>28 | Wk<br>32 | Wk<br>36 | Wk<br>40 | Wk<br>44 | Wk 48/<br>WD | SFU <sup>b</sup> |
| HADS | X <sup>f</sup> | X | X | X | X | X | X | X | X | SX | X | X | X | X |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | ΧΩ | X | X | X | X | X | X <sup>1</sup> |
| IXRS | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Bimekizumab administration m | X | X | X | X m | X m | X m | X m | X m | X m | X m | X m | X m | | |

BSA=body surface area; DLQI=Dermatology Life Quality Index; ECG=electrocardiogram; eC-SSRS=electronic Columbia-Suicide Severity Rating Scale; HADS=Hospital Anxiety and Depression Scale; IGA=Investigator's Global Assessment; IGRA=interferon gamma release assay; IXRS=interactive voice or web response system; mNAPSI=modified Nail Psoriasis Severity Index; PASI=Psoriasis Area and Severity Index; PGADA=Patient's Global Assessment of Disease Activity; PSSI=Psoriasis Scalp Severity Index; Q4W=every 4 weeks; SF-36=36-item Short Form Health Survey; SFU=Safety Follow-Up; TB=tuberculosis; WD=withdrawal; Wk=week

<sup>&</sup>lt;sup>a</sup> Visit windows of ±3 days from the first dose (Baseline) at all visits except SFU, which has a window of -3 and +7 days from scheduled visit date.

<sup>&</sup>lt;sup>b</sup> The SFU Visit will occur 20 weeks after the last dose of bimekizumab of placebo.

<sup>&</sup>lt;sup>c</sup> Ensure that the informed consent for PS0011 was completed by the subject during the Week 8 or Week 12 Visit of PS0010 (must be done before any study assessments are performed for PS0011).

<sup>&</sup>lt;sup>d</sup> To be performed prior to the first dose of bimekizumab or placebo in PS0011.

<sup>&</sup>lt;sup>e</sup> Includes evaluation of signs and symptoms of active TB and risk for exposure to TB.

The noted PS0011 Baseline assessments will be obtained at the Week 12 Visit of PS0010 and do not need to be recorded on the case report form for this study.

g Vital signs (blood pressure, pulse rate, and temperature) are to be measured prior to blood sampling and prior to dosing, where applicable.

<sup>&</sup>lt;sup>h</sup> Pregnancy testing will be urine testing at all visits except SFD, which will be a serum test.

<sup>&</sup>lt;sup>1</sup> It is recommended that the QuantiFERON TB GOLD test be performed.

Ensure that an IGRA test was performed during the Week 8 Visit of PS0010 and the result was negative.

<sup>&</sup>lt;sup>k</sup> All blood samples are to be taken prior to dosing.

<sup>&</sup>lt;sup>1</sup> Including assessment for the development of different forms of psoriasis at the SFU visit.

m Subjects who received placebo or bimekizumab 64mg, 160mg, or 320mg loading dose + 160mg Q4W in PS0010 must achieve PASI90 response at Week 12 in PS0010 to enter the PS0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving placebo or bimekizumab 64mg will be assigned to receive bimekizumab 160mg on entering PS0011. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving bimekizumab 160mg or 320mg loading dose + 160mg will be assigned to receive bimekizumab 320mg Q4W on entering PS0011. Subjects who receive bimekizumab 320mg or 480mg Q4W in PS0010 will be assigned to receive bimekizumab 320mg Q4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010. Any subject who does not achieve PASI75 response at Week 12 or later in PS0011 will be withdrawn from study treatment and will return to complete the Early Withdrawal Visit assessments.

The document control he used to support any materials altroided to support any materials and the use of the support any materials altroided to support altroided to support any materials altroided to support altroided to suppor


Figure 5-1: Schematic diagram



PASI=Psoriasis Area and Severity Index; Q4W=every 4 weeks; SFU=Safety Follow-Up

Confidential Chie

<sup>&</sup>lt;sup>a</sup> Subjects who received placebo or bimekizumab 64mg, 160mg, or 320mg loading dose + 160mg Q4W in PS0010 must achieve PASI90 response at Week 12 in PS0010 to enter the PS0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving

placebo or bimekizumab 64mg will be assigned to receive bimekizumab 160mg on entering PS0011. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving bimekizumab 160mg or 320mg loading dose + 160mg will be assigned to receive bimekizumab 320mg Q4W on entering PS0011.

b Subjects who receive bimekizumab 320mg or 480mg Q4W in PS0010 will be assigned to receive bimekizumab 320mg Q4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010.

<sup>c</sup> Any subject who does not achieve PASI75 response at Week 12 or later in PS0011 will be withdrawn from study treatment and will return to complete the Early Withdrawal Visit assessments.


## 5.4 Rationale for study design and selection of dose

PS0011 is a 48-week, double-blind, placebo-controlled, parallel-group extension study for eligible subjects who complete PS0010, a Phase 2b, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study in adult subjects with moderate to severe chronic plaque psoriasis. Because some PS0010 subjects may have severe disease, the treatment in PS0011 provides more time to respond to a potentially efficacious treatment. PS0011 also provides an opportunity for nonresponding PS0010 placebo subjects to receive bimekizumab This study will allow the collection of further data on the long-term safety, tolerability, and efficacy of bimekizumab in this subject population.

The PS0011 design (Figure 5–1) allows PASI90 responders in PS0010 to continue their dose in PS0011, thus permitting these subjects to remain on the dose that resulted in this response after 12 weeks of initial treatment in PS0010. It also provides an opportunity for an increased dose among PS0010 nonresponders (ie, <PASI90). PASI90 was selected as the response criterion in PS0010 to ensure that a sufficiently high efficacy response was achieved. This type of dose escalation for those who do not achieve a desired response after 12 weeks is common in clinical practice.

Regardless of PASI90 response at Week 12 of PS0010, subjects who received the 2 highest doses of bimekizumab (320mg and 480mg Q4W) in PS0010 will begin PS0011 on the 320mg Q4W dose. For those subjects who do achieve PASI90 response, this will allow a continuation of the PS0010 dose for subjects initially receiving 320mg Q4W and a dose down for subjects originally randomized to the 480mg Q4W dose. Because bimekizumab 480mg Q4W is the highest dose evaluated in PS0010 and because it requires 3 injections, it will be of interest to evaluate whether these subjects can maintain response in PS0011 with the lower 320mg dose. allowing the blind to be maintained with the use of only 2 injections at each study administration visit.

To protect against the possibility of exposing subjects to an ineffective treatment for extended periods of time, subjects across all treatment groups who have not achieved PASI75 response at Week 12 or later in PS0011 will be withdrawn from study treatment. Because this withdrawal decision is based strictly on the PASI response and not on the original study treatment, it can be done in such a way that will not unblind subjects or Investigators.

## **SELECTION AND WITHDRAWAL OF SUBJECTS** 6

## 6.1

To be eligible to participate in this study, all of the following criteria must be met:

- Informed Consent form is signed and dated by the subject.

  2. Subject is considered. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written
- Subject is considered reliable and capable of adhering to the protocol and visit schedule according to the judgment of the Investigator.
- 3. Subject completes all dosing requirements in PS0010 without meeting any withdrawal criteria and completes the study.

4. Female subjects of childbearing potential and male subjects with a partner of childbearing potential must continue to use an acceptable method of contraception (as detailed in PS0010) itations thereof for up to 20 weeks after the last dose of study treatment in PS0011.

### 6.2 **Exclusion criteria**

Subjects are not permitted to enroll in the study if any of the following criteria are met:

- 1. Subject has previously participated in this study.
- 2. Female subjects who plan to become pregnant during the study or within 20 weeks following last dose of study medication. Male subjects who are planning a partner pregnancy during the study or within 20 weeks following the last dose.
- 3. Subject has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study. Note: For any subject with an ongoing serious adverse event (SAE), or a history of serious infections (including herpes zoster or hospitalizations) in PS0010, the Medical Monitor must be consulted prior to the subject's entry into PS0011.
- 4. Subject must have a negative interferon gamma release assay (IGRA) as measured at Week 8 of PS0010.
- 5. Any subject who meets any withdrawal criteria in the feeder study (PS0010) is excluded from participating in the extension study (PS0011).

### 6.3 Withdrawal criteria

Subjects are free to withdraw from the study at any time, without prejudice to their continued care.

Subjects should be withdrawn from the study and will be asked to complete the Early Withdrawal Visit and SFU Visit (20 weeks after the last received dose) if any of the following events occur:

- 1. Subject withdraws his/her consent.
- 2. There is confirmation of a pregnancy in a female subject during the study, as evidenced by a positive pregnancy test.
- 3. The Sponsor or a regulatory agency requests withdrawal of the subject.
- 4. Subject develops an illness that in the opinion of the Investigator would interfere with his/her continued participation if the risk of continuing participation outweighs the potential benefit.
- 5. Subject develops erythrodermic, guttate, or pustular form of psoriasis.
- 6. Subjects considered to have either a suspected new latent tuberculosis (LTB) infection or who develop an active TB or NTMB infection during the study (including but not limited to, conversion demonstrated by IGRA or other diagnostic means) must be immediately discontinued from study medication; an Early Withdrawal Visit must be scheduled as soon as possible, but not later than the next regular visit.

Confirmed active TB is an SAE and must be captured on an SAE Report Form and provided to the Sponsor in accordance with SAE reporting requirements. As with all SAEs, periodic

follow-up reports should be completed as per protocol requirements until such time as the TB infection resolves.

- 8. Subject uses prohibited concomitant medications, with the exception of topicals, as defined in this protocol (Section 7.8.2), that may present a risk to the safety of the subject in the opinion of the Investigator and/or the Medical Monitor.

  9. Subject has a clinical laborate.
- - Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 and above: subjects must be withdrawn regardless of relationship to study drug or duration of event.
  - CTCAE Grade 2
    - Subjects may remain in the study if the event is transient. If a subject has a Grade 2 laboratory abnormality, a retest is required within 1 to 2 weeks at a scheduled or unscheduled visit. If the repeat value is below Grade 2, the subject may receive the next scheduled study treatment. If the value on the repeat is still Grade 2 or above, a second repeat test must be performed and results made available prior to the next scheduled study treatment. If this second repeat value is still Grade 2 or above, the subject must be withdrawn.
- 10. Subject has active suicidal ideation as indicated by a positive response ("Yes") to questions 4 or 5 or to the suicidal behavior questions of the "Since Last Visit" version of the self-rated electronic Columbia-Suicide Severity Rating Scale (eC-SSRS). The subject should be referred immediately to a Mental Healthcare Professional and must be withdrawn from the study.
- 11. Subjects with a HADS-D score >15 must be withdrawn. Any subject who develops a HADS-D score of >10 during the study should be referred immediately to a Mental Healthcare Professional for further evaluation and potential withdrawal by the Investigator.
- 12. Subject does not achieve PASI75 at Week 12 or later following study treatment in PS0011.
- 13. Subject experiences an AE as described below:
  - Any CTCAE Grade 3 and above adverse event (AE) that is assessed as related to study drug in the opinion of the Investigator
    - If the event is deemed to be not related to study drug by the Investigator, the subject may remain in the study after approval by the Medical Monitor.
  - Any CTCAE Grade 2 event that is evaluated as related to study drug in the opinion of the Investigator, is persistent, and falls into any of the following System Organ Classes (SOCs): "Blood and lymphatic disorders," "Cardiac disorders," or "Vascular disorders."
    - Persistent is defined as lasting 28 days or more, which spans at least 2 scheduled injections.

**UCB** 12 Aug 2016 PS0011

Investigators should attempt to obtain information on subjects in the case of withdrawal. For subjects considered as lost to follow-up, the Investigator should make an effort (at least 1 phone call and 1 written message to the subject), and document his/her effort (date and summary of the phone call and copy of the written message in the source documents) to complete the final evaluation. All results of these evaluations and observations, together with a narrative description of the reason(s) for removing the subject, must be recorded in the source documents. The eCRF must document the primary reason for withdrawal.

Investigators should contact the Medical Monitor, whenever possible, to discuss the withdrawal of a subject in advance.

### 6.3.1 **PDILI IMP discontinuation criteria**

Subjects with PDILI must be assessed to determine if investigational medicinal product (IMP) must be discontinued. In addition, all concomitant medications and herbal supplements that are not medically necessary should also be discontinued.

The PDILI criteria below require immediate and permanent discontinuation of IMP:

- Subjects with either of the following:
  - ALT or AST >5xULN
  - ALT or AST ≥3xULN and coexisting total olirubin ≥2xULN
- Subjects with ALT or AST  $\geq 3xULN$  who exhibit temporally associated symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, right upper quadrant pain or tenderness. Hypersensitivity symptoms include fever (without clear alternative cause), rash, or eosinophilia (ie, >5%).

The PDILI criterion below allows for subjects to continue on IMP at the discretion of the Investigator.

Subjects with ALT or AST  $\ge 3x$ ULN (and  $\ge 2x$  baseline) and < 5xULN, total bilirubin  $\leq$ 2xULN, and no eosinophilia (ie,  $\leq$ 5%), with no fever, rash, or symptoms of hepatitis (eg, fatigue, nausea, vomiting, right upper quadrant pain or tenderness).

Evaluation of PDILI must be initiated as described in Section 9.7.1. If subjects are unable to comply with the applicable monitoring schedule, IMP must be discontinued immediately.

Investigators should attempt to obtain information on subjects in the case of IMP discontinuation to complete the final evaluation. Subjects with PDILI should not be withdrawn from the study until investigation and monitoring are complete. All results of these evaluations and observations, as well as the reason(s) for IMP discontinuation and subject withdrawal (if applicable), must be recorded in the source documents. The eCRF must document the primary reason for IMP discontinuation.

### 7 STUDY TREATMENT

## 7.1 Description of investigational medicinal product

Placebo will be supplied as 0.9% sodium chloride aqueous solution (physiological saline, preservative free) of pharmacopoeia (USP/Ph.Eur) quality appropriate for injection.

Further details of the study medication and specifications are provided in the MMP Handling Manual.

### 7.2 Treatments to be administered

During the Treatment Period, all subjects will receive bimekizumab or placebo Q4W administered sc (refer to Figure 5–1 for further details).

Subjects who received placebo or bimekizumab 64mg, 160mg, or 320mg loading dose + 160mg Q4W in PS0010 must achieve PASI90 response at Week 12 in PS0010 to enter the PS0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while on these treatments will be assigned to receive bimekizumab 160mg or 320mg Q4W at Baseline in PS0011 as follows:

- Subjects receiving placebo and binekizumab 64mg Q4W in PS0010 will be assigned to bimekizumab 160mg Q4W in PS0001.
- Subjects receiving bimekizumab 160mg O4W and 320mg loading dose + 160mg O4W in PS0010 will be assigned to bimekizumab 320mg Q4W in PS0011.

Subjects who receive bimekizumab 320mg or 480mg Q4W in PS0010 will be assigned to receive bimekizumab 320mg Q4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010.

The study medication is to be administered in the clinic by study site staff as 2 sc injections for all study treatments in PS0011. Suitable areas for sc injections are the lateral abdominal wall and upper outer thigh. Injection sites should be rotated, and injections should not be given into areas where the skin is tender, bruised, red, or hard.

The minimum time between doses should be no less than 24 days and no more than 32 days for Q4W dosing.

An IMP Handling Manual will be provided to each site containing instructions regarding drug preparation and dosing.

## 7.3 **Packaging**

Bimekizumab and placebo will be packaged and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. It will be suitably packaged in


12 Aug 2016 PS0011

such a way as to protect the product from deterioration during transport and storage. Further information regarding storage and transport conditions are provided in the IMP Handling

Connical drug supplies will be labeled in accordance with the current International Council for Harmonisation (ICH) guidelines on Good Clinical Practice (GCP) and GMP and will include any locally required statements. If necessary, labels will be translated into the local language

7.5 Handling and storage requirements.

Bimekizuments.

Bimekizumab and placebo must be stored under refrigerated conditions (2°C to 8°C) and protected from light. The study drug must not be frozen.

The Investigator (or designee) is responsible for the safe and proper storage of IMP at the site. Investigational medicinal product stored by the Investigator is to be kept in a secured area with limited access according to the storage conditions mentioned on the label.

Appropriate storage conditions must be ensured by controlling the temperature (eg. room, refrigeration unit) and by completion of a temperature log in accordance with local requirements on a regular basis per study manuals, showing actual and minimum/maximum temperatures reached over the time interval.

Study drug will be shipped to the study sites in temperature controlled containers. Out-of-range shipping or storage conditions must be brought to the attention of the Sponsor or designee, as per instructions contained in the IMP Handling Manual. Authorization to use any out-of-range IMP must be documented and received prior to dispensing or administering the IMP at the study site.

## Drug accountability 7.6

A Drug Accountability form will be used to record IMP dispensing and return information on a by-subject basis and will serve as source documentation during the course of the study. Details of any IMP lost, damaged (due to breakage or wastage), not used, partially used, disposed of at the study site, or returned to the Sponsor or designee must also be recorded on the appropriate forms. All supplies and pharmacy documentation must be made available throughout the study for UCB (or designee) to review?

In order to maintain the blind, all IMP documentation (eg, shipping receipts, drug accountability logs, interactive web or voice response system [IXRS] treatment assignments) must be maintained and accessed only by trained unblinded site personnel. Designated unblinded site personnel must be appropriately trained and licensed (per country guidelines) to administer injections.

Blinded study staff may be delegated the responsibility to receive, inventory, and destroy the used kits. The packaging identifies each kit by a unique number that does not correlate to the contents and does not unblind study site staff. Unblinded study staff will be responsible for the preparation (eg, breaking tamper proof sticker on kit) of the IMP, including recording the administration information on the source document.

The Investigator (or designee) is responsible for retaining all used, unused, and partially used containers of IMP until returned or destroyed.


The Investigator may assign some of the Investigator's duties for drug accountability at the study site to an appropriate pharmacist/designee.

The Investigator must ensure that the IMP is used only in accordance with the protocol.

Periodically, and/or after completion of the clinical phase of the study, all used (including empty containers), partially used, unused, damaged, and/or expired IMP must be reconciled and either destroyed at the site according to local laws, regulations, and UCB SOPs or returned to UCB (or designee). Onsite destruction of used kits only may be allowed with prior approval from the Sponsor or designee after reconciliation. Investigational medicinal product intended for the study cannot be used for any other purpose than that described in this protocol.

## 7.7 Procedures for monitoring subject compliance

During the Treatment Period of this study, study medication will be administered in the clinic and compliance will be determined at the visit by study personnel. Drug accountability must be recorded on the Drug Accountability Form.

## 7.8 Concomitant medication(s)/treatment(s)

All concomitant medications, including over the counter products, herbal, traditional remedies, vitamin/mineral supplements, other dietary supplements, "nutraceuticals," and hormones must be recorded in the subject's source documentation (eg, clinical chart) and on the eCRF. This record should include the name of the drug, the dose, the route and date(s) of administration, and the indication for use.

The Investigator should examine the acceptability of all concomitant procedures, medications, topical preparations, and dietary supplements not explicitly prohibited in this study, and if necessary, discuss with the Medical Monitor.

In order to ensure that appropriate concomitant therapy is administered, subjects will be instructed to consult with the Investigator prior to taking any medication (either self-administered nonprescription drugs or prescription therapy prescribed by another physician).

## 7.8.1 Permitted concomitant treatments (medications and therapies)

## **Topical medications**

Subjects may continue to use topical moisturizers or emollients, bath oils, or oatmeal bath preparations-for skin conditions during the study, as needed. Over-the-counter shampoos for the treatment of psoriasis of the scalp are also permitted.

Subjects will be allowed to use topical medications (corticosteroids, retinoids, Vitamin D analogs coal tar, etc) as needed during this extension study.

## Other medications

Subjects who were already receiving an established nonsteroidal anti-inflammatory drug (NSAID) regimen during PS0010 may continue their use during this study. However, initiation of, or increase in dosage of, NSAIDs during the study (especially in subjects with a history of gastrointestinal [GI] intolerance to NSAIDs or a history of GI ulceration) should be done with caution. Intra-articular injections for arthritis of the knee are allowed.

Bimekizumab

Subjects who were already receiving an established anti-depressant regimen during PS0010 may continue their use during this study.

### 7.8.2 Prohibited concomitant treatments (medications and therapies)

The list of prohibited concomitant medications is provided Table 7–1.

## Prohibited psoriasis medications during PS0011

# Drug Systemic retinoids Systemic treatment (non-biological): systemic immunosuppressant agents (eg, methotrexate, cyclosporine, azathioprine, thioguanine) PACIFIC OF TO APPLICATION APPL systemic fumarate systemic corticosteroids phototherapy or chemophototherapy Anti-TNFs: infliximab (including biosimilar), golimumab etanercept (including biosimilar) certolizumab pegol adalimumab (including biosimilar) Other biologics and other systemic therapies: apremilast ustekinumab Anti-IL-17 therapy Any other antipsoriatic agent (systemic)

Any other antipsoriatic agent (topical) under investigation IL=interleukin; TNF=tumor necrosis factor

Subjects who take prohibited medications may be withdrawn from study treatment but followed until the SFU Visit. The decision to withdraw a subject for taking prohibited medications should be made in consultation with the Medical Monitor.

# Vaccines \_\_\_

Administration of live (including attenuated) vaccines is not allowed during the conduct of the study or for 20 weeks after the last dose of study drug. Administration of inactivated vaccines is allowed during the study at the discretion of the Investigator.

## Blinding

ris docur?.9 Due to differences in presentation of the IMP (bimekizumab and placebo), special precautions will be taken to ensure study blinding, and study sites will have blinded and unblinded personnel.


12 Aug 2016 PS0011

Bimekizumab and placebo injections will be prepared and administered at the study sites by unblinded dedicated study personnel who will only be responsible for dosing and drug accountability.

Study sites will be required to have a written blinding plan in place, signed by the Principal Investigator, which will detail the site's steps for ensuring that the double-blind nature of the study is maintained.

During the study, the Sponsor will provide blinded and unblinded site monitors for the purposes of verifying safety, efficacy, and drug administration and documentation records. Blinded study monitors and study site personnel, blinded to treatment assignment, will not discuss or have access to any drug-related information.

When the feeder (PS0010) study is unblinded, selected PS0010 study team members will have access to subject-level data. Because treatment assignment in PS0011 is based on PASI90 response at Week 12 of PS0010 as opposed to randomization, Sponsor personnel with such access to the PS0010 data will know the treatment assignments of all PS0010 subjects including those continuing in PS0011. This operational unblinding to PS0011 treatment assignment will pertain to selected clinical PS0010 study team members (some of whom may be involved in PS0011) but will not extend to blinded staff at the investigational sites of PS0011.

While the blinding of Sponsor clinical study team members is important for ensuring the integrity of data collection and analysis in a controlled study, this unblinding is considered acceptable because the primary evaluation of efficacy, upon which sample size calculations were based, will be performed in a blinded manner using Week 12 data of PS0010. Additionally, because investigational site staff collecting and recording study data remain blinded, those data will not be impacted by the unblinding of selected Sponsor clinical study team members. Finally, to ensure that unblinding of study team members did not impact the primary safety outcome of PS0011, sensitivity analyses will be outlined in the SAP to evaluate what, if any, impact there was on the results based on queries that resulted in changes to the AE data following the unblinding of PS0010.

Further details are provided in the study manuals and site blinding plan.

## 7.9.1 Procedures for maintaining and breaking the treatment blind

## 7.9.1.1 Maintenance of study treatment blind

All subject treatment details (bimekizumab or placebo) will be allocated and maintained by the IXRS.

# 7.9.1.2 Breaking the treatment blind in an emergency situation

The integrity of this clinical study must be maintained by observing the treatment blind. In the event of an emergency for which the appropriate treatment for a subject cannot be made without knowing the treatment assignment, it will be possible to determine to which treatment arm and dose the subject has been allocated by contacting the IXRS. All sites will be provided with details of how to contact the system for code breaking at the start of the study. The Medical Monitor or equivalent should be consulted prior to unblinding, whenever possible.


The Clinical Project Manager will be informed immediately via the IXRS when a code is broken, but will remain blinded to specific treatment information. Any unblinding of the IMP performed by the Investigator must be recorded in the source documents and on the Study Termination

No randomization will be performed in this study. An IXRS will be used for assigning eligible subjects to treatment based on a predetermined assignment schedule. An independent biostatistician or designee who is not involved in this study or the form produce this assignment schedule. Section 7.2.

Subjects will continue with the 5-digit subject numbers assigned by IXRS in the preceding study.

## STUDY PROCEDURES BY VISIT

Table 5–1 (schedule of study assessments) provides a general overview of study assessments. A list of procedures to be completed at each visit is provided in the sections that follow.

- Visit windows of  $\pm 3$  days on either side of the scheduled dosing are permitted for all visits other than the SFU Visit (see below); however, the Investigator should try to keep the subjects on the original dosing schedule. The window of  $\pm 3$  days is relative to the first dose (Baseline) and applicable for all subsequent visits. Changes to the dosing schedule outside of the 3-day window must be discussed with the Medical Monitor.
- The minimum time between doses should be no less than 24 days and no more than 32 days for Q4W dosing.
- For the SFU Visit (20 weeks after the last dose of bimekizumab or placebo), the visit should occur no more than 3 days prior to the scheduled visit date and within 7 days after the scheduled visit date (-3 days/+7 days).

## 8.1 **Baseline Visit**

The Baseline assessments noted with an \* will be obtained at the Week 12 Visit of PS0010 and do not need to be recorded on the eCRF for this study.

All procedures or assessments will be performed prior to administration of study drug, unless otherwise noted. The following procedures or assessments will be performed:

- Ensure that a separate Informed Consent Form was completed by the subject for PS0011 during the Week 8 or Week 12 Visit of PS0010 (must be done prior to any PS0011 study procedures)
- Confirm that a TB test (IGRA) was performed at the Week 8 Visit of PS0010 and the results were negative
- Assessment of inclusion/exclusion criteria
- Vital signs (blood pressure, pulse rate, and temperature)\*
- Body weight\*

- Physical examination\*
- Record 12-lead ECG\*
- eC-SSRS\*
- TB questionnaire\*
- PASI\*
- IGA\*
- DLQI\*
- BSA\*
- mNAPSI\*
- PSSI\*
- PGADA\*
- SF-36\*
- HADS\*
- Obtain blood samples for:
- btain blood samples for:

  Standard safety laboratory tests (hematology and biochemistry)\*

  Bimekizumab plasma concentration\*

  nti-bimekizumab antibodies\*

  urine sample for:

  dard safety laboratory tests (urinalysis)\*

  pregnancy test for women of ant medications

  s

  INRS
  - Bimekizumab plasma concentration\*
- Obtain urine sample for:
- Concomitant medications
- Record AEs
- Contact the IXRS
- Study medication administration (after all other visit assessments are completed)

## Week 4 (±3 days) 8.2

All procedures or assessments will be performed prior to administration of study drug, unless otherwise noted. The following procedures or assessments will be performed:

- Vital signs (blood pressure, pulse rate, and temperature)
- eC-SSRS
- **PASI**
- **IGA**
- **DLQI**
- **BSA**
- mNAPSI
- **PSSI**
- HADS
- Obtain blood samples for:
  - Standard safety laboratory tests (hematology and biochemistry)
  - Bimekizumab plasma concentration
  - Anti-bimekizumab antibodies
- Obtain urine sample for:
  - Urine pregnancy test for women of childbearing potential
- Concomitant medications
- Record AEs
- Contact the IXRS
- aial and any extensions of variations thereof.

  Ton application and any extensions of variations thereof. Study medication administration (after all other visit assessments are completed)

### Week 8 (±3 days); Week 16 (±3 days); Week 32 (±3 days); and 8.3 Week 40 (±3 days)

All procedures or assessments will be performed prior to administration of study drug (if applicable), unless otherwise noted. The following procedures or assessments will be performed:

- Vital signs (blood pressure, pulse rate, and temperature)
- eC-SSRS
- **PASI**
- **IGA**
- **BSA**
- HADŞ 🛇
- Obtain blood samples for:

Standard safety laboratory tests (hematology and biochemistry)

- Bimekizumab plasma concentration (not collected at Week 32)
- Anti-bimekizumab antibodies (not collected at Week 32)
- Obtain urine sample for:
  - Urine pregnancy test for women of childbearing potential

- Concomitant medications
- Record AEs
- Contact the IXRS
- Study medication administration (after all other visit assessments are completed)

### 8.4 Week 12 (±3 days)

The following procedures or assessments will be performed prior to administration of study drug (if applicable):

- Vital signs (blood pressure, pulse rate, and temperature)
- eC-SSRS
- TB questionnaire
- **PASI**
- **IGA**
- DLQI
- **BSA**
- mNAPSI
- **PSSI**
- **PGADA**
- SF-36
- HADS
- Obtain blood samples for:
  - Standard safety laboratory tests (hematology and biochemistry)
  - Bimekizumab plasma concentration
  - Anti-bimekizumab antibodies
- Obtain urine sample for:
  - Standard safety laboratory tests (urinalysis)
  - Urine pregnancy test for women of childbearing potential
- Concomitant medications
- Record AEs
- Contact the IXRS
- Study medication administration (after all other visit assessments are completed)

### Week 20 (±3 days); Week 28 (±3 days); and Week 44 (±3 days) 8.5

Jany extensions or variations thereof The following procedures or assessments will be performed prior to administration of study drug (if applicable):

- Vital signs (blood pressure, pulse rate, and temperature)
- eC-SSRS
- **PASI**
- **IGA**
- BSA
- **HADS**
- Obtain blood samples for:
  - Standard safety laboratory tests (hematology and biochemistry)
  - Bimekizumab plasma concentration (collected only at Week 28)
  - Anti-bimekizumab antibodies (collected only at Week 28)
- Obtain urine sample for:
  - Urine pregnancy test for women of childbearing potential
- Concomitant medications
- Record AEs
- Contact the IXRS
- Study medication administration (after all other visit assessments are completed)

### 8.6 Week 24 (±3 days)

The following procedures or assessments will be performed prior to administration of study drug (if applicable):

- Vital signs (blood pressure, pulse rate, and temperature)
- Record 12-lead ECG
- eC-SSRS
- TB questionnaire • PASI

  - **mNAPSI**

- **PSSI**
- **PGADA**
- SF-36
- **HADS**
- Obtain blood sample for:
  - Standard safety laboratory tests (hematology and biochemistry)
- Obtain urine sample for:
  - Standard safety laboratory tests (urinalysis)
  - Urine pregnancy test for women of childbearing potential
- Concomitant medications
- Record AEs
- Contact the IXRS
- Ation and any extensions or variations thereof. Study medication administration (after all other visit assessments are completed)

### 8.7 Week 36 (±3 days)

The following procedures or assessments will be performed prior to administration of study drug Vital signs (blood pressure, pulse rate, and temperature) (if applicable):

- eC-SSRS
- TB questionnaire
- **PASI**
- **IGA**
- DLQI
- **BSA**
- mNAPSI
- PSSI
- **PGADA**
- SF-36
- **HADS**
- Obtain blood sample for:
  - Standard safety laboratory tests (hematology and biochemistry)
- Obtain urine sample for:

- Standard safety laboratory tests (urinalysis)
- Urine pregnancy test for women of childbearing potential
- Concomitant medications
- Record AEs
- Contact the IXRS
- Study medication administration (after all other visit assessments are completed)

# 8.8

The following procedures or assessments will be performed:

- Vital signs (blood pressure, pulse rate, and temperature)
- Body weight
- Physical examination
- Record 12-lead ECG
- eC-SSRS
- TB questionnaire
- **PASI**
- **IGA**
- DLQI
- **BSA**
- mNAPSI
- **PSSI**
- **PGADA**
- SF-36
- **HADS**
- Obtain blood samples for:
  - TB test (IGRA; QuantiFERON TB GOLD test is recommended)
    - Standard safety laboratory tests (hematology and biochemistry)
  - Bimekizumab plasma concentration
  - Anti-bimekizumab antibodies
- Obtain urine sample for:
  - Standard safety laboratory tests (urinalysis)
  - Urine pregnancy test for women of childbearing potential

.val


- Concomitant medications
- Record AEs
- Contact the IXRS

# COPT application and any extensions of variations thereof. 8.9 SFU Visit (20 weeks after the last dose of bimekizumab or placebo: -3/+7 days)

The following procedures or assessments will be performed:

- Vital signs (blood pressure, pulse rate, and temperature)
- Body weight
- Physical examination
- eC-SSRS
- Record 12-lead ECG
- **PASI**
- IGA
- **HADS**
- Obtain blood samples for:
  - Standard safety laboratory tests (hematology and biochemistry)
  - Serum pregnancy test for women of childbearing potential
  - Bimekizumab plasma concentration
  - Anti-bimekizumab antibodies
- Obtain urine sample for:
  - Standard safety laboratory tests (urinalysis)
- Concomitant medications
- Record AEs (including assessment for development of other forms of psoriasis)
- Contact the IXRS

# **Early Withdrawal Visit**

Subjects withdrawing early from the study (see Section 6.3) will undergo the same assessments as the Week 48 Visit (see Section 8.4) and will enter the SFU Period.

# **Unscheduled Visit**

This document At the Investigator's discretion, an Unscheduled Visit may be completed at any time during the study, but prior to the SFU Visit, if deemed necessary for the subject's safety and well-being.

If an additional visit (or unscheduled visit) is conducted due to safety or efficacy reasons, an eC-SSRS assessment will be performed with the subject during the visit. If an additional visit (or


12 Aug 2016 PS0011

unscheduled visit) is conducted for reasons other than safety or efficacy concerns any extensions or variations thereof. (eg, replacement of lost medication, repeated collection of a laboratory specimen due to collection or analysis issues), an eC-SSRS will not be required at these visits.

At this visit, any of the following assessments may be performed, depending on the reason for the visit:

- Vital signs
- Physical examination
- Record 12-lead ECG
- eC-SSRS
- If medically indicated, obtain blood sample(s) for:
  - Standard safety laboratory tests (hematology and biochemistry)
  - The blood sample may also be used for PK assessments, if needed
- Obtain urine sample for standard safety laboratory tests (urinalysis; including urine pregnancy test)
- Concomitant medications
- Record AEs

### ASSESSMENT OF SAFET 9

### Adverse events 9.1

### **Definition of AE** 9.1.1

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

In order to ensure complete safety data collection, all AEs occurring during the study (ie, after the signing of the Informed Consent form), including any pretreatment and posttreatment periods required by the protocol, must be reported in the eCRF even if no IMP was taken but specific study procedures were conducted. This includes all AEs not present prior to the initial visit and all AEs that recurred or worsened after the initial visit.

Signs or symptoms of the condition/disease for which the IMP is being studied should be recorded as AEs only if their nature changes considerably or their frequency or intensity increases in a clinically significant manner as compared to the clinical profile known to the Investigator from the subject's history or the Baseline Period.

# 9.1.2 Procedures for reporting and recording AEs

The subject will be given the opportunity to report AEs spontaneously. A general prompt will also be given at each study visit to detect AEs. For example:

"Did you notice anything unusual about your health (since your last visit)?"

In addition, the Investigator should review any self-assessment procedures employed in the study.

# 9.1.3 Description of AEs

When recording an AE, the Investigator should use the overall diagnosis or syndrome using standard medical terminology, rather than recording individual symptoms or signs. The eCRF and source documents should be consistent. Any discrepancies between the subject's own words on his/her own records and the corresponding medical terminology should be clarified in the source documentation.

When recording the severity of an AE in the CRF (ie, mild, moderate, or severe), the Investigator must refer to the CTCAE Version 4

(http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm). Details for completion of the AE eCRF (including judgment of severity and relationship to IMP) are described in the eCRF Completion Guidelines.

# 9.1.4 Follow up of AEs

An AE should be followed until it has resolved, has a stable sequelae, the Investigator determines that it is no longer clinically significant, or the subject is lost to follow up. Further details regarding follow up of PDILI events are provided in Section 9.7.1.4.

If an AE is ongoing at the end of the study for a subject, follow up should be provided until resolution/stable level of sequelae is achieved, or until the Investigator no longer deems that it is clinically significant, or until the subject is lost to follow up. If no follow up is provided, the Investigator must provide a justification. The follow up will usually be continued for 20 weeks after the subject has discontinued his/her IMP.

# 9.1.5 Rule for repetition of an AE

An increase in the intensity of an AE should lead to the repetition of the AE being reported with:

- The outcome date of the first AE that is not related to the natural course of the disease being the same as the start date of the repeated AE, and the outcome of "worsening"
- The AE verbatim term being the same for the first and repeated AE, so that the repeated AE can be easily identified as the worsening of the first one

# 9.1.6 Pregnancy

If an Investigator is notified that a subject has become pregnant after the first intake of any IMP, the Investigator must immediately notify UCB's Patient Safety (PS) department by providing the completed Pregnancy Report and Outcome form (for contact details see SAE reporting information at the beginning of this protocol). The subject should be withdrawn from the study as soon as pregnancy is known (by positive pregnancy test), and the following should be completed:


- The subject should return for an Early Withdrawal Visit.
- The subject should immediately stop the intake of the IMP.
- A SFU Visit should be scheduled 20 weeks after the subject has discontinued her IMP.

The Investigator must inform the subject of information currently known about potential risks and about available treatment alternatives.

The pregnancy will be documented on the Pregnancy Report and Outcome form provided to the Investigator. The progression of the pregnancy and the eventual birth (if applicable) must be followed up using the Pregnancy Report and Outcome form in which the Investigator has to report on the health of the mother and of the child. Every reasonable attempt should be made to follow the health of the child for 30 days after birth for any significant medical issues. In certain circumstances, UCB may request that follow up is continued for a period longer than 30 days. If the subject is lost to follow up and/or refuses to give information, written documentation of attempts to contact the subject needs to be provided by the Investigator and filed at the site. UCB's PS department is the primary contact for any questions related to the data collection for the pregnancy, eventual birth, and follow up.

In cases where the partner of a male subject enrolled in a clinical study becomes pregnant, the Investigator or designee is asked to contact the subject to request consent of the partner via the Partner Pregnancy Consent form that has been approved by the responsible IRB/IEC and should be available in the Investigator site file. In case of questions about the consent process, the Investigator may contact the UCB/Contract Research Organization (CRO) contract monitor for the study. The Investigator will complete the Pregnancy Report and Outcome form and send it to UCB's PS department (for contact details see SAE reporting information at the beginning of this protocol) only after the partner has agreed that additional information can be captured and has provided the signed Partner Pregnancy Consent form. UCB's PS department is also the primary contact for any questions related to the data collection for the partner pregnancy, eventual birth, and follow up.

A pregnancy becomes an SAE in the following circumstances: miscarriage, abortion (elective or spontaneous), unintended pregnancy after hormonal contraceptive failure (if the hormonal contraceptive was correctly used), ectopic pregnancy, fetal demise, or any congenital anomaly/birth defect of the baby. Those SAEs must be additionally reported using the Investigator SAE Report form.

# 9.1.7 Suspected transmission of an infectious agent via a medicinal product

For the purposes of reporting, any suspected transmission of an infectious agent via a medicinal product should be considered as an SAE; such cases must be reported immediately, recorded in the AE module of the eCRF, and followed as any other SAE. Any organism, virus, or infectious particle (eg, prion protein transmitting transmissible spongiform encephalopathy), pathogenic or nonpathogenic, is considered an infectious agent.

# 9.1.8 Overdose of investigational medicinal product

Excessive dosing (beyond that prescribed in the protocol and including overdose) should be recorded in the eCRF. Any SAE or nonserious AE associated with excessive dosing must be

followed as any other SAE or nonserious AE. These events are only considered AEs or SAEs if there are associated clinical signs and symptoms or if the act of taking the excess medicine itself is an AE or SAE (eg., suicide attempt).

### 9.1.9 Safety signal detection

Selected data from this study will be reviewed periodically to detect as early as possible any safety concern(s) related to the IMP so that Investigators, clinical study subjects, regulatory authorities, and IRBs/IECs will be informed appropriately and as early as possible.

In addition, an independent Data Monitoring Committee (DMC) will periodically review and monitor the safety data from this study and advise UCB. Details are provided in the DMC Charter. A Cardiovascular Adjudication Committee will also periodically review and monitor the safety data from this study and advise UCB. Details are provided in the Cardiovascular Adjudication Committee Charter.

The Study Physician or medically qualified designee/equivalent will conduct an ongoing review of SAEs and perform ongoing SAE reconciliations in collaboration with the PS representative.

As appropriate for the stage of development and accumulated experience with the IMP, medically qualified personnel at UCB may identify additional safety measures (eg, AEs, vital signs, laboratory, or ECG results) for which data will be periodically reviewed during the course of the study.

### Serious adverse events 9.2

### 9.2.1 **Definition of SAE**

Once it is determined that a subject experienced an AE, the seriousness of the AE must be determined. An SAE must meet 1 or more of the following criteria:

- Death
- Life-threatening

(Life-threatening does not include a reaction that might have caused death had it occurred in a more severe form.)

- Significant or persistent disability/incapacity
- Congenital anomaly/birth defect (including that occurring in a fetus)
- Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious

Important medical events may include, but are not limited to, potential Hy's Law [see Section 9.5], allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.)

Initial inpatient hospitalization or prolongation of hospitalization

(A patient admitted to a hospital, even if he/she is released on the same day, meets the criteria for the initial inpatient hospitalization. An emergency room visit that results in admission to the hospital would also qualify for the initial inpatient hospitalization criteria.

Hospitalizations for reasons not associated with the occurrence of an AE [eg, preplanned surgery or elective surgery for a pre-existing condition that has not worsened or manifest in an unusual or uncharacteristic manner] do not qualify for report. for this condition, it is not appropriate to record the surgery or hospitalization as an SAE, since there is no AE upon which to assess the serious criteria. Please note that, if the pre-existing condition has worsened or manifested in an unusual or uncharacteristic manner, this would then qualify as an AE and, if necessary, the seriousness of the event would need to be determined.)

Note: Confirmed active TB is always to be considered as an SAE and must be captured on an SAE Report Form and provided to the Sponsor in accordance with SAE reporting requirements.

### **Procedures for reporting SAEs** 9.2.2

If an SAE is reported, UCB must be informed within 24 hours of receipt of this information by the site (see contact information for SAE reporting listed in the SAE Reporting section at the front of the protocol). The Investigator must forward to UCB (or its representative) a duly completed "Investigator SAE Report Form for Development Drug" (SAE report form) provided by UCB, even if the data are incomplete, or if it is obvious that more data will be needed in order to draw any conclusions. Information recorded on this form will be entered into the global safety database.

An Investigator SAE report form will be provided to the Investigator. The Investigator SAE Report form must be completed in English.

It is important for the Investigator, when completing the SAE report form, to include the assessment as to a causal relationship between the SAE and the IMP administration. This insight from the Investigator is very important for UCB to consider in assessing the safety of the IMP and in determining whether the SAE requires reporting to the regulatory authorities in an expedited manner.

Additional information (eg. autopsy or laboratory reports) received by the Investigator must be provided within 24 hours. All documents in the local language must be accompanied by a translation in English, or the relevant information included in the same document must be summarized in the Investigator SAE report form.

The Investigator is specifically requested to collect and report to UCB (or its representative) any SAEs (even if the Investigator is certain that they are in no way associated with the IMP), up to 30 days from the end of the study for each subject, and to also inform participating subjects of the need to inform the Investigator of any SAE within this period. Serious AEs that the Investigator thinks may be associated with the IMP must be reported to UCB regardless of the time between the event and the end of the study.

12 Aug 2016 PS0011

Upon receipt of the SAE report form, UCB will perform an assessment of expectedness of the reported SAE. The assessment of the expectedness of the SAE is based on the IB.

Information on SAEs obtained after clinical database lock will be captured through the PS database without limitation of time.

9.3 Immediate reporting of AEs

The following AEs must be reported.

- SAE: AE that the Investigator classifies as serious by the definitions in Section 9.2.1 regardless of causality
- Suspected transmission of an infectious agent via a medicinal product
- AEs of special interest as defined in Section 9.5

### 9.4 **Anticipated SAEs**

The following Anticipated SAEs (Table 9–1) are anticipated to occur in the population studied in this protocol at some frequency that is independent of drug exposure. This original list will remain in effect for the duration of the protocol. Note that listed events will not be regarded as anticipated SAEs if they are life-threatening or if they result in the death of the study subject.

This list does not change the Investigator's obligation to report all SAEs (including Anticipated SAEs) as detailed in Section 9.2.2.

Table 9–1: Anticipated SAEs for the population of subjects with moderate to severe chronic plaque psoriasis

| MedDRA® system order class | MedDRA preferred term |
|---|---|
| Skin and subcutaneous tissue disorders | Any psoriatic condition HLT |
| Musculoskeletal and connective tissue disorders | Psoriatic arthropathy |

HLT=high level term, MedDRA=Medical Dictionary for Regulatory Activities; SAE=serious adverse event Note: Exception Listed events will not be regarded as anticipated SAEs if they are life-threatening or if they result in the death of the study subject.

# Adverse events of special interest

An AE of special interest is any AE that a regulatory authority has mandated be reported on an expedited basis, regardless of the seriousness, expectedness, or relatedness of the AE to the administration of a UCB product/compound.

Potential Hy's Law, defined as  $\ge 3xULN$  ALT or AST with coexisting  $\ge 2xULN$  total bilirubin in the absence of  $\geq 2xULN$  ALP, with no alternative explanation for the biochemical abnormality, must ALWAYS be reported to UCB as an AE of special interest (ie, without waiting for any additional etiologic investigations to have been concluded). Follow-up information should then


be reported if an alternative etiology is identified during investigation and monitoring of the subject.

# 9.6 Adverse events for special monitoring

UCB has identified AEs for special monitoring (AESM). An AESM is an AE or safety topic for which special monitoring, additional data collection activities, and/or enhanced signal detection activities (within UCB), are considered appropriate. Identified AESM can be of particular interest based on findings from the IMP clinical program to date, potential risks generally associated with biologic immunomodulators, or comorbidities and risk factors prevalent in the study population.

Adverse events for special monitoring for this study include: serious infections (including opportunistic infections and TB; see Section 9.8.1), cytopenias, hypersensitivities, suicide ideation or behavior (assessed using the eC-SSRS; see Section 9.8.6), depression and anxiety (assessed using the HADS; see Section 12.9), major cardiovascular events, and liver function test changes/enzyme elevations (ALT, AST, bilirubin; see Section 9.7.1), malignancies, and inflammatory bowel diseases.

# 9.7 Laboratory measurements

Clinical laboratory assessments consist of serum chemistry, hematology, and urinalysis. A centralized laboratory will be used to supply all laboratory test supplies and analyze all blood and urine samples for hematology, biochemistry, and urinalysis measurements. Any unscheduled laboratory testing should also be collected using the central laboratory. Laboratory parameters to be measured are listed in Table 9–2.

Specific details regarding the handling and processing of serum chemistry, hematology, and urinalysis samples are provided in the study laboratory manuals.

Table 9-2: Laboratory measurements

| Hematology | Chemistry | Urinalysis |
|---|---|---|
| Basophils | Calcium | Albumin |
| Eosinophils | Chloride | Bacteria |
| Lymphocytes | CRP | Crystals |
| Atypical lymphocytes | Magnesium | Glucose |
| Monocytes | Potassium | pH |
| Neutrophils | Sodium | RBC |
| Hematocrit | Glucose | WBC |
| Hemoglobin | BUN | Urine dipstick for pregnancy testing <sup>a</sup> |
| MCH | Creatinine | |
| MCHC | ALP | |
| MCV | AST | |

### Table 9-2: Laboratory measurements

| Hematology | Chemistry | Urinalysis |
|----------------|--------------------------------------|------------|
| Platelet count | ALT | |
| RBC count | GGT | |
| WBC count | Total bilirubin | oliolia . |
| | LDH | 2,70 |
| | Total cholesterol | ans |
| | Serum pregnancy testing <sup>a</sup> | 3/15/10 |

ALP=alkaline phosphatase; ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; CRP=C-reactive protein; GGT=gamma glutamyltransferase; LDH=lactate dehydrogenase; MCH=mean corpuscular hemoglobin; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell; WBC=white blood cell

Assessments of PK variables are described in Section 10. Assessments of immunological variables are described in Section 11.

### 9.7.1 **Evaluation of PDILI**

The PDILI IMP discontinuation criteria for this study are provided in Section 6.3.1, with the accompanying required follow-up investigation and monitoring detailed below. All PDILI events must be reported as an AE and reported to the study site and Sponsor within 24 hours of learning of their occurrence. Any PDILI event that meets the criterion for potential Hy's Law must be reported as an AE of special interest (see Section 9.5), and, if applicable, also reported as an SAE (see Section 9.2.1).

Evaluation of PDILI consists of the diagnostic testing and continued monitoring included in Table 9-3 (specific tests dependent on laboratory results and corresponding symptoms) and consultation with a local hepatologist (if applicable; discussed in Section 9.7.1.1). The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist. Additional investigation and monitoring may be required and adapted based on the diagnosis after the cause of the liver injury/abnormality is confirmed (details in Section 9.7.1.4).

The results of all monitoring, including laboratory testing and other testing, should be made available to the study site and sponsor.

All initial tests resulting in abnormal hepatic laboratory values need to be repeated, but appropriate medical action must not be delayed waiting for the repeat result.

If tests are done locally for more rapid results, a concurrent sample should also be sent to the central laboratory whenever possible. Medical care decisions are to be made initially using the most rapidly available results and a conservative approach must be taken if the results from the

<sup>&</sup>lt;sup>a</sup> Pregnancy testing will be done in all women of childbearing potential and will consist of serum testing at the Safety Follow-Up Visit and urine testing at all other visits.

2 laboratory tests are significantly different. Data from the local and central laboratory are to be recorded on the applicable eCRF pages.

Table 9-3 summarizes the

ast to he pation of the sead to support any marketing astructural transfer the sead to support any marketing astructural transfer the sead to support any marketing astructural transfer to the sead to support as th

**Table 9-3:** Required investigations and follow-up for PDILI

| Clinical Study Protocol Table 9-3: Required investigations and follow-up for PDILI | | | | | aidions | |
|---|---|---|---|---|---|---|
| Labora | tory value | Symptoms a of | Imn | nediate | | Follow up |
| ALT or<br>AST | Total<br>bilirubin | hepatitis or<br>hypersensitivity | Consultation requirements | Actions | Testing | Evaluation |
| ≥3xULN | ≥2xULN <sup>b</sup> | NA | Hepatology consult. <sup>c</sup> Medical Monitor must be notified | Immediate, permanent IMP discontinuation. | Essential: Must have repeat liver chemistry values | Monitoring of liver<br>chemistry values at least<br>twice per week until values |
| ≥3xULN | NA | Yes | within 24 hours (eg, by laboratory alert) and subject discussed with Medical Monitor ASAP. | OPT application | and additional<br>testing completed<br>ASAP (see<br>Section 9.7.1.3);<br>recommended to<br>occur at the site | normalize, stabilize, or return to within baseline values. d |
| ≥5xULN | NA | NA | Need for hepatology consult to be discussed (required if ALT or AST ≥8xULN). Medical Monitor must be notified within 24 hours (eg, by laboratory alert) and subject discussed with Medical Monitor ASAP. | TED COPY application | with HCP. | |

Table 9-3: Required investigations and follow-up for PDILI

| Labora | tory value | Symptoms a of | Immediate | | | Follow up |
|---|---|---|---|---|---|---|
| ALT or<br>AST | Total<br>bilirubin | hepatitis or<br>hypersensitivity | Consultation requirements | Actions | Testing rejons | Evaluation |
| ≥3xULN<br>(and ≥2x<br>baseline)<br>and<br><5xULN<br>(and ≥2x<br>baseline) | <2xULN | No | Discussion with Medical Monitor required. Consider need for hepatology consult if there is no evidence of resolution (see Follow up requirements). c | Further investigation – immediate IMP discontinuation not required (see Section 9.7.1.2). IMP discontinuation required if any of the following occur: • Subject cannot comply with monitoring schedule. • Liver chemistry values continue to increase. • Liver chemistry values remain ≥3xULN (and ≥2x baseline) after 2 weeks of monitoring without evidence of resolution. | Essential: Every attempt must be made to have repeat liver chemistry values and additional testing completed within 48 hours at the site with HCP (see Section 9.7.1.3). | Monitoring of liver chemistry values at least twice per week for 2 weeks. d • Immediate IMP discontinuation required if liver chemistry values continue to increase. After 2 weeks of monitoring liver chemistry values: • Discontinue IMP if levels remain ≥3xULN (and ≥2x baseline) without evidence of resolution d • Continue to monitor until values normalize, stabilize, or return to within baseline values. d |

ALT=alanine aminotransferase; ASAP=as soon as possible; AST=aspartate aminotransferase; HCP=healthcare practitioner; IMP=investigational medicinal product; NA=not applicable; PDILI=potential drug-induced liver injury; ULN=upper limit of normal

<sup>&</sup>lt;sup>a</sup> Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative cause).

<sup>&</sup>lt;sup>b</sup> If the subject also has  $\ge 2x$ ULN alkaline phosphatase, the possibility of an indication of biliary obstruction should be discussed with the Medical Monitor.

<sup>&</sup>lt;sup>c</sup> Details provided in Section 9.7 D1. The local hepatologist is the expert usually consulted by the treating physician for assessment and management of potential hepatic disease. This would usually be a hepatologist, but may be a gastroenterologist.

<sup>&</sup>lt;sup>d</sup> Unless an alternative monitoring schedule is agreed by the Investigator and UCB responsible physician. Determination of stabilization is at the discretion of the Investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

### 9.7.1.1 Consultation with Medical Monitor and local hepatologist

Potential drug-induced liver injury events require notification of the Medical Monitor within All PDILI events require immediate action, testing, and monitoring.

The immediate action is dependent on the laboratory values and symptoms of hepatitis or hypersensitivity and ranges from continuation of IMP (followed by immediate investigation) to immediate and permanent discontinuation (see Section 6.3.1 and Table 9-3 for details).

When IMP is discontinued, all concomitant medications and herbor eduction for medically necessary should also be discontinued. The eduction for medically necessary concomination of imperior immediate and permanent discontinued.

### 9.7.1.3 Testing: identification/exclusion of alternative etiology

The measurements and additional information required for the assessment of PDILI events when there is a reasonable possibility that they may have been caused by the IMP include, but are not limited to, those listed in Table 9-4 (laboratory measurements) and Table 9-5 (additional information). Results of the laboratory measurements and information collected are to be submitted to the sponsor on the corresponding eCRF. If the medical history of the subject indicates a requirement for other assessments not included below, these additional assessments should be completed and submitted as applicable.

All blood samples should be stored, if possible. If tests are done locally for more rapid results, a concurrent sample must also be sent to the central laboratory.

.surer, cannot be used to st The laboratory measurements to be assessed are presented in Table 9-4.


### **Table 9-4: PDILI laboratory measurements**

| Virology- | Hepatitis A IgM antibody |
|---|---|
| related | HBsAg |
| | Hepatitis E IgM antibody |
| | HBcAb-IgM |
| | Hepatitis C RNA |
| | Cytomegalovirus IgM antibody |
| | Epstein-Barr viral capsid antigen IgM antibody (if unavailable, obtain heterophile antibody or monospot testing) |
| Immunology | Anti-nuclear antibody (qualitative and quantitative) |
| | Anti-smooth muscle antibody (qualitative and quantitative) |
| | Type 1 anti-liver kidney microsomal antibodies (qualitative and/or quantitative) |
| Hematology | Eosinophil count |
| Urinalysis | Toxicology screen <sup>a</sup> |
| Chemistry | Amylase |
| | If total bilirubin ≥1.5xULN, obtain fractionated bilirubin to obtain % direct bilirubin |
| | Serum CPK and LDH to evaluate possible muscle injury causing transaminase elevation |
| Additional | Prothrombin time/INR <sup>b</sup> |
| | Serum pregnancy test |
| | PK sample |

ALT=alanine aminotransferase; CPK=creatine phosphokinase; HBcAb-IgM=hepatitis B core antibody-IgM; HBsAg=hepatitis B surface antigen; IgM=immunoglobulin M; INR=international normalized ratio; LDH=lactate dehydrogenase; PDILI=potential drug-induced liver injury; PK=pharmacokinetic; RNA=ribonucleic acid; ULN=upper limit of normal

Additional information to be collected is presented in Table 9-5.

For detecting substances (ie, amphetamines, benzodiazepines, opioids, marijuana, cocaine, phencyclidine, and tricyclic antidepressants), additional tests may be performed based on the Investigator's medical judgment and patient's history.

b Measured only for subjects with ALT >8xULN, elevations in total bilirubin, and symptoms of hepatitis or hypersensitivity. Hepatitis symptoms include fatigue, nausea, vomiting, and right upper quadrant pain or hie doci Ada. tenderness; hypersensitivity symptoms include eosinophilia (>5%), rash, and fever (without clear alternative

### PDILI information to be collected **Table 9-5:**

# New or updated information

Concomitant prescription and over-the-counter medications (eg, acetaminophen, herbal remedies, vitamins); dosages and dates should be included.

Pertinent medical history, including the following:

- History of liver disease (eg, autoimmune hepatitis, nonalcoholic steatohepatitis or other "fatty liver disease")
- Adverse reactions to drugs
- Allergies
- Relevant family history or inheritable disorders (eg. Gilbert's syndrome, alpha-1 antitrypsin deficiency)
- Recent travel
- Progression of malignancy involving the liver (Note: Metastatic disease to the liver, by itself, should not be used as an explanation for significant AST and/or ALT elevations.)

The appearance or worsening of clinical symptoms of hepatitis or hypersensitivity (eg., fatigue, nausea, vomiting, right upper quadrant pain or tenderness, decreased appetite, abdominal pain, jaundice, fever, or

Recent clinically significant hypotension or hypoxemia with compromised cardiopulmonary function

Alcohol and illicit drug use

Results of liver imaging or liver biopsy, if done

Results of any specialist or hepatology consult, if done

Any postmortem/pathology reports

ALT=alanine aminotransferase; AST=aspartate aminotransferase; PDILI=potential drug-induced liver injury

### Follow-up evaluation 9.7.1.4

Potential drug-induced liver injury events require follow-up monitoring as described in Table 9-3. Monitoring should continue until liver chemistry values normalize, stabilize, or return to baseline. Determination of stabilization is at the discretion of the investigator in consultation with the hepatologist (as applicable) and UCB responsible physician, as needed.

# Other safety measurements 9.8

### Assessment and management of TB and TB risk factors 9.8.1

At the Baseline Visit of PS0011, all subjects will undergo physical symptoms of TB and must be care? All subjects will be assessed for TB through physical examination for signs and symptoms of

At the Baseline Visit of PS0011, all subjects will undergo physical examination for signs and symptoms of TB and must be confirmed to have undergone an IGRA test (QuantiFERON TB GOLD is recommended) at the Week 8 Visit of PS0010 with negative results. In addition, each subject will complete a TB questionnaire with questions directed at symptoms of TB and potential exposure to TB.

# Exclusion criteria at Baseline of PS0011

Subjects with known TB infection, at high risk of acquiring TB infection, or latent TB infection are excluded.

- a. Known TB infection whether present or past is defined as:
- History of active TB infection involving any organ system or findings in other organ systems consistent with TB infection, unless adequately treated and proven to be finding recovered upon consult with a TB specialist

  Any evidence by radiography or other active TB infection.
  - Any evidence by radiography or other imaging modalities consistent with previously active TB infection that is not reported in the subject's medical history.
- b. High risk of acquiring TB infection is defined as:
  - Known exposure to another person with active TB infection within the 3 months prior to enrollment
  - Time spent in a healthcare delivery setting or institution where individuals infected with TB are housed and where the risk of transmission of infection is high
- c. Latent TB infection is defined as:
  - The absence of signs, symptoms (ie, evidence of organ-specific involvement), or physical findings suggestive of TB infection with a positive IGRA test (or 2 indeterminate IGRA test results) and a chest x-ray (or other imaging) without evidence of TB infection. If the result of the IGRA test is indeterminate, the particular IGRA test previously performed may be repeated once; if positive or indeterminate on retest, the subject may not be enrolled in the study. The retest must be done prior to entry in PS0011.

Note: If available, respiratory or other specimens must also be smear and culture negative for TB (Centers for Disease Control diagnosis of LTB infection) http://www.cdc.gov/TB/topic/testing/default.htm)

d. Current or history of NTMB infection

# Signs and Symptoms

The Investigator should consider all potential sites of infection when assessing for TB during the physical examination and other evaluations, and based on the subject's medical or social history.

The most common primary focus of TB is the lung. Other sites may include GI system, grands and meni grands and meni compared to the normal population.

Some common symptom infection bone/joints, lymph glands and meninges, etc. However, in immune compromised patients and/or patients treated with TNF inhibitors, extrapulmonary manifestations of TB are common

Some common symptoms that the subject may present are dependent on the primary focus of infection and may include cough, blood in sputum, night sweats, lymphadenitis, joint pain/swelling, spinal deformity, headache/confusion, abdominal pain (mimicking inflammatory bowel disease), etc. Unusual presentations should always be considered.

Latent TB infection is defined in the "Exclusion Criteria" above. If the result of the IGRA is indeterminate, the particular IGRA previously performed may be repeated once; if positive or indeterminate on retest, the subject may not be enrolled in the study without further evaluation specified withdrawal procedures. Laboratory diagnosis should be undertaken via mycobacteria culture media (or if available by preferred nucleic acid amplification test such as the Xpert MTB RIF test) and the result must be negative for TB inducing pathogens.

Test Conversion

Tuberculosis test conversion is defined as a positive IGRA result for the current test when previous IGRA test results were negative. All subjects and the current test when stop study drug of the current test wh

stop study drug administration. In case of a TB test conversion, the subject must be considered as having either a suspected new latent or an active TB infection and be promptly referred to an appropriate specialist (eg, pulmonologist, infectious disease specialist) for further evaluation. If test conversion indicates LTB infection, active TB, or NTMB then, per UCB TB working instructions, TB test conversion (confirmed) should be classified adequately, either as due to LTB infection, active TB infection, or NTMB, respectively. Additional assessments (eg. blood tests or IGRA, chest x-rays, or other imaging) should be performed where medically relevant and documented. Such conversions should be reported to the UCB PS function.

# LTB

In case the evaluation by the appropriate specialist indicates a new LTB infection during the study, a prophylactic TB treatment should be initiated and the subject must be withdrawn from the study. Every related action should be discussed in advance with the Medical Monitor.

Once withdrawn from study treatment, subjects should return for the Week 48/Withdrawal Visit, complete all Early Withdrawal Visit assessments, and complete a SFU Visit (20 weeks after the last dose of study medication).

# Active TB or NTMB infection

Subjects who develop active TB or NTMB infection during the study must be withdrawn from the study. The subject must be immediately discontinued from study medication and an Early Withdrawal Visit must be scheduled as soon as possible, but no later than the next scheduled visit. The subject should be encouraged to keep the SFU Visit as specified by the protocol. Treatment should be started immediately.

Note that subjects with history of NTMB or active NTMB infection are excluded from the study regardless of prior or current therapy for this condition.

### 9.8.13 TB assessment by IGRA

During conduct of the study, the TB assessment by IGRA (QuantiFERON TB GOLD is recommended) will be performed at Week 8 of PS0010 and should be repeated at Week 48/Early Withdrawal Visit for all subjects. The test results will be reported as positive, negative, or indeterminate. UCB also recommends that a TB specialist be consulted where TB (latent or active) is suspected or if there are doubts regarding test results. If latent or active TB is identified, the subject must undergo appropriate study-specified withdrawal procedures. In the event of an indeterminate test result, the retest must be done prior to the next visit.

### 9.8.1.2 Chest x-ray for TB

Chest x-ray will be performed in PS0011 only when required to confirm or exclude TB. Any new clinically significant findings post-Baseline on chest x-ray must be documented in the

Ine questionnaire "Evaluation of signs and symptoms of tuberculosis" should be used as a source document. The questionnaire will be completed at the Baseline Visit of PS0011, and at the Week 12, Week 24, Week 36, and Week 48/Withdrawal Visit. The questionnaire will with the identification of subjects who may require therapy for TP ^ "Yes" to the question

the questionnaire at any visit should trigger further careful assessment to determine if subject has LTB or active TB.

Subjects with a latent or active TB infection must be withdrawn from the study.

### 9.8.1.4 TB management

LTB infection and active TB identified during study

During the study, subjects who develop evidence of LTB infection or active TB must immediately stop further administration of study medication and will be referred to an appropriate TB specialist (pulmonologist or infectious disease specialist) for further evaluation. Evidence of LTB infection is defined as the subject's IGRA test converts to positive or indeterminate (and confirmed indeterminate on repeat), or the subject's questionnaire or history and physical indicates that TB infection or exposure may have occurred. Evidence of active TB includes, in addition to the aforementioned tests, signs and symptoms of organ involvement. In either situation, the subject should be carefully assessed by a TB specialist for active TB. Subjects diagnosed with active TB of LTB infection should be withdrawn from the study and receive appropriate TB or prophylaxis therapy.

Any presumptive diagnosis or diagnosis of a TB infection is a reportable event. Confirmed active TB must be reported as an SAE. The Investigator is to complete and submit the TB follow up form provided.

The subject should be transferred to the care of his/her physician and managed according to the best available standard of care. Subjects identified as having converted to active TB during the study must be withdrawn and scheduled to return for the Week 48/Withdrawal Visit as soon as possible, but no later than the next scheduled study visit, and complete all Week 48/Withdrawal Visit assessments.

The subject should be encouraged to complete a SFU Visit (20 weeks after the last dose of study medication).

If infection with NTMB is identified during the study, the same procedure as for active TB acquired during the study must be followed.


### 9.8.2 **Pregnancy testing**

Pregnancy testing will consist of serum testing at the SFU Visit and urine testing at all other visits.

The Baseline Visit urine pregnancy test result must be negative prior to enrollment of the subject. A negative urine pregnancy test result should be obtained immediately prior to each administration of study drug and at all subsequent visits. Pregnancy tests should be administered to all female subjects of children to all female subjects of childbearing potential, regardless of their use of birth control.

### 9.8.3 Vital signs

Vital signs will be collected at every visit and will include systolic and diastolic blood pressure, pulse rate, and body temperature (oral, axillary, or otic). Subjects should be sitting for 5 minutes before and during vital signs assessments.

Vital signs are to be measured prior to blood sampling, and prior to dosing, where applicable.

Body weight will be measured at the time points specified in the schedule of study assessments (Table 5–1).

### 12-lead ECGs 9.8.4

Twelve-lead standard ECGs will be recorded at the visits specified in Table 5–1, and read by a central ECG laboratory.

Full details of ECG recording will be provided in the ECG Manual.

### **Physical examination** 9.8.5

The physical examination will include general appearance; ear, nose, and throat; eyes, hair, and skin; respiratory; cardiovascular; GI; musculoskeletal; hepatic; neurological (including limb reflexes); and mental status. Physical examination will be performed at the at the time points specified in the schedule of study assessments (Table 5–1). Findings considered clinically significant changes since the physical examination at the Screening Visit of PS0010 will be recorded as AEs.

### 9.8.6 Assessment of suicidal ideation and behavior

Suicidal ideation and behavior will be assessed by trained study personnel using the eC-SSRS. This scale will be used to assess suicidal ideation and behavior that may occur during the study. The visits at which the eC-SSRS assessments will be performed are specified in the schedule of study assessments (Table 5–1).

The eC-SSRS is a standardized and validated instrument developed for the assessment of the severity and frequency of suicidal ideation and behavior (Mundt et al., 2010; Posner et al., 2011). defines five subtypes of suicidal ideation and behavior in addition to self-injurious behavior with no suicidal intent. The eC-SSRS takes approximately 3 to 10 minutes to complete.

Refer to Section 6.3 for eCSSRS-related withdrawal criteria

### 9.8.7 **Data Monitoring Committee**

The DMC membership includes clinicians knowledgeable about the disease or the treatment. The DMC will include a statistician, and at a minimum, specialists in dermatology and infectious

disease. All members have experience and expertise in clinical trials. Board members may not participate in the study as principal or co-Investigators, or as study subject care physicians. The duration of membership for the DMC will be inclusive of planned analyses for PS0011. The

The DMC procedures will ensure that data remain blind to the study team and Investigators at all times throughout the conduct of the study.

A Cardiovascular Adjudication Committee will also restaudy. Details will be described.

### ASSESSMENT OF PHARMACOKINETIC VARIABLES 10

Blood samples for measurement of PK (Section 4.2) will be collected at the time points specified in the schedule of study assessments (Table 5–1).

At dosing visits, blood samples will be drawn prior to dosing, and will be drawn at the same time of the sampling for clinical laboratory tests. The time and date of collection will be recorded in the eCRF.

Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the laboratory manual for this study. Detailed information on sample analysis will be provided in a bioanalytical report.

### **ASSESSMENT OF IMMUNOLOGICAL VARIABLES** 11

Blood samples for measurement of antibodies to bimekizumab will be collected at the visits specified in Table 5–1. The threshold for antibody positivity will be defined prior to analysis.

At dosing visits, blood samples will be drawn prior to dosing, and will be drawn at the same time of the sampling for clinical laboratory tests. The time and date of collection will be recorded in the eCRF.

Instructions pertaining to sample collection, processing, storage, labeling, and shipping are provided in the laboratory manual for this study. The presence of antibodies to bimekizumab will be determined using a validated bioanalytical method. Detailed information on sample analysis will be provided in a bioanalytical report.

# XSSESSMENT OF EFFICACY 12

### **Psoriasis Area and Severity Index** 12.1

The PASI is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies (Feldman, 2004). The PASI quantifies the severity and extent of the disease and weighs these with the percentage of BSA involvement.

The degree of involvement is estimated across 4 body areas; head, upper limbs, trunk, and lower limbs and then transferred into a grade (Table 12–1).

The Investigator assesses the average redness, thickness, and scaliness of lesions in each body area (each on a 5-point scale); 0=none, 1=slight, 2=moderate, 3=marked, and 4=very marked.


The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity.

Table 12–1: Body areas for calculation of percent BSA for PASI

| Body area | Details of area | BSA | Degree of involvement of body area <sup>a</sup> |
|---|---|---|---|
| Head | Face, back of head | 10% | 0 to 6 |
| Upper limbs | Left, right, upper lower, flexor surface, extensor surface | 20% | 0 to 6 |
| Trunk | Front, back, groin | 30% | 0 to 6 |
| Lower limbs | Left, right, upper lower, flexor surface, extensor surface, including buttocks | 40% | 0 to 6 tension |
| Total | | 100% | del |

BSA=body surface area; PASI=Psoriasis Area and Severity Index

The PASI50, PASI75, PASI90, and PASI100 responses are based on at least 50%, 75%, 90%, and 100% improvement in the PASI score. The improvement will be based on changes from the PASI score at the Baseline of PS0010.

The PASI will be completed at the visits specified in Table 5–1.

# 12.2 Investigator's Global Assessment

A static IGA for psoriasis will be used to assess disease severity in all subjects during the study. The IGA will be completed at the visits specified in Table 5–1.

The Investigator will assess the overall severity of psoriasis using the following 5-point scale:

| 5 point In | 5 point Investigator's Global Assessment | |
|---|---|---|
| Score | Short Descriptor | Detailed Descriptor |
| 0 | Clear Suppor | No signs of psoriasis; post-inflammatory hyperpigmentation may be present |
| 1 | Almost clear | No thickening; normal to pink coloration; no to minimal focal scaling |
| 2 | Mild | Just detectable to mild thickening; pink to light red coloration; predominately fine scaling |
| 3 | Moderate | Clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling |
| Aeril | Severe | Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions |

<sup>&</sup>lt;sup>a</sup> Where 0=none; 1=1% to <10% affected, 2=10% to <30% affected, 3=30% to <50% affected, 4=50% to <70% affected, 5=70% to <90% affected, 6=90% to 100% affected.

### 12.3 **Dermatology Life Quality Index**

The DLOI is a questionnaire designed for use in adult subjects with psoriasis. The DLOI is a skin ocen shown to be valid and reproducible in psoriasis patients. The DLQI score ranges from 0 to 30 with higher scores indicating lower health related QOL. A 5-point change in the DLQI score (DLQI response) has been reported to be meaningful for the patient (within-patient minimal important difference); while a DLQI absolute score of 0 or 1 in 1 in impact of the disease on health related QQL. disease-specific questionnaire aimed at the evaluation of how symptoms and treatment affect outlined in the Schedule of Study Assessments (Table 5–1). Study site personnel should ensure

The BSA palm method will be used for the evaluation of BSA as follows:

Body surface area estimation uses the palm (subject's Given included) as representing palms)

palms)

runk=30% (30 palms)

Lower extremities=40% (40 palms)

Total BSA=100%

luation of BSA will be completed at a strength of the part of t Body surface area estimation uses the palm (subject's flat hand and thumb together, fingers

**UCB** 

Evaluation of BSA will be completed at the visits specified in Table 5–1.

# 12.5

Psoriatic nail disease will be evaluated at the Baseline Visit of PS0010 using the mNAPSI. All affected nails will be scored (0 to 3) for onycholysis/oil drop dyschromia, nail plate crumbling, and pitting and will be scored (0 for "no" or 1 for "yes") for leukonychia, nail bed hyperkeratosis, splinter haemorrhages and red spots in the lunula. The score for an individual nail ranges from 0 to 13 with higher scores indicative of more severe nail disease. The total mNAPSI score is the sum of the scores for each individual nail. If a nail is unaffected, it will be recorded as such and will not contribute to the total mNAPSI score. Subjects with nail disease at Baseline are defined as those with an mNAPSI score >0 at Baseline of PS0010.

The mNAPSI will be assessed at the visits specified in Table 5–1.

# **Psoriasis Scalp Severity Index**

(His docurate) The PSSI considers both the extent of the area of involvement and the severity based on the scoring scales outlined in Table 12–2. The assessment considers erythema, induration, and desquamation on the scalp. For each of these 3 elements, the scores of the area and severity are multiplied. Then, the score from each element is totaled to obtain the PSSI score. As with the

PASI, the PSSI score ranges from 0 to 72 with a higher score indicating increased scalp disease severity.

The PSSI will be assessed at the visits specified in Table 5–1.

Table 12-2: Parameters assessed for the PSSI

| Assessment of extent of scalp psoriasis | |
|-----------------------------------------|-----------------------------|
| Score | Definition |
| 1 | <10% |
| 2 | 10-29% |
| 3 | 30-49% |
| 4 | 50-69% |
| 5 | 70-89% |
| 6 | 90-100% |
| Assessme | ent of clinical symptoms |
| (erythema, ind | luration, and desquamation) |
| Score | Definition |
| 0 | Absent |
| 1 | Slight |
| 2 | Moderate |
| 3 | Severe |
| 4 | Severest possible |

PSSI=Psoriasis Scalp Severity Index

# 12.7 PGADA for the arthritis VAS

The PGADA for the arthritis VAS will be used to provide an overall evaluation of arthritis disease symptoms. Subjects will respond to the question, "Considering all the ways your arthritis affects you, please mark a vertical line on the scale below to show how you are feeling today," using a VAS where 0 is "very good, no symptoms" and 100 is "very poor, severe symptoms."

Each subject will complete the PGADA at the visits specified in Table 5–1.

# 12.8 36-Item Short Form Health Survey

The SF-36 (Version 2, standard recall) is a 36-item generic health-related QOL instrument that uses a recall period of 4 weeks. Items are grouped into 8 domains as follows: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items), and 1 item for perceived stability or change in health (Health Transition) during the last year. The concepts represented by these domains contribute to physical, mental, and social aspects of health-related QOL. In addition to domain scores, the PCS and MCS scores are calculated from the 8 domains (excluding the Health Transition item). Component scores

appreciate the impact of each domain on physical and mental health status (Maruish, 2011). Each of the 8 domain scores and the component summary scores range from 0 to 100, with a higher ions or variations thereof score indicating a better health status. The domains and the 2 component summary scores are standardized with a mean of 50 and a standard deviation of 10 in the general USA population. The minimally important differences, in terms of T-score points, for SF-36 domains and component summaries are as follows: PCS, 2; MCS, 3; Physical Functioning, 3; Role-Physical, 3; Bodily Pain, 3; General Health, 2; Vitality, 2; Social Functioning, 3; Role-Emotional, 4; and Mental Health, 3 (Maruish, 2011).

The SF-36 will be completed by the subject the visits specified in Table 5–1.

### 12.9 **Hospital Anxiety and Depression Scale**

The HADS was chosen for its well-established psychometric properties and its use in clinical research on biological therapy in subjects with chronic plaque psoriasis (Dauden et al, 2009; Langley et al, 2010). The HADS scores for anxiety and for depression range from 0 to 21 with higher scores indicating worse state. A score below 8 is considered to be normal (Snaith and Zigmond, 1994).

### STUDY MANAGEMENT AND ADMINISTRATION 13

### 13.1 Adherence to protocol

The Investigator should not deviate from the protocol. However, the Investigator should take any measure necessary in deviation from or not defined by the protocol in order to protect clinical study subjects from any immediate hazard to their health and safety. In this case, this action should be taken immediately, without prior notification of the regulatory authority, IRB/IEC, or Sponsor.

After implementation of such measure, the Investigator must notify the Clinical Project Manager of the Sponsor within 24 hours and follow any local regulatory requirements.

### 13.2 **Monitoring**

UCB (or designee) will monitor the study to meet the Sponsor's monitoring Standard Operating Procedures (SOPs), ICH-GCP guideline, and applicable regulatory requirements, and to ensure that study initiation, conduct, and closure are adequate. Monitoring of the study may be delegated by UCB to a CRO or a contract monitor.

The Investigator and his/her staff are expected to cooperate with UCB (or designee) and to be available during the monitoring visits to answer questions sufficiently and to provide any missing information. The Investigator(s)/institution(s) will permit direct access to source data/documents for study-related monitoring, audits, IRB/IEC review, and regulatory inspection(s).

The Investigator will allow UCB (or designee) to periodically review all eCRFs and corresponding source documents (eg, hospital and laboratory records for each study participant). Monitoring visits will provide UCB (or designee) with the opportunity to evaluate the progress of the study, verify the accuracy and completeness of eCRFs, ensure that all protocol requirements, applicable authorities regulations, and Investigator's obligations are being fulfilled, and resolve any inconsistencies in the study records.

# 13.2.1 Definition of source data

All source documents must be accurate, clear, unambiguous, permanent, and capable of being audited. Source documentation should be made using some permanent form of recording (ink, typing, printing, optical disc). They should not be obscured by correction fluid or have temporary attachments (such as removable self-stick notes). Photocopies of eCRFs are not considered acceptable source documents. Source documents are original records in which raw data are first recorded. These may include hospital/clinic/general practitioner records, charts, diaries, x-rays, laboratory results, printouts, pharmacy records, care records, ECG or other printouts, completed scales, or QOL questionnaires, for example. Source documents should be kept in a secure.

The Sponsor or designee will review to ensure that computerized source documents produced by the site are compliant with Food and Drug Administration (FDA) Part 11 requirements and document appropriately. Source documents that are computer generated and stored electronically that are not FDA Part 11 compliant, must be printed for review by the monitor (eg, ECG reports). Once printed, these copies should be signed and dated by the Investigator and become a permanent part of the subject's source documents. The Investigator will facilitate the process for enabling the monitor to compare the content of the printout and the data stored in the computer to ensure all data are consistent.

Electronic data records, such as Holter monitor records or electroencephalogram records, must be saved and stored as instructed by the Sponsor or designee.

Patient Reported Outcome (PRO) measures (eg, DLQI, SF-36, and PGADA) will be completed by each subject utilizing electronic data capture.

# 13.2.2 Source data verification

Source data verification ensures accuracy and credibility of the data obtained. During monitoring visits, reported data are reviewed with regard to being accurate, complete, and verifiable from source documents (eg, subject files, recordings from automated instruments, tracings [ECG], x-ray films, laboratory notes). All data reported on the eCRF should be supported by source documents, unless otherwise specified in Section 13.2.1.

# 13.3 Data handling

# 13.3.1 eCRF completion

This study will use electronic data capture (EDC); the Investigator is responsible for prompt reporting of accurate, complete, and legible data in the eCRF and in all required reports.

This study will use an electronic device to capture patient reported outcomes (see Section 13.2.1).

Serious AE reporting will be done using the SAE Form (see Section 9.2.2) while also entering the event in the appropriate eCRF section. The safety database and the clinical database will be reconciled during the study and discrepancies will be corrected as needed.

The Investigator should maintain a list of personnel authorized to enter data into the eCRF. Access to the EDC will be given after training has been received. A training certificate will be provided and filed.

Detailed instructions on the use of the EDC will be provided in the eCRF Completion Guidelines.

Database entry and reconciliation

Case Report Forms/external electronic data will be entered/loaded into a validated electronic database using a clinical data management system. Computerized data cleaning checks will used in addition to manual review to check for discrepancies and to analyte data. This study is performed using EDC: the database using a clinical data management system.

An electronic audit trail system will be maintained to track all data changes in the database once the data have been saved initially into the system or electronically loaded. Regular backups of the electronic data will be performed.

### 13.3.3 Subject Enrollment log/Subject Identification Code list

The subject's enrollment will be recorded in the Subject Enrollment Log.

The Investigator will keep a Subject Identification Code list. This list remains with the Investigator and is used for unambiguous identification of each subject.

The subject's consent and enrollment in the study must be recorded in the subject's medical record. These data should identify the study and document the dates of the subject's participation.

### Termination of the study 13.4

UCB reserves the right to temporarily suspend or prematurely discontinue this study either at a single site, multiple sites, or at all sites at any time for reasons including, but not limited to, safety or ethical issues, inaccurate or incomplete data recording, noncompliance, or unsatisfactory enrollment with respect to quality or quantity.

If the study is prematurely terminated or suspended, UCB (or its representative) will inform the Investigators/institutions and the regulatory authority(ies) of the termination or suspension and the reason(s) for the termination or suspension, in accordance with applicable regulatory requirement(s). The IRB/IEC should also be informed and provided with reason(s) for the termination or suspension by the Sponsor or by the Investigator/institution, as specified by the applicable regulatory requirement(s). In addition, arrangements will be made for the return of all unused MP and other material in accordance with UCB procedures for the study.

# 13:5<sup>5</sup> Archiving and data retention

The Investigator will maintain adequate records for the study, including eCRFs, medical records, laboratory results, Informed Consent documents, drug dispensing and disposition records, safety reports, information regarding participants who discontinued, and other pertinent data.

All essential documents are to be retained by the Investigator until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or at least 2 years have elapsed since the formal discontinuation of clinical development of the IMP. These documents should be retained for a longer period, however, if required by the applicable regulatory requirement(s) or by an agreement with UCB (Committee for Proprietary Medicinal Products [CPMP]/ICH/135/95, 2002 [Section 4.9.5]). The Investigator will contact UCB for authorization prior to the destruction of any study records or in the event of accidental loss or destruction of any study records. The Investigator will also notify UCB should he/she relocate or move the study-related files to a location other than that specified in the Sponsor's study master file.

Bimekizumab

# 13.6 Audit and inspection

The Investigator will permit study-related audits mandated by UCB, after reasonable notice, and inspections by domestic or foreign regulatory authorities.

The main purposes of an audit or inspection are to confirm that the rights and well-being of the subjects enrolled have been protected, that enrolled subjects (ie, signing consent and undergoing study procedures) are appropriate for the study, and that all data relevant for the evaluation of the IMP have been processed and reported in compliance with the planned arrangements, the protocol, investigational site, and IRB/IEC SOPs, ICH GCP, and applicable regulatory requirements.

The Investigator will provide direct access to all study documents, source records, and source data. If an inspection by a regulatory authority is announced the Investigator will immediately inform UCB (or designee).

# 13.7 Good Clinical Practices

Noncompliance with the protocol, ICH-GCP, or local regulatory requirements by the Investigator, institution, institution staff, or designees of the Sponsor will lead to prompt action by UCB to secure compliance. Continued noncompliance may result in the termination of the site's involvement in the study.

# 14 STATISTICS

A description of statistical methods is presented below and will be described in more detail in the Statistical Analysis Plan (SAP).

# 14.1 Definition of analysis sets

The Enrolled Set (ES) will consist of all subjects who have given informed consent for PS0011.

The Safety Set (\$\section{S}\$) will consist of all subjects who receive at least 1 dose of the study medication in PS0011.

The Full Analysis Set (FAS) will consist of all enrolled subjects who receive at least 1 dose of the study medication in PS0011 and have a valid efficacy measurement for PASI at Baseline of PS0011.

The Pharmacokinetics Per-Protocol Set (PK-PPS) will consist of all enrolled subjects who receive at least 1 dose of the study medication in PS0011 and provide at least 1 quantifiable plasma concentration postdose in PS0011.

### 14.2 General statistical considerations

No inferential statistical analyses are planned for this extension study. Instead, all variables will be presented using summary statistics. For categorical variables, counts and percentages will be

Because subjects entering PS0011 may or may not be continuing on the same dose as that received in PS0010, there are various combinations of treatment that could be received when considering both PS0010 and PS0011 together. For describing the summaries to be produced treatment groups will be categorized as either the PS0011 treatment are treatment groups. These categorizations are outlined.

# **PS0011 treatment groups**

This refers to the study treatment assigned to the subject at the beginning of PS0011 and does not account for the treatment received in PS0010. The PS0011 treatment groups are as follows:

- Placebo
- Bimekizumab 64mg Q4W
- Bimekizumab 160mg Q4W
- Bimekizumab 320mg Q4W
- All Bimekizumab (optional to be used only if specified)

# PS0010/PS0011 treatment groups

This refers to the combination of the randomized treatment in PS0010 and the treatment assigned at the beginning of PS0011. Some groups have been combined where it is considered appropriate to do so. The PS0010/PS0011 treatment groups with descriptions are as follows:

- Placebo to Placebo Subjects randomized to placebo in PS0010 who achieve PASI90 response at Week 12 of PS0010 and continue to receive placebo in PS0011.
- Placebo to Bimekizumab 160mg Q4W Subjects randomized to placebo in PS0010 who do not achieve PASI90 response at Week 12 of PS0010 and are treated with bimekizumab 160mg Q4W in PS0011.
- Bimekizumab 64mg to Bimekizumab 64mg Subjects randomized to bimekizumab 64mg Q4W in PS0010 who achieve PASI90 response at Week 12 of PS0010 and continue to receive bimekizumab 64mg O4W in PS0011.
- Bimekizumab 64mg to Bimekizumab 160mg Subjects randomized to bimekizumab 64mg Q4W in PS0010 who do not achieve PASI90 response at Week 12 of PS0010 and are treated with bimekizumab 160mg Q4W in PS0011.
- Bimekizumab 160mg Q4W to Bimekizumab 160mg Q4W Subjects randomized to bimekizumab 160mg Q4W or bimekizumab 320mg loading dose + 160mg Q4W in PS0010 who achieve PASI90 response at Week 12 of PS0010 and continue to receive bimekizumab

160mg Q4W in PS0011. Note that the PS0010 160mg Q4W groups with and without the loading dose are combined here.

- Bimekizumab 160mg Q4W to Bimekizumab 320mg Q4W Subjects randomized to bimekizumab 160mg Q4W or bimekizumab 320mg loading dose + 160mg Q4W in PS0010 who do not achieve PASI90 response at Week 12 of PS0010 and are treated with bimekizumab 320mg Q4W in PS0011. Note that the PS0010 160mg Q4W groups with and without the loading dose are combined here.
   Bimekizumab 320mg Q4W to Bimekizumab 320mg Q4W.
- Bimekizumab 320mg Q4W to Bimekizumab 320mg Q4W Subjects randomized to bimekizumab 320mg Q4W in PS0010 and continue on 320mg Q4W in PS0011. No distinction will be made between subjects that were or were not PASI90 responders at Week 12 of PS0010.
- Bimekizumab 480mg Q4W to Bimekizumab 320mg Q4W Subjects randomized to bimekizumab 480mg Q4W in PS0010 and continue on 320mg Q4W in PS0011. No distinction will be made between subjects that were or were not PASI90 responders at Week 12 of PS0010.

The treatment groups to be used in the presentations of safety and efficacy will depend on the objective of the summaries and will be specified accordingly.

# 14.3 Planned safety analyses

Safety variables will be analyzed for all subjects in the SS.

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA®). Treatment-emergent AEs will be defined as events that have a start date on or following the first administration of study treatment in PS0011 through the final administration of study treatment +140 days (covering the 20-week SFU Period). Treatment-emergent AEs will be categorized by PS0011 treatment group. Tables will include columns for placebo, bimekizumab 64mg Q4W, bimekizumab 160mg Q4W, bimekizumab 320mg, and All bimekizumab (ie, any dose of bimekizumab).

# 14.3.1 Primary safety analysis

All TEAEs will be summarized descriptively by PS0011 treatment group, primary SOC, high level term (HLT), and preferred term (PT). This summary will include the exposure adjusted incidence rate (EAIR) with associated 95% confidence interval and the exposure adjusted event rate (EAER).

For EAIR, the numerator will be the total number of subjects experiencing the AE. The denominator will be 100 subject-years; that is, the total summation of individual subject-years at risk up to the first occurrence of the AE for subjects with that AE, and the total subject-years at risk for those subjects not experiencing that AE, divided by 100. Exposure adjusted incidence rates will be presented with a 95% exact confidence interval based upon the Chi-Square distribution (Ulm, 1990).

For EAERs, the numerator will be the number of AEs including repeat occurrences in individual subjects; the denominator will be 100 subject-years. That is, the total summation of individual subject-years at risk divided by 100. No confidence interval will be computed for EAER.

Patient exposure at risk in days will be defined as date of last administration of study medication - date of first administration of study medication in PS0011 + 140 days (ie, the duration of the lations thereof SFU Period). If a subject dies, patient exposure at risk is censored at the date of death. The sum of these exposure days at risk across subjects is converted to years for the EAIR and EAER calculations described above.

### 14.3.2 Other safety analyses

Additional tables will summarize TEAEs by intensity and relationship to study medication, TEAEs leading to withdrawal from the study, treatment-emergent SAEs, and deaths. Other AE summaries to be included will be specified in the SAP. All AE tables will be presented by PS0011 treatment group (including the All bimekizumab group).

Extent of exposure to study medication in PS0011 will be summarized using descriptive statistics by PS0011 treatment group.

Change from Baseline in laboratory values, ECGs, and vital signs will be presented using descriptive statistics by PS0010/PS0011 treatment group. As these variables are summarized over time and the initial values can be impacted by the randomized treatment in PS0010, the presentation by PS0010/PS0011 treatment group is intended to provide perspective on the change in these values starting with the initial PS0010 randomization through the 48-week Treatment Period of PS0011. The table presentations will display descriptive statistics for the PS0010 Baseline followed by descriptive statistics for the observed, change from PS0010 Baseline, and change from PS0011 results by scheduled visit for PS0011.

### Planned PK analyses 14.4

14.4 Planned PK analyses
Pharmacokinetic variables will be analyzed for all subjects in the PK-PPS.

Bimekizumab plasma concentrations will be summarized by PS0010/PS0011 treatment group at each scheduled visit. Descriptive statistics for the plasma concentrations at PS0010 Baseline will be presented followed by descriptive statistics for the observed, change from PS0010 Baseline, and change from PS0011 Baseline results for scheduled visits in PS0011. Summarizing in this manner based on the PS0010/PS0011 treatment group will allow for an evaluation of how changing doses (where applicable) impacted plasma concentrations relative to both the original (PS0010) Baseline as well as the new (PS0011) Baseline. For the descriptive statistics, geometric mean, geometric coefficient of variation, and 95% confidence interval for the geometric mean will be used instead of the arithmetic mean and standard deviation.

# Planned immunological analyses 14.5

Immunological variables will be analyzed for all subjects in the PK-PPS.

Anti-bimekizumab antibody data will be summarized by PS0010/PS0011 treatment group at each scheduled visit. The summary of anti-bimekizumab antibody levels will follow a similar approach to that used for the summary of bimekizumab plasma concentrations. Additional analyses related to antibody positivity will be performed and will be described in greater detail in the SAP.

### 14.6 Planned efficacy analyses

Efficacy variables will be summarized based on the FAS. The summaries described in this section will provide data on maintenance of effect of study treatment over 48 weeks.

Responder efficacy variables (PASI75, PASI90, PASI100, IGA, and DLQI score of 0 or 1) will be summarized descriptively using counts and percentages by scheduled visit and PS0010/PS0011 treatment group. The PASI responder variables will be derived relative to both the PS0010 Baseline and the PS0011 Baseline with responder rates being presented side-by-side in applicable summary tables. Missing data will be handled by using nonresponder imputation (NRI), meaning that subjects that discontinue early or who have missing data at a given time point are imputed as though they did not achieve the given response. Supportive summaries will be based on observed case data.

Continuous efficacy variables based on the change from Baseline (PASI, DLQI, BSA, mNAPSI, PSSI, PGADA, SF-36, and HADS) will be summarized using descriptive statistics by scheduled visit and PS0010/PS0011 treatment group. The table presentations will display descriptive statistics for the PS0010 Baseline, followed by descriptive statistics for the observed, change from PS0010 Baseline, and change from PS0011 Baseline results by scheduled visit for PS0011. Figures for selected variables will also be generated in order to demonstrate the kinetics of response over time. Missing data will be handled by using multiple imputation (MI) via the Markov-Chain Monte Carlo (MCMC) method. Supportive summaries will be based on observed case data.

# 14.7 Planned interim analysis and data monitoring

A DMC will review the safety data on a recurring basis as outlined in the DMC charter. In addition to these ongoing reviews, an analysis combining safety data from PS0010 and PS0011 will be performed when the PS0010 study database is locked. This analysis will account for data in PS0010 as well as the accrued safety data in PS0011 available at the time of the PS0010 database lock. At the time of the interim analysis, the DMC will be unblinded; however, the Sponsor study team will remain blind. The details of this combined safety analysis of PS0010 and PS0011, including the events of interest to be considered, will be outlined in the DMC charter.

# 14.8 Determination of sample size

Up to 240 subjects are anticipated to enroll in PS0011. This number is based on the fact that 240 subjects are planned to be randomized in the feeder study, PS0010. The calculations to reach that sample size are outlined in the PS0010 protocol. As the primary objective of this study is to assess the long-term safety and tolerability of bimekizumab 320mg Q4W, the number of subjects anticipated is based on the number of subjects completing PS0010 and meeting eligibility requirements for PS0011.

# 15 ETHICS AND REGULATORY REQUIREMENTS

# 15.1 Informed consent

Subject's informed consent must be obtained and documented in accordance with local regulations, ICH-GCP requirements, and the ethical principles that have their origin in the principles of the Declaration of Helsinki.

Prior to obtaining informed consent, information should be given in a language and at a level of complexity understandable to the subject in both oral and written form by the Investigator (or designee). Each subject will have the opportunity to discuss the study and its alternatives with the Investigator.
Prior to participation in the study, the written Informed Consent Form should be signed and personally dated by the subject and by the person who conducted the informed consent discussion (Investigator or designee). The subject must receive a copy of the signed and dated If the Informed Consent Form is amended during the study, the Investigator (or the Sponsor, if applicable) must follow all applicable regulatory requirements pertaining to the approval of the amended Informed Consent Form by the IRB/IEC and use of the amended IRB/IEC and use of the amended IRB/IEC and use

All studies conducted at centers in the United States must include the use of a Health Insurance Portability and Accountability Act Authorization form.

The subject may withdraw his/her consent to participate in the study at any time. A subject is considered as enrolled in the study when he/she has signed the Informed Consent Form. An eCRF must not be started, nor may any study specific procedure be performed for a given subject, without having obtained his/her written consent to participate in the study.

#### 15.2 Subject identification cards

Upon signing the Informed Consent, the subject will be provided with a subject identification card in the language of the subject. The Investigator will fill in the subject identifying information and medical emergency contact information. The Investigator will instruct the subject to keep the card with him/her at all times.

#### 15.3 **IRBs and IECs**

The study will be conducted under the auspices of an IRB/IEC, as defined in local regulations, ICH-GCP, and in accordance with the ethical principles that have their origin in the Declaration of Helsinki.

The Investigator/UCB will ensure that an appropriately constituted IRB/IEC that complies with the requirements of the current ICH-GCP version or applicable country-specific regulations will be responsible for the initial and continuing review and approval of the clinical study. Prior to initiation of the study, the Investigator/UCB will forward copies of the protocol, Informed Consent Form, IB, Investigator's curriculum vitae (if applicable), advertisement (if applicable), and all other subject-related documents to be used for the study to the IRB/IEC for its review and approval.

Before initiating a study, the Investigator will have written and dated full approval from the responsible IRB/IEC for the protocol.

The Investigator will also promptly report to the IRB/IEC all changes in the study, all unanticipated problems involving risks to human subjects or others, and any protocol deviations, to eliminate immediate hazards to subjects.

The Investigator will not make any changes in the study or study conduct without IRB/IEC approval, except where necessary to eliminate apparent immediate hazards to the subjects. For minor changes to a previously approved protocol during the period covered by the original approval, it may be possible for the Investigator to obtain an expedited review by the IRB/IEC as allowed.

As part of the IRB/IEC requirements for continuing review of approved studies, the Investigator will be responsible for submitting periodic progress reports to the IRB/IEC (based on IRB/IEC requirements), at intervals appropriate to the degree of subject risk involved, but no less than once per year. The Investigator should provide a final report to the IRB/IEC following study completion.

UCB (or its representative) will communicate safety information to the appropriate regulatory authorities and all active Investigators in accordance with applicable regulatory requirements. The appropriate IRB/IEC will also be informed by the Investigator or the Sponsor, as specified by the applicable regulatory requirements in each concerned country. Where applicable, Investigators are to provide the Sponsor (or its representative) with evidence of such IRB/IEC notification.

#### 15.4 Subject privacy

UCB staff (or designee) will affirm and uphold the subject's confidentiality. Throughout this study, all data forwarded to UCB (or designee) will be identified only by the subject number assigned at Screening.

The Investigator agrees that representatives of UCB, its designee, representatives of the relevant IRB/IEC, or representatives of regulatory authorities will be allowed to review that portion of the subject's primary medical records that directly concerns this study (including, but not limited to, laboratory test result reports, ECG reports, admission/discharge summaries for hospital admissions occurring during a subject's study participation, and autopsy reports for deaths occurring during the study).

#### Protocol amendments 15.5

Protocol changes may affect the legal and ethical status of the study and may also affect the statistical evaluations of sample size and the likelihood of the study fulfilling its primary objective.

Significant changes to the protocol will only be made as an amendment to the protocol and must be approved by UCB, the IRB/IEC, and the regulatory authorities (if required), prior to being implemented.

#### FINANCE, INSURANCE, AND PUBLICATION 16

Insurance coverage will be handled according to local requirements.

Finance, insurance, and publication rights are addressed in the Investigator and/or CRO agreements, as applicable.

# **REFERENCES**

Augustin M, Glaeske G, Radtke MA, Christophers E, Reich K, Schäfer I. Epidemiology and

Christophers E, Barker JN, Griffiths CF David Topographic Control Cont Christophers E, Barker JN, Griffiths CE, Daudén E, Milligan G, Molta C, et al. The risk of psoriatic arthritis remains constant following initial diagnosis of psoriasis among patients seen in European dermatology clinics. J Eur Acad Dermatol Venereol. 2010;24:548-54.

Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0. National Institutes of Health, National Cancer Institute, Division of Cancer Treatment and Diagnosis. http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm. Updated

Dauden E, Griffiths CE, Ortonne JP, Kragballe K, Molta CT, Robertson D, et al. Improvements in patient-reported outcomes in moderate-to-severe psoriasis patients receiving continuous or paused etanercept treatment over 54 weeks: the CRYSTEL at 1

Dowlatshahi EA, Wakkee M, Arends LR, Nijsten T. The prevalence and odds of depressive symptoms and clinical depression in psoriasis patients: a systematic review and meta-analysis. J Invest Dermatol. 2014;134:1542-51.

Feldman SR. A quantitative definition of severe psoriasis for use in clinical trials. J Dermatolog Treat. 2004;15(1):27-9.

Gelfand JM, Neimann AL, Shin DB, Wang X, Margolis DJ, Troxel AB. Risk of myocardial infarction in patients with psoriasis. JAMA. 2006;296:1735-41

Gisondi P, Tessari G, Conti A, Piaserico S, Schianchi S, Peserico A, et al. Prevalence of metabolic syndrome in patients with psoriasis: a hospital-based case-control study. Br J Dermatol. 2007;157:68-73.

Gottlieb AB. Psoriasis: Emerging therapeutic strategies. Nat Rev Drug Discov. 2005;4:19-34.

Icen M, Crowson CS, McEvoy MT, Dann FJ, Gabriel SE, Maradit Kremers H. Trends in incidence of adult-onset psoriasis over three decades: a population-based study. J Am Acad Dermatol. 2009;60:394-401.

Krueger G, Ellis CN. Psoriasis—recent advances in understanding its pathogenesis and treatment. J Am Acad Dermatol. 2005;53(1 Suppl 1):S94-100.

Krueger G, Koo J, Lebwohl M, Menter A, Stern RS, Rolstad T. The impact of psoriasis on quality of Life. Results of a 1998 National Psoriasis Foundation patient-membership survey. Arch Dermatol. 2001;137:280-4.

Kurd SK, Smith N, Van Voorhees A, Troxel AB, Badmaev V, Seykora JT, et al. Oral curcumin in the treatment of moderate to severe psoriasis vulgaris: a prospective clinical trial. J Am Acad Dermatol. 2008;58:625-31.

Kurd SK Gelfand JM. The prevalence of previously diagnosed and undiagnosed psoriasis in US adults: results from NHANES 2003-2004. J Am Acad Dermatol. 2009;60:218-24.

Langley RG, Krueger GG, Griffiths CEM. Psoriasis: epidemiology, clinical features, and quality of life. Ann Rheum Dis. 2005;64(Suppl II):ii18–ii23.

Langley RG, Feldman SR, Han C, Schenkel B, Szapary P, Hsu MC, et al. Ustekinumab significantly improves symptoms of anxiety, depression, and skin-related quality of life in patients with moderate-to-severe psoriasis: Results from a randomized, double-blind, placebo-controlled phase III trial. J Am Acad Dermatol. 2010;63(3):457-65.

Maruish ME, editor. User's manual for the SF-36v2 Health Survey. 3rd ed. Lincoln, RI: QualityMetric Incorporated; 2011.

Mukhtar R, Choi J, Koo JY. Quality of life issues in psoriasis. Dermatol Clin. 2004;22:389-95.

Mundt JC, Greist JH, Gelenberg AJ, Katzelnick DJ, Jefferson JW, Model JG. Feasibility and validation of a computer-automated Columbia-Suicide Severity Rating Scale using Interactive Voice Response Technology. J Psychiatric Res. 2010;44:1224-1228.

Ortonne JP. Redefining clinical response in psoriasis: targeting the pathological basis of disease. J Drugs Dermatol. 2004;3:13-20.

Parisi R, Symmons DP, Griffiths CE, Ashcroft DM. Identification and Management of Psoriasis and Associated ComorbidiTy (IMPACT) project team. Global epidemiology of psoriasis: A systematic review of incidence and prevalence. J Invest Dermatol. 2013;133:377–385.

Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, et al. The Columbia-Suicide Severity Rating Scale: Initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011;168:1266-1277.

Rachakonda TD, Schupp CW, Armstrong AW. Psoriasis prevalence among adults in the United States. J Am Acad Dermatol. 2014;70:512-6.

Raychaudhuri SP, Gross J. A comparative study of pediatric onset psoriasis with adult onset psoriasis. Pediatric Dermatology. 2000;17(3):174–178.

Snaith RP, Zigmond AS. The Hospital Anxiety and Depression Scale Manual. NFER: Nelson, Windsor; 1994.

Ulm K. A simple method to calculate the confidence interval of a standardized mortality ratio. Am J Epidemiol. 1990;131(2):373-375.

Yeung H, Takeshita J, Mehta NN, Kintmel SE, Ogdie A, Margolis DJ, et al. Psoriasis severity and the prevalence of major medical comorbidity: a population-based study. JAMA Dermatol. 2013;149:1173-9.

#### **APPENDICES** 18

#### 18.1 **Protocol Amendment 1**

nus, the study design changed from an open-label to a double-blind, placebo-controlled, parallel-group extension study with additional treatment groups included to be consistent with the feeder study, PS0010.

The other changes in this amendment are as follows:

Provide details of the study of the study blind.

The other changes in this amendment are as follows:

Bimekizumab

- Provide details of the revised PS0011 study including the study type and description
- Clarify the treatments to be administered and the criteria for assigning subjects to treatment in PS0011
- Reduce the number of secondary objectives to reflect the revised study design
- Reassign the PK and immunological variables from secondary objectives to other objectives
- Reassign the secondary safety variables to other safety variables
- Remove severity and frequency of TEAEs as a safety variable
- Remove the population PK from PS0011
- Classify the efficacy variables into secondary efficacy variables and other efficacy variables
- Extend the timing of the SFU Visit to 20 weeks after the last dose of study medication
- Extend the maximum duration of subject participation to 64 weeks
- Increase the frequency of safety laboratory testing (hematology/biochemistry)
- Clarify the frequency of safety laboratory testing (urinalysis)
- Revise the frequency of blood sampling for bimekizumab plasma concentrations and anti-bimekizumab antibody levels after Week 16
- Revise the frequency of completion of HADS
- Provide a rationale for the revised study design
- Facility to consent will not be included in the study

  resmove specific details on contraception but clarify that continued use of an acceptable forms of contraception (as specified in PS0010) is required in PS0011 for up to 20 weeks after the last dose of study treatment

  Remove reference to subjects who may have a strength of the significant infection and the study of the study

  - Include the requirement that subjects must have a negative IGRA to be eligible for PS0011 (obtained in PS0010)


- Clarify that subject must complete PS0010 to be eligible to participate in PS0011
- Provide more detail in the Withdrawal Criterion regarding subjects that develop illnesses that would interfere with study participation
- Clarify that topicals are not considered prohibited concomitant medication that would result in subject withdrawal in the Withdrawal Office 1.

- Provide more detail in the Withdrawal Criteria regarding the withdrawal of subjects due to AEs and clinical laboratory values
- Clarify the PASI threshold for withdrawal of a subject in the Withdrawal Criteria
- Revised IMP description to include bimekizumab and placebo
- Provide details on maintaining the blind during the study (eg, drug accountability, drug preparation and administration, and study monitoring) even though some clinical study team members will be unblinded to treatment assignments in PS0011
- Provide details on the procedures for breaking the blind in an emergency situation
- Provide further details on the assignment of subject to treatment by the IXRS
- Provide additional detail and a reference for recording the severity of AEs
- Extend the follow up of AE to 20 weeks after the last dose of IMP
- Clarify the adverse events for special monitoring
- Remove the requirement to test for alcohol in the PDILI urine toxicology screen
- Remove reference to Screening Log for PS0011
- Clarify in FAS and PK-PPS that 1 dose of study medication refers to the PS0011 to avoid confusion with study medication in PS0010
- Add section (General statistical considerations) to provide details on what constitutes descriptive statistics and to define 2 different sets of treatment groups that will be used when summarizing the data
- Update treatment emergent definition in the planned safety analyses to match with the revised 20-week SFU period and provide details on treatment groups used for summaries of AEs
  - Remove other safety analysis based on adjuster status as this is no longer applicable given the revised study design
- Provide additional details to specify what types of summaries will be done for PK and immunogenicity data

#### **Modifications and changes**

#### Global changes

The following changes were made throughout the protocol

- Treatment groups were added to be consistent with the feeder study PS0010 (with the exception of the bimekizumab 480mg Q4W treatment group)

  Secondary objectives were reduced to just 1 efficacy objective

  PK and immunological variables were assistant with the secondary safety as safety

- The timing of the SFU Visit was changed from 17 weeks after the last dose of study medication to 20 weeks after the last dose of study medication
- The maximum study duration for subjects was changed from 61 weeks to 64 weeks
- The frequency of safety laboratory testing (hematology/biochemistry) was increased from every 8 weeks to every 4 weeks (at every visit), including the SFU Visit
- The frequency of safety laboratory testing (urinalysis) was decreased from every 8 weeks to every 12 weeks, including the SFU Visit
- After the Week 16 Visit, the timing of blood samples for the measurement of PK and antibodies to bimekizumab was changed from every 8 weeks, followed by the SFU Visit to every 12 weeks (up to Week 40), followed by Week 48 and the SFU Visit
- The frequency of the HADS assessment was changed from every 12 weeks to every 4 weeks (at every visit) and the SFU Visit
- The term "photochemotherapy" was changed to "chemophototherapy" throughout for consistency
- Changes made throughout the statistics section to clarify which treatment groups would be used when summarizing data.
- Multiple changes made to account for the fact that summaries of change from Baseline variables would be calculated relative to the PS0010 Baseline and PS0011 Baseline, with both being presented in summary tables.
  - The List of Abbreviations was revised
- Minor editorial revisions were made

12 Aug 2016 PS0011

# Change #1

#### TITLE

A MULTICENTER, 48-WEEK, OPEN-LABEL EXTENSION STUDY TO ASSESS THE LONG-TERM SAFETY, TOLERABILITY, AND EFFICACY OF BIMEKIZUMAB IN ADULT SUBJECTS WITH MODERATE TO SEVERE CHRONIC PLAQUE PSORIASIS

#### Has been changed to:

A MULTICENTER, 48-WEEK, OPEN LABELDOUBLE-BLIND,
PLACEBO-CONTROLLED, PARALLEL-GROUP EXTENSION STUDY TO ASSESS
THE LONG-TERM SAFETY, TOLERABILITY, AND EFFICACY OF BIMEKIZUMAB IN
ADULT SUBJECTS WITH MODERATE TO SEVERE CHRONIC PLAQUE PSORIASIS

## Change #2

LIST OF ABBREVIATIONS

The following abbreviation has been added

CTCAE Common Terminology Criteria for Adverse Events

Change #3

LIST OF ABBREVIATIONS

ICH International council on Harmonisation

Has been changed to:

ICH International Council foron Harmonisation

Change #4

LIST OF ABBREVIATIONS

IMP investigational medicinal product

Has been changed to:

IMP investigational medicinal product(s)

Change #5

**Section 1 Summary** 

PS0011 is a multicenter, 48-week, open-label extension study to assess the long-term safety, tolerability, and efficacy of bimekizumab in eligible adult subjects with moderate to severe


chronic plaque psoriasis who complete PS0010. At Week 12 of PS0010, all eligible subjects continuing into PS0011 will undergo the PS0010 Week 12 study assessments and PS0011 Baseline assessments, and will then receive their first open-label dose of bimekizumab.

open label extension study to assess the long-term safety, tolerability, and efficacy of bimekizumab in eligible adult subjects with moderate to severe chronic plaque psoriasis who complete PS0010. At Week 12 of PS0010, all eligible subjects continuing into PS0011 will undergo the PS0010 Week 12 study assessments and any additional assessments, and will then receive their from PS0011. and any extensil PS0011.

## Change #6

#### **Section 1 Summary**

During the Open-Label Treatment Period, subjects will attend study visits at the site every 4 weeks (Q4W) for study assessments and administration of bimekizumab (if applicable) by study site staff through Week 48. Following completion or early withdrawal from the 48-week Open-Label Treatment Period, subjects will return for a Safety Follow-Up (SFU) Visit at 17 weeks after their last dose of bimekizumab. Subjects withdrawing early from the study will undergo the Early Withdrawal Visit assessments and will enter the SFU Period.

# Has been changed to:

During the **Open Label** Treatment Period, subjects will attend study visits at the **study** site every 4 weeks (Q4W) for study assessments and administration of bimekizumab or placebo (if applicable) by study site staff through Week 48. Any subject who does not achieve a Psoriasis Area and Severity Index (PASI) 75 response (defined as a 75% reduction in the PASI score from the Baseline of PS0010) at Week 12 or later in PS0011 will be withdrawn from study treatment and will return to complete the Early Withdrawal Visit assessments. Following completion or early withdrawal from the 48-week Open Label Treatment Period, subjects will return for a Safety Follow-Up (SFU) Visit at 17 20 weeks after their last dose of bimekizumab or placebo in PS0011.

Subjects withdrawing early from the study will undergo the Early Withdrawal Visit assessments and will enter the SFU Period.

The following text has been deleted

Section 1 Summary
The following Bimekizumab will initially be administered at a dose of 320mg Q4W subcutaneously (sc) during the 48 week Open Label Treatment Period, with an option to reduce the dose to 160mg Q4W at the discretion of the Investigator if the subject achieves a Psoriasis Area


**UCB** 12 Aug 2016 Bimekizumab PS0011

and Severity Index (PASI) 90 response (defined as a 90% reduction in the PASI score from the Baseline of PS0010) for at least 2 consecutive visits (not including the PS0011 Baseline sions or variations thereof. Visit). If the subject's disease is not adequately controlled on the 160mg Q4W dose, they may return to 320mg Q4W. The decision to return to 320mg Q4W dosing should be based upon treatment response, tolerability, and Investigator discretion, with the aim to use the dosing regimen that achieves the optimal benefit risk for each subject.

## Change #8

**Section 1 Summary** 

The following text has been added

Subjects who received placebo or bimekizumab 64mg, 160mg, or 320mg loading dose + 160mg Q4W in PS0010 must achieve PASI90 response at Week 12 in PS0010 to enter the PS0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving placebo or bimekizumab 64mg Q4W will be assigned to receive bimekizumab 160mg Q4W on entering PS001 I. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving bimekizumab 160mg or 320mg loading dose + 160mg Q4W will be assigned to receive bimekizumab 320mg Q4W on entering PS0011. Subjects who receive bimekizumab 320mg or 480mg Q4W in PS0010 will be assigned to receive bimekizumab 320mg Q4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010

## Change #9

#### **Section 1 Summary**

The primary objective of the study is to assess the long-term safety and tolerability of bimekizumab. Secondary objectives of the study are to assess the safety and tolerability of reduction of the dose of bimekizumab from 320mg Q4W to 160mg Q4W; to assess the pharmacokinetics (PK) of bimekizumab; to assess the immunogenicity of bimekizumab; and to assess the efficacy of open-label bimekizumab 320mg Q4W administered over 48 weeks with and without dose reduction.

# Has been changed to:

The primary objective of the study is to assess the long-term safety and tolerability of bimekizumab. The Ssecondary objectives of the study is are to assess the safety and tolerability of reduction of the dose of bimekizumab from 320mg Q4W to 160mg Q4W; to assess the pharmacokinetics (PK) of bimekizumab; to assess the pharmacokinetics (PK) of bimekizumab; to assess the immunogenicity of bimekizumab; and to assess the efficacy of open label bimekizumab 320mg O4W administered O4W over 48 weeks, with and without dose reduction. The other objectives of the study are to assess the pharmacokinetics (PK) and immunogenicity of bimekizumab.

#### **Section 1 Summary**

The primary safety variable is the incidence of treatment-emergent adverse events (TEAEs) adjusted by duration of subject exposure to treatment. The secondary safety variables are severity and frequency of TEAEs and change from Baseline of PS0010 in clinical laboratory values (chemistry, hematology, and urinalysis), vital signs, physical examination, and 12-lead electrocardiogram (ECG) results.

## Has been changed to:

The primary safety variable is the incidence of treatment-emergent adverse events (TEAEs) adjusted by duration of subject exposure to treatment. The **other secondary** safety variables are **severity and frequency of TEAEs and** change from Baseline of PS0010 **and PS0011** in clinical laboratory values (chemistry, hematology, and urinalysis), vital signs, physical examination, and 12-lead electrocardiogram (ECG) results.

## Change #11

#### **Section 1 Summary**

Pharmacokinetic variables are plasma concentrations of bimekizumab and population PK (CL/F, V/F). The immunological variable is anti-bimekizumab antibody levels prior to and following study treatment.

## Has been changed to:

The Pharmacokinetic PK variables are is plasma concentrations of bimekizumab and population PK (CL/F, V/F). Tthe immunological variable is anti-bimekizumab antibody levels prior to and following study treatment.

# Change #12

#### **Section 1 Summary**

The efficacy assessments are PASI, Investigator's Global Assessment (IGA), Dermatology Life Quality Index (DLQI), body surface area (BSA) affected by psoriasis, modified Nail Psoriasis Severity Index (mNAPSI) score, Psoriasis Scalp Severity Index (PSSI), Patient's Global Assessment of Disease Activity (PGADA), 36-item Short Form Health Survey (SF-36), and the Hospital Anxiety and Depression Scale (HADS); a detailed list of efficacy variables is presented in Section 4.4.

# Has been changed to:

The efficacy assessments are PASI, Investigator's Global Assessment (IGA) Dermatology Life Quality Index (DLQI), body surface area (BSA) affected by psoriasis, modified Nail Psoriasis Severity Index (mNAPSI) score, Psoriasis Scalp Severity Index (PSSI), Patient's Global Assessment of Disease Activity (PGADA), 36-item Short Form Health Survey (SF-36), and the

Hospital Anxiety and Depression Scale (HADS); a detailed list of the secondary and other

efficacy variables is presented in Section 4.4.

Therapy for patients with psoriasis varies according to the severity of disease. Limited or mild disease is often treated with topical therapies such as corticosteroids and vitamin D analogs. Patients with more severe disease are often treated with photochemotherapid oral phosphodiesterase 4 (PDE4) inhibitor (P necrosis factor (TNF) antagonists, interleukin (IL) 12/23 inhibitors, and IL-17A inhibitors. The effectiveness of TNF inhibitors in the treatment of psoriasis has been demonstrated in many Phase 3 clinical studies and has led to the approval of multiple TNF inhibitors for use in patients with moderate to severe psoriasis. Interleukin inhibitors include secukinumab and ixekizumab, IL-17A inhibitors approved for treatment of moderate to severe psoriasis. Ustekinumab is an IL-12/23 antagonist approved for use in patients with moderate to severe psoriasis, and brodalumab, an IL-17 receptor antagonist, has completed pivotal Phase 3 studies in psoriasis. Standard therapies for psoriasis are listed below:

#### Has been changed to:

Therapy for patients with psoriasis varies according to the severity of disease. Limited or mild disease is often treated with topical therapies such as corticosteroids and vitamin D analogs. Patients with more severe disease are often treated with photochemophototherapy, methotrexate, the oral phosphodiesterase 4 (PDE4) inhibitor (apremilast), or biologic agents, such as tumor necrosis factor (TNF) antagonists, interleukin (IL) 12/23 inhibitors, and IL-17A inhibitors. The effectiveness of TNF inhibitors in the treatment of psoriasis has been demonstrated in many Phase 3 clinical studies and has led to the approval of multiple TNF inhibitors for use in patients with moderate to severe psoriasis. Interleukin inhibitors include secukinumab and ixekizumab, 12-17A inhibitors approved for treatment of moderate to severe psoriasis. Ustekinumab is an IL-12/23 antagonist approved for use in patients with moderate to severe psoriasis, and brodalumab, an IL-17 receptor antagonist, has completed pivotal Phase 3 studies in psoriasis. Standard therapies for psoriasis are listed below:

# Change #14

#### Section 2.1.2 Current treatments for psoriasis

Photochemotherapy is a frequent option for moderate to severe patients, but the inconvenience of multiple treatment visits and varying efficacy limits its use in the market.

Has been changed to:

• Photos C' **Photoe**Chemophototherapy is a frequent option for moderate to severe patients, but the inconvenience of multiple treatment visits and varying efficacy limits its use in the market.


#### Section 2.2.1 Clinical

profession engible subjects who appears and profession of the subjects who appears and profession of the subjects with moderate to severe chronic plaque psoriasis. In PS0010, subjects will be randomized 1:1:1:1:1 to receive the following blinded study treatment regimens for a treatment period of 12 weeks:

Has been changed to:

The current study, PS0011, is a 48-week open label extension study for eligible subjects who complete PS0010, a Phase 2b, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study in adult subjects with moderate to severe chronic plaque psoriasis. In PS0010, subjects will be randomized 1:1:1:1:1:1 to receive the following blinded study treatment regimens for a treatment period of 12 weeks:

## Change #16

#### Section 3.2 Secondary objectives

Secondary objectives of the study are:

- To assess the safety and tolerability of reduction of the dose of bimekizumab from 320mg Q4W to 160mg Q4W
- To assess PK of bimekizumab
- To assess the immunogenicity of bimekizumab
- To assess the efficacy of open-label bimekizumab 320mg Q4W administered over 48 weeks with and without dose reduction

# Has been changed to:

# Section 3.2 Secondary objectives

The Secondary objectives of the study is are:

- To assess the safety and tolerability of reduction of the dose of bimekizumab from 320mg Q4W to 160mg Q4W
- To assess PK of bimekizumab
- Fo assess the immunogenicity of bimekizumab
- To assess the efficacy of open label bimekizumab 320mg Q4W administered Q4W over 48 weeks. with and without dose reduction

#### **Section 3.3 Other objectives (new section)**

The other objectives of the study are:

- To assess PK of bimekizumab
- To assess the immunogenicity of bimekizumab

# Change #18

#### Section 4.1.2 Secondary safety variables

Change from Baseline variables will be defined relative to the Baseline measurement from PS0010.

The secondary safety variables are:

- Severity and frequency of TEAEs
- Change from Baseline in clinical laboratory values (chemistry, hematology, and urinalysis)
- Change from Baseline in vital signs
- Change from Baseline in physical examination
- Change from Baseline in 12-lead ECG results

# Has been changed to:

# Section 4.1.2 Other Secondary safety variables

Change from Baseline variables will be defined relative to the Baseline measurements from **both** PS0010 **and PS0011**.

The **secondary** other safety variables are:

- Severity and frequency of TEAEs
- Change from Baseline in clinical laboratory values (chemistry, hematology, and urinalysis)
- Change from Baseline in vital signs
- Change from Baseline in physical examination
- Change from Baseline in 12-lead ECG results

# Change #19

#### Section 4.2 Pharmacokinetic variables

The PK variables are:

Plasma concentrations of bimekizumab and population PK (CL/F, V/F)

## Has been changed to:

#### Section 4.2 Pharmacokinetic variables

The PK variables are: is Pplasma concentrations of bimekizumab and population PK (CL/F, <del>V/F)</del>.

## Change #20

#### Section 4.4 Efficacy variables

Change from Baseline variables will be defined relative to the Baseline measurement from PS0010

## Has been changed to:

Change from Baseline variables will be defined relative to the Baseline measurements from both

- Change #21
  Section 4.4.1 Secondary efficacy variables (new section)

  The secondary efficacy variables are:

  PASI90 response over time

  IGA response (Clear or Almost Clear with at least a 2 category improvement from Baseline on a 5-point scale) over time Baseline on a 5-point scale) over time

# Change #22

Section 4.4.2 Other efficacy variables (new section; text previously under Section 4.4 **Efficacy variables**)

The following variables have been designated as secondary efficacy variables and have been deleted from the list of other efficacy variables

- PASI75, PASI90, and PASI100 response
- IGA response (Clear or Almost Clear with at least a 2 category improvement from Baseline on a 5-point scale)

# Change #23

#### **Section 5.1 Study description**

PS0011 is a multicenter, 48-week, open-label extension study to assess the long-term safety, tolerability, and efficacy of bimekizumab in eligible adult subjects with moderate to severe chronic plaque psoriasis who complete PS0010. At Week 12 of PS0010, all eligible subjects


Bimekizumab

continuing into PS0011 will undergo the PS0010 Week 12 study assessments and PS0011 Baseline assessments, and will then receive their first open-label dose of bimekizumab.

#### Has been changed to:

PS0011 is a multicenter, 48-week, double-blind, placebo-controlled, parallel-group open label extension study to assess the long-term safety, tolerability, and efficacy of bimekizumab in eligible adult subjects with moderate to severe chronic plaque psoriasis who complete PS0010. At Week 12 of PS0010, all eligible subjects continuing into PS0011 will undergo the PS0010 Week 12 study assessments and any additional PS0011 Baseline assessments, and will then receive their first open label dose of bimekizumab or placeboin **PS0011.** 

## Change #24

#### **Section 5.1 Study description**

During the Open-Label Treatment Period, subjects will attend study visits at the site Q4W for study assessments and administration of bimekizumab (if applicable) by study site staff through Week 48. Following completion or early withdrawal from the 48-week Open-Label Treatment Period, subjects will return for a SFU Visit at 17 weeks after their last dose of bimekizumab. Subjects withdrawing early from the study will undergo the Early Withdrawal Visit assessments and will enter the SFU Period.

Has been changed to:

During the Open Label Treatment Period, subjects will attend study visits at the study site every 4 weeks (O4W) for study assessments and administration of bimekizumab or placebo (if applicable) by study site staff through Week 48. Any subject who does not achieve PASI75 response at Week 12 or later in PS0011 will be withdrawn from study treatment and will return to complete the Early Withdrawal Visit assessments. Following completion or early withdrawal from the 48-week **Open Label** Treatment Period, subjects will return for a Safety Follow-Up (SFU) Visit at 17.20 weeks after their last dose of bimekizumab or placebo in PS0011.

Subjects withdrawing early from the study will undergo the Early Withdrawal Visit assessments and will enter the SFU Period.

# Change #25

Section 5.1 Study description

The following text has been deleted

Bimekizumab will initially be administered at a dose of 320mg O4W se during the 48 week Open Label Treatment Period, with an option to reduce the dose to 160mg O4W at the discretion of the Investigator if the subject achieves a PASI90 response (90% reduction in the PASI score from the Baseline of PS0010) for at least 2 consecutive visits (not including the PS0011 Baseline Visit). If the subject's disease is not adequately controlled on the




Bimekizumab

160mg Q4W dose, they may return to 320mg Q4W. The decision to return to 320mg Q4W dosing should be based upon treatment response, tolerability, and Investigator discretion, with the aim to use the dosing regimen that achieves the optimal benefit risk for each subject.

## Change #26

**Section 5.1 Study description** 

The following text has been added

Subjects who received placebo or bimekizumab 64mg, 160mg, or 320mg loading dose + 160mg Q4W in PS0010 must achieve PASI90 response at Week 12 in PS0010 to enter the PS0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving placebo or bimekizumab 64mg Q4W will be assigned to receive bimekizumab 160mg Q4W on entering PS0011. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving bimekizumab 160mg or 320mg loading dose + 160mg Q4W will be assigned to receive bimekizumab 320mg Q4W on entering PS0011. Subjects who receive bimekizumab 320mg Q4W in PS0010 will be assigned to receive bimekizumab 320mg Q4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010.

#### Change #27

# Section 5.1.1 Study duration per subject

The study duration for each subject is estimated to be up to a maximum of 61 weeks:

- Open-Label Treatment Period: up to 48 weeks
- SFU Visit: 17 weeks after the last dose of bimekizumab

The end of the study is defined as the date of the last visit of the last subject in the study.

# Has been changed to:

The study duration for each subject is estimated to be up to a maximum of 6164 weeks:

- Open Label Treatment Period: up to 48 weeks
- SFU Visit: 2017 weeks after the last dose of bimekizumab or placebo

The end of the study is defined as the date of the last visit of the last subject in the study.

# Table 5 1

Table 5-1 Schedule of study assessments

 Table 5-1:
 Schedule of study assessments

| Visit Week <sup>a</sup> | 750011 | Open-Label Treatment Period | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | PS0011<br>Baseline | Wk<br>4 | Wk<br>8 | Wk<br>12 | Wk<br>16 | Wk<br>20 | Wk<br>24 | Wk<br>28 | Wk<br>32 | Wk<br>36 | Wk<br>40 | Wk<br>44 | Wk 48/<br>WD | SFU <sup>b</sup> |
| Hematology/biochemistry/urinalysis | X <sup>f</sup> | | X | | X | | X | | XX | S | X | | X | X |
| Blood sample for bimekizumab plasma concentrations k | X <sup>f</sup> | X | X | X | X | | X | , 8 | NX T | | X | | X | X |
| Blood sample for anti-bimekizumab antibodies <sup>k</sup> | X <sup>f</sup> | X | X | X | X | | X | ano | X | | X | | X | X |
| HADS | X <sup>f</sup> | | | X | | | X | | | X | | | X | |

# Has been changed to:

Table 5-1: Schedule of study assessments

| Visit Week <sup>a</sup> | PS0011<br>Baseline | Open Label Treatment Period | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Protocol activity | | Wk<br>4 | Wk <sup>2</sup> | Wk<br>12 | Wk<br>16 | Wk<br>20 | Wk<br>24 | Wk<br>28 | Wk<br>32 | Wk<br>36 | Wk<br>40 | Wk<br>44 | Wk 48/<br>WD | SFU b |
| Hematology/biochemistry/urinalysis | X <sup>f</sup> | X.O | X | X | X | X | X | X | X | X | X | X | X | X |
| Urinalysis | X <sup>f</sup> | 17 | | X | | | X | | | X | | | X | X |
| Blood sample for bimekizumab plasma concentrations k | Xfr | X | X | X | X | | X | X | X | | X | | X | X |
| Blood sample for anti-bimekizumab antibodies k | Xf | X | X | X | X | | X | X | X | | X | | X | X |
| HADS | X <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |

12 Aug 2016 PS0011

## Change #29

#### Table 5-1 Schedule of study assessments

<sup>b</sup> The SFU Visit will occur 17 weeks after the last dose.

## Has been changed to:

extensions or variations thereof. <sup>b</sup> The SFU Visit will occur **2017** weeks after the last dose **of bimekizumab or placebo**.

## Change #30

#### Table 5-1 Schedule of study assessments

<sup>d</sup> To be performed prior to the first dose of open-label bimekizumab.

## Has been changed to:

<sup>d</sup> To be performed prior to the first dose of <del>open label</del> bimekizumab **or placebo in PS0011**.

# Change #31

Table 5-1 Schedule of study assessments

The following footnote has been deleted

<sup>m</sup> Bimekizumab will be administered at a dose of 320mg Q4W with an option to reduce the dose to 160mg Q4W at the discretion of the investigator if the subject achieves a PASI90 response (90% reduction in the PASI score from the Baseline of PS0010) for at least 2 consecutive visits (not including the PS0011 Baseline Visit). If the subject's disease is not adequately controlled on the 160mg O4W dose, they may return to 320mg O4W based on treatment response, tolerability, and Investigator discretion, with the aim to use the dosing regimen that achieves the optimal benefit risk for each subject.

# Change #32

Table 5-1 Schedule of study assessments

The following footnote has been added

<sup>m</sup> Subjects who received placebo or bimekizumab 64mg, 160mg, or 320mg loading dose + 160mg 04W in PS0010 must achieve PASI90 response at Week 12 in PS0010 to enter the PS0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving placebo or bimekizumab 64mg Q4W will be assigned to receive bimekizumab 160mg Q4W on entering PS0011. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving bimekizumab 160mg or 320mg loading dose + 160mg Q4W will be assigned to receive bimekizumab 320mg O4W on entering PS0011. Subjects who receive bimekizumab 320mg or 480mg O4W in PS0010 will be assigned to receive bimekizumab 320mg Q4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010. Any subject who does not

 The document control be used to support any materials alterial and any state of the control of t




BL=Baseline; PASI=Psoriasis Area and Severity Index; Q4W=every 4 weeks; sc=subcutaneously

<sup>&</sup>lt;sup>a</sup> Bimekizumab will be administered at a dose of 320mg Q4W sc with an option to reduce the dose to 160mg Q4W at the discretion of the Investigator if the subject achieves PASI90 response (90% reduction in the PASI score from the Baseline of PS0010) for at least 2 consecutive visits (not including the PS0011 Baseline Visit). If the subject's disease is not adequately controlled on the 100mg Q4W dose, they may return to 320mg Q4W. The decision to return to 320mg Q4W dosing should be based upon treatment response, tolerability, and Investigator discretion, with the aim to use the dosing regimen that achieves the optimal benefit-risk for each subject.

#### Has been changed to:



PASI=Psoriasis Area and Severity Index; Q4W=every 4 weeks; SFU=Safety Follow-Up

<sup>&</sup>lt;sup>a</sup> Subjects who received placebo or bimekizumab 64mg, 160mg, or 320mg loading dose + 160mg Q4W in PS0010 must achieve PASI90 response at Week 12 in PS0010 to enter the PS0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in

PS0010 while receiving placebo or bimekizumab 64mg will be assigned to receive bimekizumab 160mg on entering PS0011. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while receiving bimekizumab 160mg or 320mg loading dose + 160mg will be assigned to receive bimekizumab 320mg Q4W on entering PS0011.

b Subjects who receive bimekizumab 320mg or 480mg Q4W in PS0010 will be assigned to receive bimekizumab 320mg Q4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010.

<sup>c</sup> Any subject who does not achieve PASI75 response at Week 12 or later in PS0011 will be withdrawn from study treatment and will return to complete the Early Withdrawal Visit assessments.


#### Section 5.4 Rationale for study design and dose selection

mouerate to severe chronic plaque psoriasis. This study will allow the collection of further data on the long-term safety, tolerability, and efficacy of bimekizumab in this subject population and access/continued access to bimekizumab for subjects who received either bimekizumab or placebo in the lead-in study.

Has been changed to:

PS0011 is a 48-week. double study.

study for eligible subjects who complete PS0010, a Phase 2b, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study in adult subjects with moderate to severe chronic plaque psoriasis. Because some PS0010 subjects may have severe disease, the treatment in PS0011 provides more time to respond to a potentially efficacious treatment. PS0011 also provides an opportunity for nonresponding PS0010 placebo subjects to receive **bimekizumab.** This study will allow the collection of further data on the long-term safety, tolerability, and efficacy of bimekizumab in this subject population. and access/continued access to bimekizumab for subjects who received either bimekizumab or placebo in the Change #35
Section 5.4 Rationale for study design and dose selection

The following rationale has been deleted

In this study, bimekizumab will initially be administered at a dose of 320mg Q4W se, with an option to reduce the dose to 160mg Q4W at the discretion of the Investigator if the subject achieves a PASI90 response (90% reduction in the PASI score from the Baseline of PS0010) for at least 2 consecutive visits (not including the PS0011 Baseline Visit). If the subject's disease is not adequately controlled on the 160mg Q4W dose, they may return to 320mg Q4W. The decision to return to 320mg Q4W dosing should be based upon treatment response, tolerability, and Investigator discretion, with the aim to use the dosing regimen that achieves the optimal benefit risk for each subject. This will allow the assessment of safety, tolerability, and efficacy following a reduction in the bimekizumab dose to 160mg Q4W.

The rationale for the selection of the 320mg Q4W dose for this study is based on the following:

- The optimal therapeutic dose of bimekizumab will not yet be known at the time subjects begin entering PS0011 from PS0010.
- Stratification of dosing in PS0011 based on prior dose in PS0010 would result in unblinding of PS0010.

- The 320mg Q4W dose is within the range of doses that have already been explored by iv administration. This dose was selected based on modeling using the currently available data and may be modified, if appropriate, as further data are collected on the optimal dose of bimekizumab.
- Based on currently available data and modeling, few subjects are expected to have a robust response to bimekizumab 64mg Q4W in PS0010. The 320mg Q4W dose allows subjects who received placebo or bimekizumab 64mg Q4W in PS0010 to receive a potentially effective dose in this extension study. Although some subjects may have had some response to a lower dose in PS0010 (eg, 64mg or 160mg), the increased dose in PS0011 could provide additional benefit, resulting in an improved response or remission.
- The 320mg Q4W dose decreases the risk that subjects who responded to treatment in PS0010 experience a loss of efficacy due to a dose reduction upon entry into PS0011. Importantly, subjects who are nonresponders after 12 weeks of treatment in PS0011 will be withdrawn. This minimizes exposure to a possibly noneffective treatment.

Section 5.4 Rationale for study design and dose selection.

The following rationale has been added.

The PSO011-3-4 The PS0011 design (Figure 5-1) allows PASI90 responders in PS0010 to continue their dose in PS0011, thus permitting these subjects to remain on the dose that resulted in this response after 12 weeks of initial treatment in PS0010. It also provides an opportunity for an increased dose among PS0010 nonresponders (ie, <PASI90). PASI90 was selected as the response criterion in PS0010 to ensure that a sufficiently high efficacy response was achieved. This type of dose escalation for those who do not achieve a desired response after 12 weeks is common in clinical practice.

Regardless of PASI90 response at Week 12 of PS0010, subjects who received the 2 highest doses of bimekizumab (320mg and 480mg Q4W) in PS0010 will begin PS0011 on the 320mg Q4W dose. For those subjects who do achieve PASI90 response, this will allow a continuation of the PS0010 dose for subjects initially receiving 320mg Q4W and a dose down for subjects originally randomized to the 480mg Q4W dose. Because bimekizumab 480mg O4W is the highest dose evaluated in PS0010 and because it requires 3 injections, it will be of interest to evaluate whether these subjects can maintain response in PS0011 with the lower 320mg dose, allowing the blind to be maintained with the use of only 2 injections at each study administration visit.

To protect against the possibility of exposing subjects to an ineffective treatment for extended periods of time, subjects across all treatment groups who have not achieved PASI75 response at Week 12 or later in PS0011 will be withdrawn from study treatment. Because this withdrawal decision is based strictly on the PASI response and not on the original study treatment, it can be done in such a way that will not unblind subjects or Investigators.

#### Section 6.1 Inclusion criteria

1. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the subject or by the parent(s) or legal representative.

## Has been changed to:

1. An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the subject. or by the parent(s) or legal anyextension representative.

## Change #38

#### Section 6.1 Inclusion criteria

2. Subject/legal representative is considered reliable and capable of adhering to the protocol and visit schedule according to the judgment of the Investigator.

## Has been changed to:

2. Subject/legal representative is considered reliable and capable of adhering to the protocol and visit schedule according to the judgment of the Investigator.

# Change #39

Section 6.1 Inclusion criteria

3. Subject completes all dosing requirements in PS0010 without meeting any withdrawal criteria.

# Has been changed to:

3. Subject completes all dosing requirements in PS0010 without meeting any withdrawal criteria and completes the study.

# Change #40 🔊

#### Section 6.1 Inclusion criteria

4. Female subjects must be postmenopausal (at least 1 year; to be confirmed hormonally at the PS0011 Baseline Visit, if less than 2 years since last menstrual period), permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy) or, if of childbearing potential, must be willing to use a highly effective method of contraception up until 20 weeks after last administration of study medication (anticipated 5 half lives), and have a negative pregnancy test at Visit 1 (Baseline) and immediately prior to first dose. The following methods are considered highly effective when used consistently and correctly:

- -combined (estrogen and progestogen) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)

- intrauterine hormone releasing system

- receasing system

   vascetomized partner (where postvasectomy testing had demonstrated sperm clearance).

   sexual abstinence if it is in accordance with a subject's proceediffestyle. Subjects who use abstinence as a formabstain from heterosexual into medication. Start accordance with the subject's lifestyle at regular intervals during the study.

Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, up till 20 weeks after the last administration of study medication (anticipated 5 half lives).

## Has been changed to:

4. Female subjects of childbearing potential and male subjects with a partner of childbearing potential must continue to use an acceptable method of contraception (as detailed in PS0010) for up to 20 weeks after the last dose of study treatment in PS0011.

# Change #41

Section 6.2 Exclusion criteria

Exclusion criterion #4 has been deleted

4. Subject has any current sign or symptom that may indicate a medically significant infection.

# Change #42

Section 6.2 Exclusion criteria

Exclusion criterion #5 has been deleted

S. Subject has current clinically active infection with Histoplasma, Coccidiodes, Paracoccidioides, Pneumocystis, tuberculosis (TB), nontuberculous mycobacteria (NTMB), Blastomyces, Aspergillus, or Candidiasis (systemic). Any subject diagnosed with Histoplasmosis, Coccidiodes, Paracoccidiodes, Pneumocystis, TB, NTMB, Blastomyces, Aspergillus, or Candidiasis (systemic) during PS0010 is excluded from **PS0011** even if treatment has been completed.

#### Section 6.2 Exclusion criteria

The following exclusion criterion has been added

4. Subject must have a negative interferon gamma release assay (IGRA) as measured at Week 8 of PS0010.

# Change #44

Section 6.2 Exclusion criteria (now exclusion criterion #5; previously exclusion criterion #6)

6. Any subject who meets any withdrawal criteria in the feeder study (PS0010) is excluded from participating in the open-label extension study (PS0011).

## Has been changed to:

5. Any subject who meets any withdrawal criteria in the feeder study (PS0010) is excluded from COPY application participating in the open label extension study (PS0011).

## Change #45

#### Section 6.3 Withdrawal criteria

Subjects should be withdrawn from the study and will be asked to complete the Early Withdrawal Visit and SFU Visit (17 weeks after the last received dose) if any of the following events occur

# Has been changed to:

Subjects should be withdrawn from the study and will be asked to complete the Early Withdrawal Visit and SFU Visit (17-20 weeks after the last received dose) if any of the following events occur:

# Change #46

#### Section 6.3 Withdrawal criteria

4. Subject develops an illness that would interfere with his/her continued participation.

.. Judgect develops an illness that in the opinion of the Investigator would interfere with this/her continued participation if the risk of continuing participation outweighs the potential benefit. 4. Subject develops an illness that in the opinion of the Investigator would interfere with

#### Section 6.3 Withdrawal criteria

5. Subject develops erythrodermic, guttate, or generalized pustular form of psoriasis.

## Has been changed to:

5. Subject develops erythrodermic, guttate, or generalized pustular form of psoriasis.

#### Change #48

Section 6.3 Withdrawal criteria

The following text has been added to withdrawal criterion #6

Additional information on TB policies are provided in Section 9.8.1.

## Change #49

#### Section 6.3 Withdrawal criteria

and any extensions or variations thereof.

Pication and any extensions

Pres 8. Subject uses prohibited concomitant medications that may present a risk to the safety of the subject in the opinion of the Investigator and/or the Medical Monitor

## Has been changed to:

8. Subject uses prohibited concomitant medications, with the exception of topicals, as defined in this protocol (Section 7.8.2), that may present a risk to the safety of the subject in the opinion of the Investigator and/or the Medical Monitor.

# Change #50

Section 6.3 Withdrawal criteria

9. Subject develops laboratory abnormalities (with or without clinical symptoms) of neutropenia <1.0x10<sup>9</sup>/L, lymphopenia <0.5x10<sup>9</sup>/L, or other clinically relevant laboratory abnormalities consistent with rheumatology Common Terminology Criteria (CTC) Grade 3 or higher. (Refer to Section 6.3.1 for withdrawal criteria in relation to potential drug induced liver injury [PDILI]).

## Has been changed to:

- 9. Subject has a clinical laboratory value meeting the following criteria:
  - CTCAE Grade 3 and above: subjects must be withdrawn regardless of relationship to study drug or duration of event.
  - **CTCAE Grade 2** 
    - Subjects may remain in the study if the event is transient. If a subject has a Grade 2 laboratory abnormality, a retest is required within 1 to 2 weeks at a scheduled or unscheduled visit. If the repeat value is below Grade 2, the subject

may receive the next scheduled study treatment. If the value on the repeat is still Grade 2 or above, a second repeat test must be performed and results made available prior to the next scheduled study treatment. If this second repeat value is still Grade 2 or above, the subject must be withdrawn.

## Change #51

#### Section 6.3 Withdrawal criteria

11. Subjects with a HADS-D score ≥15 must be withdrawn. Any subject who has a HADS-D score of ≥10 should be referred immediately to a Mental Healthcare Professional for further evaluation and potential withdrawal by the Investigator.

## Has been changed to:

11. Subjects with a HADS-D score ≥15 must be withdrawn. Any subject who **develops has** a HADS-D score of ≥10 during the study should be referred immediately to a Mental Healthcare Professional for further evaluation and potential withdrawal by the Investigator.

## Change #52

#### Section 6.3 Withdrawal criteria

12. Subject does not achieve a PASI50 at Week 12 or later following open-label treatment in PS0011.

# Has been changed to:

12. Subject does not achieve **a PASI50 PASI75** at Week 12 or later following **open label study** treatment in PS0011.

# Change #53

#### Section 6.3 Withdrawal criteria

#### The following withdrawal criterion for AEs has been added

- 13. Subject experiences an AE as described below:
  - Any CTCAE Grade 3 and above adverse event (AE) that is assessed as related to study drug in the opinion of the Investigator
    - If the event is deemed to be not related to study drug by the Investigator, the subject may remain in the study after approval by the Medical Monitor.
  - Any CTCAE Grade 2 event that is evaluated as related to study drug in the opinion of the Investigator, is persistent, and falls into any of the following System Organ Classes (SOCs): "Blood and lymphatic disorders," "Cardiac disorders," or "Vascular disorders."
    - Persistent is defined as lasting 28 days or more, which spans at least 2 scheduled injections.

#### Section 7.1 Description of investigational medicinal product

The IMP used in this study is bimekizumab.

#### Has been changed to:

The IMP used in this study is are bimekizumab and placebo.

## Change #55

Section 7.1 Description of investigational medicinal product

The following description of placebo has been added

tensions of variations thereof. Placebo will be supplied as 0.9% sodium chloride aqueous solution (physiological saline, preservative free) of pharmacopoeia (USP/Ph.Eur) quality appropriate for injection.

## Change #56

#### Section 7.2 Treatments to be administered

During the Treatment Period, all subjects will receive bimekizumab 320mg Q4W sc administered for up to 48 weeks in an open-label manner. At the discretion of the Investigator, and if the subject achieves PASI90 response (90% reduction in the PASI score from the Baseline of PS0010) for at least for at least 2 consecutive visits (not including the PS0011 Baseline Visit), the bimekizumab dose may be reduced to 160mg Q4W sc. If the subject's disease is not adequately controlled on the 160mg Q4W dose, they may return to 320mg Q4W. The decision to return to 320mg O4W dosing should be based upon treatment response, tolerability, and Investigator discretion, with the aim to use the dosing regimen that achieves the optimal benefitrisk for each subject.

# Has been changed to:

During the Treatment Period, all subjects will receive bimekizumab or placebo 320mg Q4W se administered sc for up to 48 weeks in an open label manner. (refer to Figure 5-1 for further details). At the discretion of the Investigator, and if the subject achieves a PASI90 response (90% reduction in the PASI score from the Baseline of PS0010) for at least for at least 2 consecutive visits (not including the PS0011 Baseline Visit), the bimekizumab dose may be reduced to 160mg Q4W se. If the subject's disease is not adequately controlled on the 160mg 04W dose, they may return to 320mg 04W. The decision to return to 320mg 04W dosing should be based upon treatment response, tolerability, and Investigator discretion, this docular subject. with the aim to use the dosing regimen that achieves the optimal benefit risk for each


#### Section 7.2 Treatments to be administered

Paccoo or bimekizumab 64mg, 160mg, or 320mg loading dose + 100mg Q4W in PS0010 must achieve PASI90 response at Week 12 in PS0010 to enter the PS0011 extension study on the same treatment dose. Subjects who do not achieve PASI90 response at Week 12 in PS0010 while on these treatments will be assigned to receive bimekizumab 160mg or 320mg Q4W at Baseline in PS0011 as follows:

• Subjects receiving:

- bimekizumab 160mg Q4W in PS0011.
- Subjects receiving bimekizumab 160mg Q4W and 320mg loading dose # 160mg Q4W in PS0010 will be assigned to bimekizumab 320mg O4W in PS0011.

Subjects who receive bimekizumab 320mg or 480mg Q4W in PS0010 will be assigned to gardh gardh copy it Zajion application receive bimekizumab 320mg Q4W on entering PS0011, regardless of their PASI90 response at Week 12 in PS0010.

## Change #58

## Section 7.2 Treatments to be administered

The study medication is to be administered in the clinic by study site staff as 2 sc injections for the 320mg dose or 1 sc injection for the 160mg dose. Suitable areas for sc injections are the lateral abdominal wall and upper outer thigh, Injection sites should be rotated and injections should not be given into areas where the skin is tender, bruised, red, or hard.

# Has been changed to:

The study medication is to be administered in the clinic by study site staff as 2 sc injections for the 320mg dose or 1 sc injection for the 160mg dose for all study treatments in PS0011. Suitable areas for sc injections are the lateral abdominal wall and upper outer thigh. Injection sites should be rotated and injections should not be given into areas where the skin is tender, bruised, red, or hard.

# Change #59

# Section 7.3 Packaging

Bimekizumab will be packaged and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. It will be suitably packaged in such a way as to protect the product from deterioration during transport and storage. Further information regarding storage and transport conditions are provided in the IMP Handling Manual.

# Has been changed to:

Bimekizumab and placebo will be packaged and labeled according to Good Manufacturing Practice (GMP) guidelines and applicable laws or regulations. It will be suitably packaged in Bimekizumab

such a way as to protect the product from deterioration during transport and storage. Further information regarding storage and transport conditions are provided in the IMP Handling Manual.

Clinical drug supplies will be labeled in accordance with the current International Council on Harmonisation (ICH) guidelines on Good Clinical Practice (GCP) and GMP and will include locally required statements. If necessary, labels will be translated into 41.

Has been changed to:

Clinical drug

Clinical drug supplies will be labeled in accordance with the current International Council onfor Harmonisation (ICH) guidelines on Good Clinical Practice (GCP) and GMP and will include any locally required statements. If necessary, labels will be translated into the local language.

## Change #61

## Section 7.5 Handling and storage requirements

The IMP must be stored under refrigerated conditions (2°C to 8°C) and protected from light. The study drug must not be frozen.

## Has been changed to:

The IMP Bimekizumab and placebo must be stored under refrigerated conditions (2°C to 8°C) and protected from light. The study drug must not be frozen.

# Change #62

Section 7.6 Drug Accountability

The following text has been added

In order to maintain the blind, all IMP documentation (eg, shipping receipts, drug accountability logs, interactive web or voice response system [IXRS] treatment assignments) must be maintained and accessed only by trained unblinded site personnel. Designated unblinded site personnel must be appropriately trained and licensed (per country guidelines) to administer injections.

Blinded study staff may be delegated the responsibility to receive, inventory, and destroy the used kits. The packaging identifies each kit by a unique number that does not correlate to the contents and does not unblind study site staff. Unblinded study staff will be responsible for the preparation (eg, breaking tamper proof sticker on kit) of the IMP, including recording the administration information on the source document.

#### Section 7.8.1 Permitted concomitant treatments (medications and therapies)

#### **Topical medications**

Subjects will be allowed to use topical medications (corticosteroids, retinoids, Vitamin D analogs coal tar, etc) as needed during this open-label extension.

## Has been changed to:

#### **Topical medications**

Subjects will be allowed to use topical medications (corticosteroids, retinoids, Vitamin D analogs coal tar, etc) as needed during this open label extension study.

# Change #64

Section 7.9 Prohibited concomitant treatments (medications and therapies)

The following text has been deleted

Subjects who use prohibited medications will be withdrawn from study treatment but followed until the SFU Visit.

# Change #65

Table 7-1 Prohibited psoriasis medications during PS0011

phototherapy or photochemotherapy

# Has been changed to:

phototherapy or **chemophototherapy** photochemotherapy

# Change #66

Section 7.9 Blinding

The following text has been deleted

This is an open label extension study and no blinding will be performed. All subjects' treatment assignments during PS0010 will remain blinded until database lock of PS0010. This document can't

12 Aug 2016

PS0011

## Change #67

#### **Section 7.9 Blinding**

The following text has been added

Due to differences in presentation of the IMP (bimekizumab and placebo), special precautions will be taken to ensure study blinding, and study sites will have blinded and unblinded personnel.

Bimekizumab and placebo injections will be prepared and administered at the study sites by unblinded dedicated study personnel who will only have responsibility for dosing and drug accountability.

Study sites will be required to have a written blinding plan in place, signed by the Principal Investigator, which will detail the site's steps for ensuring that the double-blind nature of the study is maintained.

During the study, the Sponsor will provide blinded and unblinded site monitors for the purposes of verifying safety, efficacy, and drug administration and documentation records. Blinded study monitors and study site personnel, blinded to treatment assignment, will not discuss or have access to any drug-related information.

When the feeder (PS0010) study is unblinded, selected PS0010 study team members will have access to subject-level data. Because treatment assignment in PS0011 is based on PASI90 response at Week 12 of PS0010 as opposed to randomization, Sponsor personnel with such access to the PS0010 data will know the treatment assignments of all PS0010 subjects including those continuing in PS0011. This operational unblinding to PS0011 treatment assignment will pertain to selected clinical PS0010 study team members (some of whom may be involved in PS0011) but will not extend to blinded staff at the investigational sites of PS0011.

While the blinding of Sponsor clinical study team members is important for ensuring the integrity of data collection and analysis in a controlled study, this unblinding is considered acceptable because the primary evaluation of efficacy, upon which sample size calculations were based, will be performed in a blinded manner using Week 12 data of PS0010. Additionally, because investigational site staff collecting and recording study data remain blinded, those data will not be impacted by the unblinding of selected Sponsor clinical study team members. Finally, to ensure that unblinding of study team members did not impact the primary safety outcome of PS0011, sensitivity analyses will be outlined in the SAP to evaluate what, if any, impact there was on the results based on queries that resulted in changes to the AE data following the unblinding of PS0010.

Further details are provided in the study manuals and site blinding plan.

# Change #68

Section 7.9.1 Procedures for maintaining and breaking the treatment blind (new section)

This new section has been added and subdivided (see Change #69 and Change #70)

Section 7.9.1.1 Maintenance of study treatment blind (new subsection)

The following text has been added

All subject treatment details (bimekizumab or placebo) will be allocated and maintained by the IXRS.

## Change #70

Section 7.9.1.2 Breaking the treatment blind in an emergency situation (new subsection)

The following text has been added

The integrity of this clinical study must be maintained by observing the treatment blind. In the event of an emergency for which the appropriate treatment for a subject cannot be made without knowing the treatment assignment, it will be possible to determine to which treatment arm and dose the subject has been allocated by contacting the IXRS. All sites will be provided with details of how to contact the system for code breaking at the start of the study. The Medical Monitor or equivalent should be consulted prior to unblinding, whenever possible.

The Clinical Project Manager will be informed immediately via the IXRS when a code is broken, but will remain blinded to specific treatment information. Any unblinding of the IMP performed by the Investigator must be recorded in the source documents and on the Study Termination eCRF page.

# Change #71

# Section 7.10 Randomization and numbering of subjects

This is an open-label extension study and no randomization will be performed. All subjects will receive bimekizumab 320mg Q4W sc with an option to reduce the dose to 160mg Q4W at the discretion of the Investigator (see Section 7.2 for further details).

Subjects will continue with the 5-digit subject numbers assigned by the interactive web or voice response system (XRS) in the preceding study. The randomization number must be incorporated into the eCRF.

# Has been changed to:

This is an open label extension study and nNo randomization will be performed in this study. An IXRS will be used for assigning eligible subjects to study treatment based on a predetermined assignment schedule. An independent biostatistician or designee who is not involved in this study or the feeder study, PS0010, will produce this assignment schedule. Details of the study treatments in PS0011 are presented in Section 7.2. All subjects will receive bimekizumab 320mg Q4W sc with an option to reduce the dose to 160mg Q4W at the discretion of the Investigator (see Section 7.2 for further details).
Subjects will continue with the 5-digit subject numbers assigned by the interactive web or voice response system (IXRS) in the preceding study. The randomization number must be incorporated into the eCRF.

#### Change #72

#### **Section 8 Study procedures by visit**

For the SFU Visit (17 weeks after the last dose), the visit should occur no more than 3 days prior to the scheduled visit date and within 7 days after the scheduled visit date (-3 days/+7 days).

### Has been changed to:

• For the SFU Visit (2017 weeks after the last dose of bimekizumab or placebo), the visit should occur no more than 3 days prior to the scheduled visit date and within 7 days after the scheduled visit date (-3 days/+7 days).

#### Change #73

Section 8.2 Week 4 (±3 days)

The following assessment has been added

**HADS** 

### Change #74

Section 8.2 Week 4 (±3 days)

A blood sample for safety laboratory testing has been added

- Obtain blood samples for:
  - Standard safety laboratory tests (hematology and biochemistry)

# Change #75

Section 8.3 Week 8 (±3 days); Week 16 (±3 days); Week 32 (±3 days); and Week 40 (±3 days)

rhis document HADS The following assessment has been added

Section 8.3 Week 8 (±3 days); Week 16 (±3 days); Week 32 (±3 days); and Week 40 (±3 days)

- Obtain blood samples for:
  - Bimekizumab plasma concentration
  - Anti-bimekizumab antibodies

#### Has been changed to:

- Obtain blood samples for:
  - Bimekizumab plasma concentration (not collected at Week 32)
  - Anti-bimekizumab antibodies (not collected at Week 32)

#### Change #77

Section 8.3 Week 8 (±3 days); Week 16 (±3 days); Week 32 (±3 days); and Week 40  $(\pm 3 \text{ days})$ 

A urine sample for safety laboratory testing has been deleted

- Obtain a urine sample for:
  - Standard safety laboratory tests (urinalysis)

#### Change #78

Section 8.4 Week 12 (±3 days)

A blood sample for safety laboratory testing has been added

- Obtain blood samples for:
  - Standard safety laboratory tests (hematology and biochemistry)

### Change #79

Section 8.4 Week 12 (±3 days)

sample for safety l

or Obtain urine sample for:

- Standard safe

'itis A urine sample for safety laboratory testing has been added

- - Standard safety laboratory tests (urinalysis)

**UCB** 

Section 8.5 Week 20 (±3 days); Week 28 (±3 days); and Week 44 (±3 days)

The following assessment has been added

HADS

#### Change #81

Section 8.5 Week 20 (±3 days); Week 28 (±3 days); and Week 44 (±3 days)

Blood samples for safety laboratory testing and for measuring PK and antibodies to bimekizumab have been added

- **Obtain blood samples for:** 
  - Standard safety laboratory tests (hematology and biochemistry)
  - Bimekizumab plasma concentration (collected only at Week 28)
  - Anti-bimekizumab antibodies (collected only at Week 28)

### Change #82

Section 8.6 Week 24 (±3 days)

A blood sample for measuring PK and antibodies to bimekizumab has been deleted

- Obtain blood samples for:
  - **Bimekizumab plasma concentration**
  - Anti bimekizumab antibodies

### Change #83

Section 8.7 Week 36 (±3 days)

A blood sample for safety laboratory testing has been added

- **Obtain blood sample for:** 
  - Standard safety laboratory tests (hematology and biochemistry)

## Change #84

Section 8.7 Week 36 (±3 days)

A urine sample for safety laboratory testing has been added

- Obtain a urine sample for:
  - Standard safety laboratory tests (urinalysis)

Section 8.9 SFU Visit (17 weeks after the last dose; -3/+7 days)

#### Has been changed to:

Ation and any extensions or variations thereof. Section 8.9 SFU Visit (1720 weeks after the last dose of bimekizumab or placebo; -3/+7 days)

#### Change #86

Section 8.9 SFU Visit (17 weeks after the last dose; -3/+7 days)

The following assessment has been added

HADS

#### Change #87

**Section 9.1.3 Description of AEs** 

Details for completion of the AE eCRF (including judgment of relationship to IMP) are described in the eCRF Completion Guidelines.

#### Has been changed to:

When recording the severity of an AE in the CRF (ie, mild, moderate, or severe), the **Investigator must refer to the CTCAE Version 4** 

(http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm). Details for completion of the AE eCRF (including judgment of severity and relationship to IMP) are described in the eCRF Completion Guidelines.

### Change #88

## Section 9.1.4 Follow up of AEs

If an AE is ongoing at the end of the study for a subject, follow up should be provided until resolution/stable level of sequelae is achieved, or until the Investigator no longer deems that it is clinically significant, or until the subject is lost to follow up. If no follow up is provided, the Investigator must provide a justification. The follow up will usually be continued for 17 weeks after the subject has discontinued his/her IMP.

### Has been changed to:

If an AE is ongoing at the end of the study for a subject, follow up should be provided until resolution/stable level of sequelae is achieved, or until the Investigator no longer deems that it is clinically significant, or until the subject is lost to follow up. If no follow up is provided, the Investigator must provide a justification. The follow up will usually be continued for 1720 weeks after the subject has discontinued his/her IMP.

#### **Section 9.1.6 Pregnancy**

A SFU Visit should be scheduled 17 weeks after the subject has discontinued her IMP.

#### Has been changed to:

A SFU Visit should be scheduled 1720 weeks after the subject has discontinued her IMP.

#### Change #90

#### Section 9.6 Adverse events for special monitoring

sions or variations thereof. Adverse events for special monitoring for this study include: serious infections (including opportunistic infections and TB; see Section 9.8.1), cytopenias, hypersensitivities, suicide ideation or behavior (assessed using the eC-SSRS; see Section 9.8.6), depression and anxiety (assessed using the HADS; see Section 12.9), major cardiac events, and liver function test changes/enzyme elevations (ALT, AST, bilirubin; see Section 9.7.1), malignancies, and inflammatory bowel diseases.

### Has been changed to:

Adverse events for special monitoring for this study include: serious infections (including opportunistic infections and TB; see Section 9.8.1), cytopenias, hypersensitivities, suicide ideation or behavior (assessed using the eC-SSRS; see Section 9.8.6), depression and anxiety (assessed using the HADS; see Section 12.9), major eardiac cardiovascular events, and liver function test changes/enzyme elevations (ALT, AST, bilirubin; see Section 9.7.1), malignancies, and inflammatory bowel diseases.

## Change #91

## **Table 9-4 PDILI laboratory measurements**

<sup>a</sup> For detecting substances (ie, alcohol, amphetamines, benzodiazepines, opioids, marijuana, cocaine, phencyclidine, and tricyclic antidepressants), additional tests may be performed based on the Investigator's medical judgment and patient's history.

## Has been changed to:

<sup>a</sup> For detecting substances (ie, alcohol amphetamines, benzodiazepines, opioids, marijuana, cocaine, phencyclidine, and tricyclic antidepressants), additional tests may be performed based on the Investigator's medical judgment and patient's history.

#### Section 9.8.1 Assessment and management of TB and TB risk factors

#### LTB

Once withdrawn from study treatment, subjects should return for the Week 48/Withdrawal Visit, complete all Early Withdrawal Visit assessments, and complete a SFU Visit (17 weeks after the last dose of study medication).

#### Has been changed to:

Once withdrawn from study treatment, subjects should return for the Week 48/Withdrawal Visit, complete all Early Withdrawal Visit assessments, and complete a SFU Visit (2017 weeks after tion and any exten the last dose of study medication).

#### Change #93

#### Section 9.8.1.4 TB management

LTB infection and active TB identified during study

The subject should be encouraged to complete a SFU Visit (1) weeks after the last dose of study medication).

### Has been changed to:

The subject should be encouraged to complete a SFU Visit (2017 weeks after the last dose of study medication).

## Change #94

### Section 13.3.3 Subject Screening and Enrollment log/Subject Identification Code list

The subject's screening and enrollment will be recorded in the Subject Screening and Enrollment Log.

## Has been changed to:

#### Section 13.3.3 Subject Screening and Enrollment log/Subject Identification Code list

The subject's screening and enrollment will be recorded in the Subject Screening and Enrollment Log.

## Change #95

#### Section 14.1 Definition of analysis sets

The Full Analysis Set (FAS) will consist of all enrolled subjects who receive at least 1 dose of the study medication and have a valid efficacy measurement for PASI at Baseline of PS0011.

#### Has been changed to:

The Full Analysis Set (FAS) will consist of all enrolled subjects who receive at least 1 dose of the study medication **in PS0011** and have a valid efficacy measurement for PASI at Baseline of PS0011.

#### Change #96

#### **Section 14.1 Definition of analysis sets**

The Pharmacokinetics Per-Protocol Set (PK-PPS) will consist of all enrolled subjects who receive at least 1 dose of the study medication and provide at least 1 quantifiable plasma concentration postdose in PS0011.

#### Has been changed to:

The Pharmacokinetics Per-Protocol Set (PK-PPS) will consist of all enrolled subjects who receive at least 1 dose of the study medication **in PS0011** and provide at least 1 quantifiable plasma concentration postdose in PS0011.

#### Change #97

Section 14.2 General statistical considerations (new section)

The following text has been added

No inferential statistical analyses are planned for this extension study. Instead, all variables will be presented using summary statistics. For categorical variables, counts and percentages will be displayed. For continuous variables, summary statistics will consist of the number of available observations, arithmetic mean, standard deviation, median, minimum, and maximum unless stated otherwise.

Because subjects entering PS0011 may or may not be continuing on the same dose as that received in PS0010, there are various combinations of treatment that could be received when considering both PS0010 and PS0011 together. For describing the summaries to be produced, treatment groups will be categorized as either the PS0011 treatment groups or PS0010/PS0011 treatment groups. These categorizations are outlined below.

### **PS0011 treatment groups**

This refers to the study treatment assigned to the subject at the beginning of PS0011 and does not account for the treatment received in PS0010. The PS0011 treatment groups are as follows:

Placebo

- Bimekizumab 64mg Q4W
- Bimekizumab 160mg Q4W
- Bimekizumab 320mg Q4W
- All Bimekizumab (optional to be used only if specified)

#### PS0010/PS0011 treatment groups

This refers to the combination of the randomized treatment in PS0010 and the treatment assigned at the beginning of PS0011. Some groups have been combined where it is considered appropriate to do so. The PS0010/PS0011 treatment groups with descriptions are as follows:

- Placebo to Placebo Subjects randomized to placebo in PS0010 who achieve PASI90 response at Week 12 of PS0010 and continue to receive placebo in PS0011.
- Placebo to Bimekizumab 160mg Q4W Subjects randomized to placebo in PS0010 who do not achieve PASI90 response at Week 12 of PS0010 and are treated with bimekizumab 160mg Q4W in PS0011.
- Bimekizumab 64mg to Bimekizumab 64mg Subjects randomized to bimekizumab 64mg Q4W in PS0010 who achieve PASI90 response at Week 12 of PS0010 and continue to receive bimekizumab 64mg Q4W in PS0011.
- Bimekizumab 64mg to Bimekizumab 160mg Subjects randomized to bimekizumab 64mg Q4W in PS0010 who do not achieve PASI90 response at Week 12 of PS0010 and are treated with bimekizumab 160mg Q4W in PS0011.
- Bimekizumab 160mg Q4W to Bimekizumab 160mg Q4W Subjects randomized to bimekizumab 160mg Q4W or bimekizumab 320mg loading dose + 160mg Q4W in PS0010 who achieve PASI90 response at Week 12 of PS0010 and continue to receive bimekizumab 160mg Q4W in PS0011. Note that the PS0010 160mg Q4W groups with and without the loading dose are combined here.
- Bimekizumab 160mg Q4W to Bimekizumab 320mg Q4W Subjects randomized to bimekizumab 160mg Q4W or bimekizumab 320mg loading dose + 160mg Q4W in PS0010 who do not achieve PASI90 response at Week 12 of PS0010 and are treated with bimekizumab 320mg Q4W in PS0011. Note that the PS0010 160mg Q4W groups with and without the loading dose are combined here.
- Bimekizumab 320mg Q4W to Bimekizumab 320mg Q4W Subjects randomized to bimekizumab 320mg Q4W in PS0010 and continue on 320mg Q4W in PS0011. No distinction will be made between subjects that were or were not PASI90 responders at Week 12 of PS0010.
- Bimekizumab 480mg Q4W to Bimekizumab 320mg Q4W Subjects randomized to bimekizumab 480mg Q4W in PS0010 and continue on 320mg Q4W in PS0011. No distinction will be made between subjects that were or were not PASI90 responders at Week 12 of PS0010.

The treatment groups to be used in the presentations of safety and efficacy will depend on the objective of the summaries and will be specified accordingly.

#### Section 14.2 Planned safety analyses (now Section 14.3)

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA®). Treatment-emergent AEs will be defined as events that have a start date on or following the first administration of study treatment in PS0011 through the final administration of study treatment +119 days (covering the 17-week SFU Period). Treatment-emergent AEs will be categorized to treatment group based on the dose being received at the time of onset of the event. Tables will include columns for bimekizumab 320mg Q4W, bimekizumab 160mg Q4W, and All bimekizumab (ie, either dose of bimekizumab).

Change from Baseline variables will be defined relative to the Baseline measurement from PS0010.

#### Has been changed to:

Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA®). Treatment-emergent AEs will be defined as events that have a start date on or following the first administration of study treatment in PS0011 through the final administration of study treatment + 119 140 days (covering the 1720-week SFU Period). Treatment-emergent AEs will be categorized to by PS0011 treatment group based on the dose being received at the time of onset of the event. Tables will include columns for placebo, bimekizumab 64mg Q4W, bimekizumab 160mg Q4W, bimekizumab 320mg, and All bimekizumab (ie, any dose of bimekizumab) bimekizumab 320mg Q4W, bimekizumab 160mg Q4W, and All bimekizumab (ie, either dose of bimekizumab).

Change from Baseline variables will be defined relative to the Baseline measurement from PS0010.

## Change #99

### Section 14.2.1 Primary safety analysis (now Section 14.3.1)

All TEAEs will be summarized descriptively by treatment group, primary system organ class (SOC), high level term (HLT), and preferred term (PT). This summary will include the exposure adjusted incidence rate (EAIR) with associated 95% confidence interval and the exposure adjusted event rate (EAER).

## Has been changed to:

All TEAEs will be summarized descriptively by **PS0011** treatment group, primary SOC system organ class (SOC), high level term (HLT), and preferred term (PT). This summary will include the exposure adjusted incidence rate (EAIR) with associated 95% confidence interval and the exposure adjusted event rate (EAER).

#### Section 14.2.1 Primary safety analysis (now Section 14.3.1)

medication + 119 days (ie, the duration of the SFU Period).

a subject dies, patient exposure at risk is censored at the date of death. The sum of these exposure days at risk across subjects is converted to years for the EAIR and EAER calculations described above.

Has been changed to:

Patient exposure at risk in days will be defined as date of last administration of study medication - date of first administration of study medication in PS0011 + 119 140 days (ie, the duration of the SFU Period). If a subject dies, patient exposure at risk is censored at the date of death. The sum of these exposure days at risk across subjects is converted to years for the EAIR and EAER

Section 14.2.2 Other safety analyses (now Section 14.3.2) Additional tables will summarize TEAEs by intensional tables withdrawal from the Has been at the safety analyses (now Section 14.3.2) Has been at the safety analyse (now Section 14.3.2) Has been at the safety analyse (now Section 14.3.2) Has been at the safety analyse (now Section 14.3.2) Ha Additional tables will summarize TEAEs by intensity and relationship to study medication, TEAEs leading to withdrawal from the study, treatment-emergent SAEs, and deaths.

#### Has been changed to:

Additional tables will summarize TEAEs by intensity and relationship to study medication, TEAEs leading to withdrawal from the study, treatment-emergent SAEs, and deaths. Other AE summaries to be included will be specified in the SAP. All AE tables will be presented by PS0011 treatment group (including the All bimekizumab group).

### Change #102

Section 14.2.2 Other safety analyses (now Section 14.3.2)

The following text has been deleted

In order to evaluate if there is any difference in the TEAE profile of subjects who have dose adjustments, additional summaries will be generated and are described further here. With respect to dose adjustments, subjects will be classified into 1 of the following 3 groups:

- Nonadjusters—This group consists of subjects who do not experience a dose adjustment during the study.
- Single adjusters This group consists of subjects who experience just one dose adjustment during the study. Per the protocol, if just a single adjustment occurs, then that adjustment must be to go from bimekizumab 320mg Q4W to 160mg Q4W.
- Multiple adjusters—This group consists of subjects who experience more than 1 dose adjustment during the study. This means that the subjects in this group dose adjust

from bimekizumab 320mg Q4W to 160mg Q4W and then adjust back to 320mg Q4W (with further dose adjustments possible).

, variations thereof Summaries based on these 3 groups will be done for the TEAE overview, incidence of TEAEs (by SOC, HLT, and PT), and incidence of treatment emergent SAEs.

#### Change #103

#### Section 14.2.2 Other safety analyses (now Section 14.3.2)

Extent of exposure to study medication in PS0011 will be summarized using descriptive statistics. As with the primary summaries of TEAEs, extent of exposure will be presented with columns for bimekizumab 320mg Q4W, bimekizumab 160mg Q4W, and All bimekizumab

#### Has been changed to:

Extent of exposure to study medication in PS0011 will be summarized using descriptive statistics by PS0011 treatment group. As with the primary summaries of TEAEs, extent of exposure will be presented with columns for bimekizumab 320mg Q4W, bimekizumab 160mg Q4W, and All bimekizumab.

#### Change #104

## Section 14.2.2 Other safety analyses (now Section 14.3.2)

Change from Baseline in laboratory values. ECGs, and vital signs will be presented using descriptive statistics by PS0010 randomized treatment group and overall. As these variables are summarized over time and the initial values can be impacted by the randomized treatment in PS0010, the presentation by PS0010 randomized treatment group is intended to provide perspective on the change in these values starting with the initial PS0010 randomization through the 48-week Open-Label Treatment Period of PS0011. The table presentations will display descriptive statistics for the PS0010 Baseline and the observed and change from PS0010 Baseline results by scheduled visit for PS0011.

## Has been changed to:

Change from Baseline in laboratory values, ECGs, and vital signs will be presented using descriptive statistics by PS0010/**PS0011** randomized treatment group and overall. As these variables are summarized over time and the initial values can be impacted by the randomized treatment in PS0010, the presentation by PS0010/PS0011 randomized treatment group is intended to provide perspective on the change in these values starting with the initial PS0010 randomization through the 48-week **Open Label** Treatment Period of PS0011. The table presentations will display descriptive statistics for the PS0010 Baseline followed by descriptive statistics for the observed, change from PS0010 Baseline, and change from PS0011 results by scheduled visit for PS0011

#### Section 14.3 Planned PK analyses (now Section 14.4)

Bimekizumab plasma concentrations will be summarized for each treatment at each scheduled visit.

#### Has been changed to:

Bimekizumab plasma concentrations will be summarized for each treatment by PS0010/PS0011 treatment group at each scheduled visit. Descriptive statistics for the plasma concentrations at PS0010 Baseline will be presented followed by descriptive statistics for the observed, change from PS0010 Baseline, and change from PS0011 Baseline results for scheduled visits in PS0011. Summarizing in this manner based on the PS0010/PS0011 treatment group will allow for an evaluation of how changing doses (where applicable) impacted plasma concentrations relative to both the original (PS0010) Baseline as well as the new (PS0011) Baseline. For the descriptive statistics, geometric mean, geometric coefficient of variation, and 95% confidence interval for the geometric mean will be used instead of the arithmetic mean and standard deviation.

#### Change #106

Section 14.4 Planned immunological analyses (now Section 14.5)

Anti-bimekizumab antibody data will be summarized for each treatment at each scheduled visit.

### Has been changed to:

Anti-bimekizumab antibody data will be summarized by PS0010/PS0011 treatment group for each treatment at each scheduled visit. The summary of anti-bimekizumab antibody levels will follow a similar approach to that used for the summary of bimekizumab plasma concentrations. Additional analyses related to antibody positivity will be performed and will be described in greater detail in the SAP.

### Change #107

Section 14.5 Planned efficacy analyses (now Section 14.6)

Efficacy variables will be summarized based on the FAS. The summaries described in this section will provide data on maintenance of effect of open-label bimekizumab over 48 weeks. Additionally, it will allow an assessment of the impact of dose adjustments on efficacy results.

## Has been changed to:

Efficacy variables will be summarized based on the FAS. The summaries described in this section will provide data on maintenance of effect of open label bimekizumab study treatment over 48 weeks. Additionally, it will allow an assessment of the impact of dose adjustments on efficacy results.

#### Section 14.5 Planned efficacy analyses (now Section 14.6)

Responder efficacy variables (PASI75, PASI90, PASI100, IGA, and DLQI score of 0 or 1) will be summarized descriptively using counts and percentages by scheduled visit and PS0010 randomized treatment group and overall. The PASI responder variables are derived relative to the PS0010 Baseline. Missing data will be handled by using nonresponder imputation (NRI), meaning that subjects that discontinue early or who have missing data at a given time point are imputed as though they did not achieve the given response. Supportive summaries will be based on observed case data.

#### Has been changed to:

Responder efficacy variables (PASI75, PASI90, PASI100, IGA, and DLQI score of 0 or 1) will be summarized descriptively using counts and percentages by scheduled visit and PS0010/PS0011 randomized treatment group and overall. The PASI responder variables will be derived relative to both the PS0010 Baseline and the PS0011 Baseline with responder rates being presented side-by-side in applicable summary tables. Missing data will be handled by using nonresponder imputation (NRI), meaning that subjects that discontinue early or who have missing data at a given time point are imputed as though they did not achieve the given response. Supportive summaries will be based on observed case data.

#### Change #109

# Section 14.5 Planned efficacy analyses (now Section 14.6)

Continuous efficacy variables based on the change from Baseline (PASI, DLQI, BSA, mNAPSI, PSSI, PGADA, SF-36, and HADS) will be summarized using descriptive statistics by scheduled visit and PS0010 randomized treatment group and overall. The table presentations will display descriptive statistics for the PS0010 Baseline and the observed and change from PS0010 Baseline results by scheduled visit for PS0011. Figures for selected variables will also be generated in order to demonstrate the kinetics of response over time. Missing data will be handled by using multiple imputation (MI) via the Markov-Chain Monte Carlo (MCMC) method. Supportive summaries will be based on observed case data.

## Has been changed to:

Continuous efficacy variables based on the change from Baseline (PASI, DLQI, BSA, mNAPSI, PSSI, PGADA, SF-36, and HADS) will be summarized using descriptive statistics by scheduled visit and PS0010/PS0011 randomized treatment group-and overall. The table presentations will display descriptive statistics for the PS0010 Baseline, followed by descriptive statistics for the and the observed, and change from PS0010 Baseline, and change from PS0011 Baseline results by scheduled visit for PS0011. Figures for selected variables will also be generated in order to demonstrate the kinetics of response over time. Missing data will be handled by using multiple imputation (MI) via the Markov-Chain Monte Carlo (MCMC) method. Supportive summaries will be based on observed case data.

Section 14.5 Planned efficacy analyses (now Section 14.6)

The following text has been deleted

In addition to the summaries described above, the impact of dose adjustment on efficacy will be considered. This will be done primarily by summarizing efficacy variables by the 3 adjuster groups as defined in Section 14.3.2. Furthermore, a supportive analysis specifically for single adjusters will be performed in which PASI score will be summarized by visit, where Baseline is recalibrated for each individual subject and defined as the visit where the bimekizumab 160mg Q4W dose is initiated. The visits summarized will be in weeks relative to when the 160mg Q4W dose was started as opposed to the scheduled week of the PS0011 assessment. These summaries will be based on observed data only.

#### Change #111

# Section 14.6 Planned interim analysis and data monitoring (now Section 14.7)

A DMC will review the safety data on a recurring basis as outlined in the DMC charter. In addition to these ongoing reviews, an analysis combining safety data from PS0010 and PS0011 will be performed when the PS0010 study database is locked. This review will account for data in PS0010 as well as the accrued safety data in PS0011 available at the time of the PS0010 database lock. The details of this combined safety review of PS0010 and PS0011, including the events of interest to be considered, will be outlined in the DMC charter.

### Has been changed to:

A DMC will review the safety data on a recurring basis as outlined in the DMC charter. In addition to these ongoing reviews, an analysis combining safety data from PS0010 and PS0011 will be performed when the PS0010 study database is locked. This review analysis will account for data in PS0010 as well as the accrued safety data in PS0011 available at the time of the PS0010 database lock. At the time of the interim analysis, the DMC will be unblinded; however, the Sponsor study team will remain blind. The details of this combined safety review analysis of PS0010 and PS0011, including the events of interest to be considered, will be outlined in the DMC charter.

## Change #112

#### Section 15.1 Informed consent

Prior to participation in the study, the written Informed Consent Form should be signed and personally dated by the subject, or his/her legal representative, and by the person who conducted the informed consent discussion (Investigator or designee). The subject or his/her legal representative must receive a copy of the signed and dated Informed Consent Form. As part of the consent process, each subject must consent to direct access to his/her medical records for study-related monitoring, auditing, IRB/IEC review, and regulatory inspection.

#### Has been changed to:

Prior to participation in the study, the written Informed Consent Form should be signed and as on variations thereof. personally dated by the subject, or his/her legal representative, and by the person who conducted the informed consent discussion (Investigator or designee). The subject or his/her legal representative must receive a copy of the signed and dated Informed Consent Form. As part of the consent process, each subject must consent to direct access to his/her medical records for study-related monitoring, auditing, IRB/IEC review, and regulatory inspection.

### Change #113

#### **Section 15.2 Subject identification cards**

Upon signing the Informed Consent and Assent form (as applicable), the subject or legal representative will be provided with a subject identification card in the language of the subject. The Investigator will fill in the subject identifying information and medical emergency contact information. The Investigator will instruct the subject to keep the card with him/her at all times.

#### Has been changed to:

Upon signing the Informed Consent-and Assent form (as applicable), the subject or legal representative will be provided with a subject identification card in the language of the subject. The Investigator will fill in the subject identifying information and medical emergency contact information. The Investigator will instruct the subject to keep the card with him/her at all times.

### Change #114

**Section 17 References** 

The following reference was added

Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0. National Institutes of Health, National Cancer Institute, Division of Cancer Treatment and Diagnosis. http://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm. Louised to Lised to This document cannot be used to Updated 26 Jul 2016.

#### 19 DECLARATION AND SIGNATURE OF INVESTIGATOR

I confirm that I have carefully read and understood this protocol and agree to conduct this clinical study as outlined in this protocol, according to current Good Clinical Practice and local laws and requirements.

I will ensure that all subinvestigators and other staff members read and understand all aspects of this protocol.

I have received and read all study-related information provided to me.

The objectives and content of this protocol as well as the results deriving from it will be treated confidentially, and will not be made available to third parties without prior authorization by UCB.

All rights of publication of the results reside with UCB, unless other agreements were made in a separate contract.

| Investigator: | ication and all. |
|---|---|
| Printed name | Date/Signature |
| aused to support any mail. | |
| Printed name Printed name Printed name This document cannot be used to support any market. | |

actice.

Actice.

Act


### **PS0011 Protocol Amendment 1**

extensions of variations thereof. Aleaning of Signature

Clinical Approval

Clinical Approval

Clinical Approval

Read to support any marketing authorization application and the sead to support any marketing authorization and the sead to support any marketing authorization and the sead to support any marketing authorization and the sead to support any marketing authorization and support and support any marketing authorization and support any marketing authorization and support any marketing authorization and support any marketing authorization and support any marketing authorization and support and support any marketing authorization and support any marketing authorization and support an Server Approval Date (dd-mon-yyyy (HH:mm)) 12-Aug-2016 16:22 GMT+0 12-Aug-2016 18:33 GMT+0